

# STATISTICAL ANALYSIS PLAN

Study CRO-14-122 - Sponsor code CHL.1/02-2014

# Spinal anaesthesia with Chloroprocaine HCl 1% for elective lower limb procedures of short duration: a prospective, randomised, observer-blind study in adult patients

Prospective, single centre, randomised, parallel-group, observer-blind, three doses, efficacy and pharmacokinetic study

**EudraCT Number: 2014-003778-17** 

Investigational medicinal product: Chloroprocaine HCl 1% solution for injection (10

mg/mL), Sintetica S.A., Switzerland

Indication: Spinal anaesthesia

Sponsor: Sintetica S.A., via Penate 5, CH-6850 Mendrisio,

Switzerland

Phone: +41.91.640.42.50 Fax: +41.91.646.85.61

Study investigators: Principal Investigator: Stefano Bonarelli, MD

Istituto Ortopedico Rizzoli, SC Anestesia e Terapia

Intensiva post-operatoria e del dolore IOR-IRCCS,

via G.C. Pupilli 1 - 40136 Bologna, Italy

Phone: +39.051.6366356 Fax: +39.051.6366647

Email: stefano.bonarelli@ior.it

Development phase: Phase II

Version and date: Final version 1.0, 02FEB2016

This study was conducted in accordance with Good Clinical Practice (GCP), ICH topic E6

Property of the Sponsor.

May not be used, divulged, published or otherwise disclosed without the consent of the Sponsor

This document comprises 32 pages plus appendices



# 1 STATISTICAL ANALYSIS PLAN VERSIONS' HISTORY

| Version | Date of Issue | Reason for change |
|---|---|---|
| Draft version 0.1 | 30DEC2015 | Issue of the first draft |
| Draft version 0.2 | rsion 0.2 Updated by Matteo Rossini in order to impleme required by Chiara Leuratti | |
| Final version 1.0 | 02FEB2016 | Final version issued by Matteo Rossini |



2 STATISTICAL ANALYSIS PLAN APPROVAL AND ACKNOWLEDGEMENT

2.1 SPONSOR APPROVAL AND ACKNOWLEDGEMENT

Sintetica S.A., Switzerland

Sponsor Representative (for approval)

Elisabetta Donati, Corporate Director Scientific Affairs

03 FEB 2016

Signature



# 2.2 CRO APPROVAL AND ACKNOWLEDGEMENT

CROSS Research S.A. and CROSS Metrics S.A., sister-owned companies

| Statistical Analysis of Demo<br>Matteo Rossini, Biometry Ma<br>OZFER ZO16<br>Date | egraphy, Efficacy and Safety (for approval) anager, Unit Head Signature |
|---|---|
| Pharmacokinetic Analysis (<br>Luca Loprete, Senior Pharma | |
| Date | Signature |
| Medical Writing (for appro<br>Chiara Leuratti, Clinical Proj | ects Unit Head Clei anabenat |
| Date | Signature |
| Coordination (for acknowledgement only) Emanuela Terragni, Clinical Project Leader | |
| <u>02∓€8 2016</u><br>Date | Ema mela lovra smi<br>Signature |



| 3 | TABLE OF CONTENTS |
|---|-------------------|
| U | THE OF COLLECTE |

| | STATISTICAL ANALYSIS PLAN | 1 |
|----------|------------------------------------------------|----|
| 1 | STATISTICAL ANALYSIS PLAN VERSIONS' HISTORY | 2 |
| 2 | STATISTICAL ANALYSIS PLAN APPROVAL AND | |
| | ACKNOWLEDGEMENT | 3 |
| 2.1 | SPONSOR APPROVAL AND ACKNOWLEDGEMENT | 3 |
| 2.2 | CRO APPROVAL AND ACKNOWLEDGEMENT | 4 |
| 3 | TABLE OF CONTENTS | 5 |
| 4 | TABLES | 7 |
| 5 | LIST OF ABBREVIATIONS | 8 |
| 6 | INTRODUCTION | 10 |
| 6.1 | Changes with respect to the study protocol | 10 |
| 7 | STUDY DESCRIPTION | 11 |
| 7.1 | Study Objective | 11 |
| 7.1.1 | Primary end-point | 11 |
| 7.1.2 | Secondary end-points | 11 |
| 7.2 | Study Design | 11 |
| 8 | STUDY POPULATION | 13 |
| 8.1 | Target population | 13 |
| 8.2 | Inclusion criteria | 13 |
| 8.3 | Exclusion criteria | 13 |
| 8.3.1 | Not allowed treatments and other treatments | 14 |
| 9 | STUDY SCHEDULE | 15 |
| 9.1 | Study visits and procedures | 15 |
| 9.2 | Diet and lifestyle | 17 |
| 10 | SUBJECT IDENTIFICATION AND ASSIGNMENT OF STUDY | |
| | TREATMENT | 18 |
| 10.1 | Unique subject identifier | 18 |
| 10.2 | Randomisation | 18 |
| 10.3 | Treatment allocation | 18 |
| 10.4 | Blinding | 18 |
| 11 | EVALUATION PARAMETERS | 20 |
| 11.1 | Study variables | 20 |
| 11.1.1 | Primary variables | 20 |
| 11.1.2 | Secondary variables | 20 |
| 11.1.2.1 | Efficacy variables | 20 |
| 11.1.2.2 | Pharmacokinetic variables | 20 |
| 11.1.2.3 | Safety variables | 20 |
| 11.2 | Efficacy assessments | 21 |
| 11.3 | Pharmacokinetic assessments | 22 |
| 11.4 | Safety assessments | 22 |
| 12 | STATISTICAL METHODS | 23 |
| 12.1 | Analysis sets | 23 |




Statistical analysis plan CRO-14-122 Sponsor code CHL.1/02-2014 Chloroprocaine 1% - Spinal block Final version 1.0, 02FEB2016

| 14 | APPENDICES | 32 |
|---|---|---|
| 13 | REFERENCES | 31 |
| 12.7.8 | Sedation and premedication | 30 |
| 12.7.7 | Spinal injection | 30 |
| 12.7.6 | Modified Aldrete's scoring scale | 30 |
| 12.7.5 | Incidence of TNS at 24 h (day 2) and 6 days±1 (day 7±1) after spinal injection (T <sub>sp</sub> ) | 30 |
| 12.7.4 | Pain assessment at the site of injection and at the site of surgery | 30 |
| 12.7.3 | ECG | 30 |
| 12.7.2 | Vital signs | 29 |
| 12.7.1 | Adverse events | 29 |
| 12.7 | Safety and tolerability evaluation | 29 |
| 12.6 | Analysis of pharmacokinetic parameters | 28 |
| 12.5.4 | Effectiveness of anaesthesia and quality of spinal block | 28 |
| 12.5.3 | Time to events and maximum level of sensory block | 27 |
| 12.5.2 | Sensory and motor block assessment | 27 |
| 12.5.1 | Surgical procedure | 27 |
| 12.5 | Analysis of efficacy parameters | 27 |
| 12.4.12 | Pregnancy test | 27 |
| 12.4.11 | Subjects study visits | 27 |
| 12.4.10 | Prior and concomitant medications | 27 |
| 12.4.9 | Physical examination | 26 |
| 12.4.8 | Medical and surgical history | 26 |
| 12.4.7 | Demography | 26 |
| 12.4.6 | Discontinued subjects | 26 |
| 12.4.5 | Protocol deviations | 26 |
| 12.4.4 | Inclusion/exclusion criteria not met | 26 |
| 12.4.3 | Subjects excluded from the efficacy and/or PK and/or Safety analysis | 26 |
| 12.4.2 | Analysis sets | 26 |
| 12.4.1 | Subjects' disposition | 25 |
| 12.4 | Demographic, baseline and background characteristics | 25 |
| 12.3.3 | Missing values of safety assessments | 25 |
| 12.3.2 | Missing values of pharmacokinetic assessments | 25 |
| 12.3.1 | Missing values of efficacy assessments | 25 |
| 12.3 | Handling of missing data | 25 |
| 12.2 | Sample size and power considerations | 25 |
| 12.1.4 | Reasons for exclusion from the PK sets | 24 |
| 12.1.3 | Reasons for exclusion from the Per Protocol set | 24 |
| 12.1.2 | Reasons for exclusion from the Full Analysis Set | 24 |
| 12.1.1 | Definitions | 23 |

#### ${\it CONFIDENTIAL}$



Statistical analysis plan CRO-14-122 Sponsor code CHL.1/02-2014 Chloroprocaine 1% - Spinal block Final version 1.0, 02FEB2016

# 4 TABLES

Table 7.2.1 Study schedule

12



#### 5 LIST OF ABBREVIATIONS

ADR Adverse Drug Reaction

AE Adverse Event

ALCOA Attributable-Legible-Contemporaneous-Original-Accurate

ANOVA Analysis of Variance

ASA American Society of Anesthesiologists

BMI Body Mass Index
BP Blood Pressure
BW Body Weight
CA Competent Authority

CABA 2-chloro-4-aminobenzoic acid

CDISC Clinical Data Interchange Standards Consortium

CSF Cerebrospinal fluid
CI Confidence Interval
CNS Central Nervous System
CRF Case Report Form

CRO Contract Research Organisation

Clinical Study Protocol **CSP** Clinical Study Report **CRS** CVCoefficient of Variation **DBP** Diastolic Blood Pressure **Ethics Committee** EC **ECG** Electrocardiogram Early Termination Visit **ETV** Full Analysis Set **FAS** First Subject First Visit **FSFV GCP** Good Clinical Practice **GLP** Good Laboratory Practice

HR Heart Rate

IB Investigator's Brochure

ICH International Conference on Harmonisation

IRB/IEC Institutional Review Board/Independent Ethics Committee

IMP Investigational Medicinal Product

IUD Intra-Uterine Device

IV Intravenous

IVRA Intravenous Regional Anaesthesia

LSLV Last Subject Last Visit

MedDRA Medical Dictionary for Regulatory Activities

NA Not Applicable NRS Numerical rating scale

NSAIDs Non-Steroidal Anti-Inflammatory Drugs

OTC Over The Counter
PK Pharmacokinetic
PP Per Protocol
PT Preferred Term

PTAE Pre-Treatment Adverse Event
SAE Serious Adverse Event
SBP Systolic Blood Pressure

SB<sub>max</sub> Maximum level of sensory block SBML Sensory block metameric level

SD Standard Deviation

SmPC Summary of Product Characteristics

SOC System Organ Class

SOPStandard Operating ProcedureSpO2Peripheral oxygen saturationSDTMStudy Data Tabulation ModelTEAETreatment-Emergent Adverse Event




Statistical analysis plan CRO-14-122 Sponsor code CHL.1/02-2014 Chloroprocaine 1% - Spinal block Final version 1.0, 02FEB2016

T<sub>ea</sub> Time to regression of spinal block (i.e. end of anaesthesia)

T<sub>hd</sub> Time to eligibility for home discharge

T<sub>mb</sub> Time to onset of motor block

 $\begin{array}{ll} T_{SBmax} & Time \ to \ maximum \ level \ of \ sensory \ block \\ T_{pa} & Time \ to \ first \ post-operative \ analgesia \end{array}$ 

 $T_{ra}$  Time to administration of rescue anaesthesia or rescue analgesia

Time to regression of two dermatomers with respect to the maximum level of sensory block

 $T_{rmb}$  Time to regression of motor block  $T_{rs}$  Time to readiness for surgery

 $T_{S1}$  Time to regression of sensory block to S1

 $\begin{array}{ll} T_{sb} & Time \ to \ onset \ of \ sensory \ block \\ T_{sp} & Time \ of \ spinal \ injection \\ T_{ua} & Time \ to \ unassisted \ ambulation \\ T_{uv} & Time \ to \ first \ spontaneous \ urine \ voiding \\ TNS & Transient \ Neurological \ Symptoms \end{array}$ 

WHODDE World Health Organisation Drug Dictionary Enhanced



#### 6 INTRODUCTION

The statistical analysis of demographic, efficacy and safety data and the PK analysis will be performed by the Contract Research Organisation (CRO) Biometry Unit. The present Statistical Analysis Plan (SAP) was compiled by the CRO Biometry Unit, reviewed by the Sponsor and finalized before database lock.

# 6.1 Changes with respect to the study protocol

No changes with respect to the final version 2.0 of the study protocol (1) and the final version 1.0 of the amendment number 3 (2) are present in the SAP.



#### 7 STUDY DESCRIPTION

# 7.1 Study Objective

The objective of this study is to evaluate the effect of the three doses of Chloroprocaine HCl 1% (30, 40 and 50 mg) for spinal anaesthesia in adult patients undergoing short duration elective surgery of the lower limb.

#### 7.1.1 Primary end-point

• The primary end-point of the study is to evaluate the efficacy of the three Chloroprocaine HCl 1% doses (30 mg [D1], 40 mg [D2] and 50 mg [D3]) in terms of time to complete regression of spinal block (T<sub>ea</sub>).

# 7.1.2 Secondary end-points

- To evaluate the efficacy of three Chloroprocaine HCl 1% doses (D1, D2 and D3) in terms of time to onset of sensory block (T<sub>sb</sub>), time to onset of motor block (T<sub>mb</sub>), time to readiness for surgery (T<sub>rs</sub>), time to regression of motor block, time to unassisted ambulation (T<sub>ua</sub>), time to regression of sensory block to S1 (T<sub>S1</sub>), Sensory block metameric levels during the block, Maximum level of sensory block (SB<sub>max</sub>), time to maximum level of sensory block (T<sub>SBmax</sub>), time to regression of two dermatomers with respect to the maximum level of sensory block (T<sub>rd</sub>), time to first spontaneous urine voiding (T<sub>uv</sub>), time to administration of rescue anaesthesia or rescue analgesia (T<sub>ra</sub>), time to first post-operative analgesia (T<sub>pa</sub>), time to eligibility for home discharge (T<sub>hd</sub>), proportion of patients achieving effective anaesthesia, quality of spinal block;
- To assess the concentration of chloroprocaine and its metabolite 2-chloro-4-aminobenzoic acid (CABA) in plasma after administration of D1, D2 and D3;
- To assess the excretion of CABA in urine (as % of the administered dose);
- To investigate the safety and tolerability of the administered Chloroprocaine HCl 1% doses on the basis of treatment emergent adverse events, transient neurological symptoms (TNS), vital signs (blood pressure, heart rate and peripheral oxygen saturation [SpO<sub>2</sub>]) check and ECG recording.

# 7.2 Study Design

Prospective, single centre, randomised, parallel-group, observer-blind, three doses, efficacy and pharmacokinetic study.

For details on the study schedule see below (Table 7.2.1).



Table 7.2.1 Study schedule

| ACTIVITIES | Screening<br>Phase | Treatment<br>Phase | | Follow-up<br>Phase | |
|---|---|---|---|---|---|
| Visit | Visit 1<br>Days -14/1 | Visit 2<br>Day 1 | Final Visit<br>or ETV<br>Day1/2 | Day 2<br>24 h<br>post-surgery | Day 7±1 |
| Informed consent | X | | | | |
| Demography and lifestyle | X | | | | |
| Medical/surgical history | X | | | | |
| Physical examination | Х | | | | |
| Previous and concomitant medication | Х | X | X | Х | X |
| Height | Х | | | | |
| Body weight | Х | | | | |
| Vital signs (blood pressure, heart rate) <sup>1</sup> | Х | X | X | | |
| $SpO_2^1$ | Х | X | X | | |
| ECG <sup>1</sup> | | X | X | | |
| Pregnancy test (urine) | X | | | | |
| Inclusion/exclusion criteria | Х | X | | | |
| Enrolment and Randomisation | | X | | | |
| I.v. Midazolam premedication | | X | | | |
| Ringer's solution infusion | | $\mathbf{x}^2$ | | | |
| Spinal injection | | X | | | |
| Surgery (< 40 min) | | X | | | |
| Sensory block assessment | | x <sup>5</sup> | | | |
| Motor block assessment | | x <sup>5</sup> | | | |
| Blood sampling <sup>3</sup> | | X | | | |
| Urine collection <sup>4</sup> | | X | | | |
| Pain assessment | | $\mathbf{x}^7$ | $\mathbf{x}^7$ | $\mathbf{x}^7$ | $\mathbf{x}^7$ |
| TNS questionnaire | | | | X | X |
| Home discharge <sup>6</sup> | | | X | X | |
| Adverse events monitoring | X | X | X | Х | X |

- 1. Vital signs and SpO<sub>2</sub> at screening, at baseline, during the block until the end of the anaesthesia and during post-operative recovery (final visit). ECG (if foreseen by the standard hospital procedures) at baseline, during the block until the end of the anaesthesia and during post-operative recovery (final visit)
- 2. If needed
- 3. Blood samples for PK analysis were collected at baseline and at 5, 10, 30 and 60 min after spinal puncture
- 4. Urine was collected for PK analysis at the time of first spontaneous voiding
- 5. The evolution of both sensory and motor blocks, including sensory block metameric level, were evaluated by a blinded observer every 2 min until readiness for surgery, every 5 min until the maximum level is reached (two consecutive observations with the same level of sensory block) and then every 5 min until regression of two dermatomers with respect to the maximum level of sensory block. After that, sensory and motor block assessments were repeated every 30 min until regression of motor block and complete regression of sensory block to S1 (if compatible with surgical procedure)
- 6. Patients were discharged on Day 1 or on a following day after the criteria for discharge, including Aldrete's scoring scale criteria, are met and according to the hospital's standard procedures. In case of discontinuation, subjects underwent an early termination visit (ETV)
- 7. Pain at the site of injection and pain at the site of surgery was assessed using a 0-10 NRS, where 0 indicates "No pain" and 10 indicates "Worst imaginable pain". At 24 h (day 2) and  $6\pm 1$  days (day  $7\pm 1$ ) after spinal puncture, pain assessment was performed using the TNS questionnaire



#### 8 STUDY POPULATION

# 8.1 Target population

Forty-five (45) male/female patients, 15/dose group, aged 18-65 years, scheduled for lower limb surgery (< 40 min) under spinal block, i.e. requiring ≥ T12 metameric level of sensory block.

#### 8.2 Inclusion criteria

To be enrolled in this study, subjects must fulfil all these criteria:

- 1. Sex, age and surgery: male/female patients, 18-65 years old, scheduled for short duration (less than 40 min) lower limb surgery requiring ≥ T12 metameric level of sensory block
- 2. Body Mass Index (BMI): 18 32 kg/m<sup>2</sup> inclusive
- 3. ASA physical status: I-II
- 4. *Informed consent*: signed written informed consent before inclusion in the study
- 5. *Full comprehension*: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study

# 8.3 Exclusion criteria

Subjects meeting any of these criteria were not enrolled in the study:

- 1. *Physical findings*: clinically significant abnormal physical findings which could interfere with the objectives of the study. Contraindications to spinal anaesthesia. History of neuromuscular diseases to the lower extremities
- 2. ASA physical status: III-V
- 3. Further anaesthesia: patients expected to require further anaesthesia
- 4. *Allergy*: ascertained or presumptive hypersensitivity to the active principle and/or formulations ingredients; ascertained or presumptive hypersensitivity to the ester type and major anaesthetics
- 5. *Diseases*: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study; ascertained psychiatric and neurological diseases, sepsis, blood coagulation disorders, severe cardiopulmonary disease, thyroid disease, diabetes or other neuropathies
- 6. *Investigative drug studies*: participation in the evaluation of any investigational product for 3 months before this study, calculated from the first day of the month following the last visit of the previous study
- 7. *Drug, alcohol*: history of drug or alcohol abuse
- 8. *Blood donation*: blood donations in the 3 months before this study



- 9. *Pregnancy and lactation*: missing or positive pregnancy test at screening, pregnant or lactating women
- 10. *Chronic pain syndromes*: patients with chronic pain syndromes (taking opioids, antidepressants, anticonvulsant agents or chronic analgesic therapy)
- 11. *Medications*: medication known to interfere with the extent of spinal blocks for 2 weeks before the start of the study. Hormonal contraceptives for females are allowed.

#### 8.3.1 Not allowed treatments and other treatments

No medication known to interfere with the extent of spinal block (see chloroprocaine SmPC), in particular no therapeutic use of opioids, was allowed for 2 weeks before the start of the study and during the whole study duration. Hormonal contraceptives for women are allowed.

The area to be operated was aseptically prepared with disinfectants, e.g. chlorhexidine, not containing iodine. Iodine-based disinfectants must not be used. The information on the iodine-free disinfectant used for each patient was reported in the individual CRFs.

After admission to the operating theatre and before the spinal puncture all patients were premedicated with i.v. midazolam (about 0.03 mg/kg). In addition, only if the investigator deems it necessary, patients were premedicated with 500 or 1000 mL of Ringer's solution administered by infusion.

Post-operative analgesia was given to all patients, if necessary, according to the hospital standard procedures.



#### 9 STUDY SCHEDULE

The schedule of the study is summarised at page 12 (Table 7.2.1).

# 9.1 Study visits and procedures

The study protocol foresees a screening visit, one study treatment for each patient, followed by post-operative recovery, final visit and 2 follow-ups. Maximum study duration will be 22 days, screening visit and follow-up included. A written informed consent was obtained before any study assessment or procedure.

The first subject first visit (FSFV) is defined as the 1<sup>st</sup> visit performed at the clinical centre by the 1<sup>st</sup> screened subject. The last subject last visit (LSLV) is defined as the last telephonic follow-up performed by the last subject, i.e. the last visit foreseen by the study protocol, independently of the fact that the subject is a completer or a withdrawn subject.

The following phases, visits and procedures were performed:

#### > Screening phase

Screening - visit 1: between day -14 and day 1

# > Treatment phase

• Visit 2 - day 1: anaesthesia and surgery

#### Follow-up phase

- Post-operative recovery day 1 (immediately after surgery)
- Final visit/early termination visit (ETV). In case of early discontinuation, discontinued subjects underwent an early termination visit (ETV)
- Day 2 (i.e. 24 h after surgery) Telephonic follow-up, if the patient has left the hospital on day 1
- Day 7±1 (6±1 days after surgery) Telephonic follow-up



| | Day | Procedures/Assessments | Notes |
|---|---|---|---|
| Screening - Visit 1 | From day -14<br>to day 1 | <ul> <li>Explanation to the subject of study aims, procedures and possible risks</li> <li>Informed consent signature</li> <li>Screening number (as S001, S002, etc.)</li> <li>Demographic data and life style recording</li> <li>Previous/concomitant medications</li> <li>Routine pre-surgery assessments according to the hospital standard procedures, including medical/surgical history, physical examination, height, weight, vital signs (blood pressure, heart rate), SpO<sub>2</sub></li> <li>Urine pregnancy test for women</li> <li>Inclusion/exclusion criteria evaluation</li> <li>AE monitoring</li> </ul> | |
| Treatment - Visit 2 | Day 1 | <ul> <li>Concomitant medications</li> <li>Adverse events (before, during and after block placement and surgery)</li> <li>Inclusion/exclusion criteria evaluation</li> <li>Subject randomisation</li> <li>Vital signs, SpO<sub>2</sub> and ECG (if foreseen by the standard hospital procedures)</li> <li>Premedication 1: i.v. midazolam – all patients</li> <li>Premedication 2: 500 or 1000 mL of Ringer's solution, if needed</li> <li>Anaesthesia administration (intrathecal injection)</li> <li>Pain assessment (0-10 NRS)</li> <li>Post-operative analgesia according to the hospital standard procedures</li> <li>Sensory and motor block assessments, including sensory block metameric level</li> <li>Quality of spinal block assessment</li> <li>Surgery (&lt; 40 min)</li> <li>Blood sampling for PK analysis at pre-dose (0h) and at 5, 10, 30 and 60 min after spinal puncture</li> <li>Urine collection for PK analysis at the time of first urine voiding</li> </ul> | |
| Final Visit/ETV | Day 1/2 or<br>upon<br>discontinuation<br>for ETV | <ul> <li>Final assessments, including pain assessment (0-10 NRS), before discharge according to the hospital's standard procedures</li> <li>Aldrete's scoring scale</li> <li>Vital signs (BP, HR, SpO<sub>2</sub>) and ECG (if foreseen by the standard hospital procedures)</li> <li>AE and concomitant medications</li> <li>Discharge (when criteria for discharge are met and according to the hospital's standard procedures)</li> <li>In case of clinically significant results at the final visit, the subjects will be followed-up by the investigator until the normalisation of the concerned clinical parameter(s)</li> </ul> | Standardised meals will be served according to the hospital procedures. Patients will be discharged on Day 1 or on a following day after the criteria for discharge are met and according to the hospital's standard procedures. |



| | Day | Procedures/Assessments | Notes |
|---|---|---|---|
| Follow-up | , | <ul> <li>AE, in particular TNS (questionnaire)</li> <li>Concomitant medications</li> </ul> | |
| Follow-up | Day 7±1<br>post-surgery | <ul> <li>AE, in particular TNS (questionnaire)</li> <li>Concomitant medications</li> </ul> | |

# 9.2 Diet and lifestyle

Study participants underwent study procedures as outpatients or in-patients, according to the decision of the study investigator. Patients arrived at the clinical centre either in the morning of the scheduled surgery day or the previous evening, according to the hospital requirements, and were discharged on Day 1 or on a following day after meeting the criteria for discharge, according to the hospital procedures.

On day 1, patients were under fasting conditions before surgery. Clear fluids intake was allowed until 2 h before surgery. The patients remained under fasting conditions until surgery has been completed and according to the investigator's opinion. Meals were served according to the hospital's standard procedures.



# 10 SUBJECT IDENTIFICATION AND ASSIGNMENT OF STUDY TREATMENT

# 10.1 Unique subject identifier

All the subjects who sign the informed consent form for the present study will be coded with "unique subject identifiers" when data are extracted from the study database into the domains of the CDISC SDTM model. The unique subject identifier consists of the sponsor study code (i.e. CHL.1/2-2014), the 3-digit centre number (i.e. 001), the 4-digit screening number (e.g. S001, S002, etc.) and, if applicable, the 3-digit subject randomisation number (i.e. 001, 002, ..., 046). Study code, centre number, screening number and subject randomisation number are separated by slashes ("/"). The last 8 digits of the unique subject identifier (enrolled subjects), corresponding to the subject screening and subject randomisation numbers separated by a slash, will appear as subject identifier in the individual listings and figures of the clinical study report and will be used to identify the subjects in in-text tables or wording (if applicable).

#### 10.2 Randomisation

The randomisation list was computer generated by the Biometry Unit of the Clinical Contract Research Organization (CRO), using the PLAN procedure of the SAS® system version 9.3 (TS1M1) (4) or higher for Windows (the version will be stated in the final clinical study report). The randomisation list will be attached to the final clinical study report.

#### 10.3 Treatment allocation

Patients were allocated to D1, D2 or D3 dose group in a 1:1:1 ratio according to the study randomisation list.

Randomisation number was given to the patients on study Day 1 and was used to allocate each patient to a dose group, as detailed above.

The 5-mL ampoules with the investigational product were numbered. Each patient was allocated the product ampoule corresponding to his/her randomisation number.

#### 10.4 Blinding

This is an observer-blind study. No masking procedure was applied.

The physician preparing and the physician administering the doses was not involved in data recording and evaluation. An independent blinded observer evaluated sensory and motor blocks for each patient.

Emergency envelopes containing individual randomisation codes were sent to the clinical centre. Breaking of an individual randomisation code during the study was allowed only when knowledge of the code was essential for the patient's health. In this case, only the envelope related to the concerned subject would have been opened. Individual code breaking would have been clearly reported in the patient CRF and on the envelope.




Statistical analysis plan CRO-14-122 Sponsor code CHL.1/02-2014 Chloroprocaine 1% - Spinal block Final version 1.0, 02FEB2016

The clinical centre also received individual kit replacement envelopes. If a reserve kit needed to be used, the kit replacement envelope would be opened and the injectable solution would be prepared in such a way that the observer blind condition of the study is maintained. The date and the reason for kit replacement envelope opening would be recorded on the envelope.

No breaking of any individual randomisation code occurred during the study and the reserve kit number K050 was used for the subject with randomisation number 046, who was enrolled in addition to the originally scheduled 45 patients (2).



#### 11 EVALUATION PARAMETERS

# 11.1 Study variables

# 11.1.1 Primary variables

Time to regression of spinal block (T<sub>ea</sub>), defined as the time when Bromage score returns to 0 and sensitive perception returns to S1.

#### 11.1.2 Secondary variables

#### 11.1.2.1 Efficacy variables

- Time to onset of sensory block (T<sub>sb</sub>)
- Time to onset of motor block  $(T_{mb})$
- Time to readiness for surgery ( $T_{rs}$ ), defined as loss of pinprick sensation at the required metameric level  $\geq T12$  with a modified Bromage score  $\geq 2$
- Time to regression of motor block (Bromage score = 0;  $T_{rmb}$ )
- Time to unassisted deambulation (T<sub>ua</sub>)
- Time to regression of sensory block to S1 (T<sub>S1</sub>)
- Sensory block metameric level (SBML, assessed until resolution of sensory block to S1)
- Maximum level of sensory block (SB<sub>max</sub>)
- Time to maximum level of sensory block  $(T_{SBmax})$
- Time to regression of two dermatomers with respect to the maximum level of sensory block  $(T_{rd})$
- Time to eligibility for home discharge (T<sub>hd</sub>)
- Time to first spontaneous urine voiding (T<sub>uv</sub>)
- Time to administration of rescue anaesthesia or rescue analgesia  $(T_{ra})$
- Time to first post-operative analgesia (T<sub>pa</sub>)
- Proportion of patients achieving an effective anaesthesia
- Quality of spinal block

#### 11.1.2.2 Pharmacokinetic variables

- Plasma concentrations of chloroprocaine and CABA at baseline (i.e. before spinal puncture) and at 5, 10, 30 and 60 min after spinal puncture
- Urine excretion of CABA from spinal puncture to time of first urine voiding

#### 11.1.2.3 Safety variables

• Treatment-emergent adverse events throughout the study



- Incidence of TNS at 24 h (day 2) and 6±1 days (day 7±1) after spinal puncture (Tsp)
- Vital signs (BP, HR and SpO<sub>2</sub>), ECG
- Pain assessment at the site of injection and at the site of surgery performed immediately after regression of spinal block, at discharge (final visit/ETV), 24 h (day 2) and 6±1 days (day 7±1) after spinal puncture

# 11.2 Efficacy assessments

Sensory and motor block assessment procedures and evaluations are detailed in section 7.2 of the study protocol (1).

Efficacy assessments are based on the following variables:

| Parameter | Description |
|---|---|
| Time (min) to onset of sensory block (T <sub>sb</sub> ) | Time period from spinal injection ( $T_{sp}$ ; time 0 h) to achievement of sensory block (see section 7.2 of the study protocol [1]). |
| Time (min) to onset of motor block (T <sub>mb</sub> ) | Time period from spinal injection ( $T_{sp}$ ; time 0 h) to achievement of motor block (see section 7.2 of the study protocol [1]). |
| Time (min) to readiness for surgery $(T_{rs})$ | Time period from completion of spinal injection ( $T_{sp}$ ; time 0 h) to achievement of sensory and motor block adequate for surgery, i.e. loss of Pinprick sensation and Bromage's score $\geq$ 2 at the required metameric level $\geq$ T12 |
| Time (h) to regression of spinal block (T <sub>ea</sub> ) | Time period from spinal injection ( $T_{sp}$ ; time 0 h) to the time when the Bromage score returns to 0 and sensitive perception returns to S1 |
| Time (h) to regression of sensory block to S1 (T <sub>S1</sub> ) | Time period from spinal injection (T <sub>sp</sub> ; time 0 h) to the time when sensitive perception has returned to S1 |
| Time (h) to regression of motor block (T <sub>rmb</sub> ) | Time period from spinal injection ( $T_{sp}$ ; time 0 h) to the time when the Bromage score has returned to 0 |
| Time (h) to unassisted ambulation (T <sub>ua</sub> ) | Time period from spinal injection ( $T_{sp}$ ; time 0 h) to the time when the patient can walk unassisted |
| Sensory block metameric level (SBML) | Metameric level of sensory block assessed from spinal injection ( $T_{sp}$ ; time 0 h) until regression of sensory block to S1 |
| Maximum level of sensory block (SB <sub>max</sub> ) | Maximum metameric level of sensory block (decreased or absent sensation) achieved |
| Time (min) to maximum level of sensory block $(T_{SBmax})$ | Time period from spinal injection (Tsp; time 0 h) to the time when the maximum metameric level of sensory block is achieved (consider the time of the first of the two consecutive observations with the same level of sensory block) |



| Parameter | Description |
|---|---|
| Time (h) to regression of two dermatomers with respect to the maximum level of sensory block $(T_{rd})$ | Time period from spinal injection ( $T_{sp}$ ; time 0 h) to the time when the sensory block decrease of two dermatomers with respect to the maximum level of sensory block |
| Time (h) to eligibility for home discharge (T <sub>hd</sub> ) | Time period from spinal injection (T <sub>sp</sub> ; time 0 h) to the time when the criteria from discharge are met, even if according to the hospital procedures the patient is discharged at a later time |
| Time (h) to first spontaneous urine voiding (T <sub>uv</sub> ) | Time period from spinal injection ( $T_{sp}$ ; time 0 h) to the first time when the patient can pass urine unassisted |
| Time (h) to administration of rescue anaesthesia or rescue analgesia (T <sub>ra</sub> ) | Time from spinal injection( $T_{sp}$ ; time 0 h) to administration of first rescue anaesthesia or analgesia (if applicable) |
| Time (h) to first post-operative analgesia (T <sub>pa</sub> ) | Time from spinal injection $(T_{sp};$ time $0\ h)$ to first post-operative analgesia |

#### 11.3 Pharmacokinetic assessments

- Plasma concentrations of chloroprocaine at pre-dose and at 5, 10, 30 and 60 min after spinal injection for the three dose levels (D1, D2 and D3)
- Plasma concentrations of CABA at pre-dose and at 5, 10, 30 and 60 min after spinal injection for the three dose levels (D1, D2 and D3)
- Urinary excretion of CABA, as percentage of administered chloroprocaine dose for the three dose levels (D1, D2 and D3)

# 11.4 Safety assessments

Safety and general tolerability of the investigational anaesthetic will be based on TEAEs, TNS, physical examinations, vital signs and ECG.

In particular, ECG (if foreseen by the standard hospital procedures), blood pressure, heart rate and SpO<sub>2</sub> will be monitored as detailed in sections 7.1.1 and 7.1.2 of the study protocol (1).

Occurrence of clinically relevant hypotension or bradycardia will be monitored throughout the study and, if observed, treated according to the hospitals' standard procedures.

Patients will be questioned about the occurrence of treatment-emergent adverse events (TEAEs). Particular attention will be given to TNS symptoms. Further details on the AE assessments are given in section 7.1.4 of the study protocol (1).



#### 12 STATISTICAL METHODS

The data documented in this study and the parameters measured will be evaluated and compared using classic descriptive statistics, i.e. geometric mean (PK data only), arithmetic mean, SD, CV (%), minimum, median and maximum values for quantitative variables, and frequencies for qualitative variables.

Not available data will be evaluated as "missing values". The statistical analysis of demographic and safety data will be performed using SAS® version 9.3 (TS1M1) (4). The PK analysis will be performed using SAS® version 9.3 (TS1M1) (4) and the figures will be generated using Phoenix WinNonlin® version 6.3 (5).

#### 12.1 Analysis sets

### 12.1.1 Definitions

A subject will be defined as <u>screened</u> after the signature of the informed consent, regardless of the completion of all the screening procedures.

A subject will be defined as <u>eligible</u> if he/she respects all the inclusion/exclusion criteria. Otherwise he/she will be defined as a <u>screen failure</u>.

A subject will be defined as <u>enrolled</u> in the study if he/she is included into the treatment phase of the study. The enrolment will be performed through randomised allocation to a dose group.

A subject will be defined as <u>randomised</u> in the study when he/she is assigned to a randomised dose group.

- Enrolled set: all enrolled subjects. This analysis set will be used for demographic, baseline and background characteristics.
- Full Analysis Set (FAS): all randomised patients who fulfil the study protocol requirements in terms of study anaesthetics administration. Missing values of time to complete spinal block regression (T<sub>ea</sub>) will be replaced with the highest T<sub>ea</sub> detected in the corresponding treatment group. This analysis set will be used for sensitivity analysis.
- Per Protocol set (PP): all randomised patients who fulfil the study protocol requirements in terms of anaesthetic administration and primary efficacy evaluation, with no major deviations that could affect the primary efficacy results. This analysis set will be used for the primary efficacy analysis.
- PK Set 1 (PK 1): the PK set 1 will include all randomised patients who fulfil the study protocol requirements in terms of anaesthetic administration and have at least one post-dose blood PK sample collected.
- PK Set 2 (PK 2): the PK set 2 will include all randomised patients who fulfil the study protocol requirements in terms of anaesthetic administration and have the urine for PK analysis collected.



• Safety set: all patients who receive at least one dose of the investigational medicinal product. This analysis set will be used for the safety analyses.

Each subject will be coded by the CRO Biometry Unit as valid or not valid for the Enrolled set, FAS, PP set, PK set 1, PK set 2 and Safety set. Subjects will be evaluated according to the treatment they actually receive (Enrolled set, FAS, PP set, PK set 1, PK set 2 and Safety set).

#### 12.1.2 Reasons for exclusion from the Full Analysis Set

Reasons for the exclusion from the Full Analysis Set are the following:

- failure to be administered the investigational product
- lack of any primary efficacy data post enrolment
- failure to satisfy major inclusion/exclusion criteria (eligibility violations). Subjects who fail to satisfy an inclusion/exclusion criterion may be excluded from the analysis without the possibility of introducing bias only under the following circumstances:
  - the inclusion/exclusion criterion was measured prior to enrolment
  - the detection of the relevant eligibility violations can be made completely objectively
  - all subjects receive equal scrutiny for eligibility violations (blind review)
  - all detected violations of the particular inclusion/exclusion criterion are excluded

# 12.1.3 Reasons for exclusion from the Per Protocol set

Reasons for the exclusion from the Per Protocol set include the following:

- lack of compliance to the IMP
- exposure to an IMP different from the one assigned to the subject
- missing primary efficacy data
- more than 20% of the actual block assessment times outside the recommended ranges (see section 7.2 of the study protocol [1])
- failure to satisfy any inclusion/exclusion criteria (eligibility violations)

# 12.1.4 Reasons for exclusion from the PK sets

Reasons for the exclusion from the PK sets include the following:

- lack of compliance to the IMP
- exposure to an IMP different from the one assigned to the subject
- missing of any post-dose blood sample (PK set 1)
- missing of urine collection for PK analysis (PK set 2)
- failure to satisfy any inclusion/exclusion criteria (eligibility violations)



# 12.2 Sample size and power considerations

To calculate the required study sample size, results from a previous study with spinal injection of Chloroprocaine HCl 1% (6) were taken into consideration and normal distribution of data was assumed. Sample size was calculated using n-Query Advisor 7.0. When the sample size in each of the 3 dose groups is 13, a one-way analysis of variance will have 80% power to detect at the 0.050 level a difference in time to complete spinal block regression ( $T_{ea}$ ) means characterized by a variance of means,  $V=\Sigma(\mu i - \mu)^2 / G$  (where G=3) of 249.962, assuming that the common standard deviation is 30.011. To be more conservative and to take into account possible deviations from normality, the sample size is increased of about 15%. At least fifteen (15) patients per dose group have to be enrolled in order to have 15 administered patients per dose group.

# 12.3 Handling of missing data

# 12.3.1 Missing values of efficacy assessments

For the analysis on the Full Analysis Set, missing values of time to complete spinal block regression ( $T_{ea}$ ) will be replaced with the highest  $T_{ea}$  detected in the corresponding dose level group.

For the analysis on the Per Protocol Set and on the Full Analysis Set, any other missing values of the secondary efficacy assessments will not be replaced and will be treated as missing values.

# 12.3.2 Missing values of pharmacokinetic assessments

Missing values of the pharmacokinetic assessments will not be replaced and will be treated as missing data in the statistical analysis.

# 12.3.3 Missing values of safety assessments

Missing values of the safety assessments will not be replaced and will be treated as missing data in the statistical analysis.

# 12.4 Demographic, baseline and background characteristics

Continuous variables will be summarised by dose level group using classic descriptive statistics (i.e. mean, SD, CV%, min, median and max) and categorical variables will be summarised by dose level group using tables of frequencies.

# 12.4.1 Subjects' disposition

The disposition of all subjects enrolled in the study will be listed (Listing 16.2.4.1) and summarised by dose level and overall (Table 14.1.1.1). The number and proportion of subjects completing the study, the number and proportion of withdrawals and the reasons for withdrawal will be presented.



#### 12.4.2 Analysis sets

The subjects included in each analysis set will be listed (Listing 16.2.4.2) and summarised by dose level and overall (Table 14.1.1.2). Reason for exclusion will be listed.

# 12.4.3 Subjects excluded from the efficacy and/or PK and/or Safety analysis

All subjects excluded from the efficacy and/or PK and/or Safety analysis will be listed (Listing 16.2.3.1) and the reasons for exclusion will be reported.

#### 12.4.4 Inclusion/exclusion criteria not met

All the inclusion/exclusion criteria not met will be listed (Listing 16.2.4.4) and summarised by dose level and overall (Table 14.1.1.4) . The number and proportion of subjects for each criterion not met will be reported.

#### 12.4.5 Protocol deviations

All the protocol deviations reported during the clinical trial will be listed (Listing 16.2.2.1) and summarised by dose level and overall (Table 14.1.1.5). The number and proportion of subjects for each deviation will be reported.

#### 12.4.6 Discontinued subjects

All subjects who discontinued the clinical trial (if any) will be listed (Listing 16.2.1.1). The dose level of IMP administered, sex, age, last visit performed before discontinuation, time elapsed from IMP spinal injection (days), date of premature discontinuation and primary reason for subject premature discontinuation will be reported.

#### 12.4.7 Demography

Demographic data will be listed (Listing 16.2.4.3) and summarised by dose level and overall (Table 14.1.1.3). The number and proportion of subjects in each category for categorical variables (e.g. race) and descriptive statistics (mean, SD, CV%, minimum, median and maximum) for continous variables (e.g. age, weight) will be presented.

# 12.4.8 Medical and surgical history

All the diseases of medical history and the surgeries of all subjects enrolled in the study will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 18.1, listed (Listing 16.2.10.2) and summarised (Table 14.1.1.6). The number and proportion of subjects for each System Organ Class (SOC) and Preferred Term (PT) will be presented.

# 12.4.9 Physical examination

Date of the physical examination, ASA physical status, overall investigator's interpretation (as normal [N], abnormal not clinically significant [NCS] or abnormal clinically significant [CS]) and CS findings/illnesses (if any) will be listed (Listing 16.2.10.2).



#### 12.4.10 Prior and concomitant medications

Prior and concomitant medications/therapies will be listed (Listing 16.2.10.3) and summarised (Table 14.1.1.7) as number and proportion of subjects being treated with any type of medication/therapy classified according to the standardised product name recorded in the World Health Organization (WHO) Drug Dictionary Enhanced (WHODDE version September 1, 2015) and to the Anatomical Therapeutic Chemical (ATC) classification system.

#### 12.4.11 Subjects study visits

The dates of all subjects study visits will be listed (Listing 16.2.10.4).

# 12.4.12 Pregnancy test

The date/time of urine collection for pregnancy test and the test' result will be listed (Listing 16.2.10.5).

# 12.5 Analysis of efficacy parameters

Continuous variables will be summarised by dose level group using classic descriptive statistics (i.e. mean, SD, CV%, min, median and max) and categorical variables will be summarised by dose level group using tables of frequencies.

### 12.5.1 Surgical procedure

The type of surgery, the required metameric level of sensory block, the date/time of surgery start and end, the intake of any rescue anaesthesia or rescue analgesia administered before or during the surgical procedure and whether or not a general anaesthesia was required to complete surgery will be listed (Listing 16.2.6.1).

# 12.5.2 Sensory and motor block assessment

The scheduled assessment time, the assessment date and time, the metameric level of sensory block and the Bromage score will be listed (Listing 16.2.6.2).

# 12.5.3 Time to events and maximum level of sensory block

The time to regression of spinal block ( $T_{ea}$ ), time to onset of sensory block ( $T_{sb}$ ), time to onset of motor block ( $T_{mb}$ ), time to readiness for surgery ( $T_{rs}$ ), time to regression of sensory block to S1 ( $T_{S1}$ ), time to regression of motor block ( $T_{rmb}$ ), time to unassisted ambulation ( $T_{ua}$ ), time to maximum level of sensory block ( $T_{SBmax}$ ), time to regression of two dermatomers with respect to the maximum level of sensory block ( $T_{rd}$ ), time to eligibility for home discharge ( $T_{hd}$ ), time to first spontaneous urine voiding ( $T_{uv}$ ), time to administration of rescue anaesthesia or rescue analgesia ( $T_{ra}$ ) and time to first post-operative analgesia ( $T_{pa}$ ) will be listed (Listing 16.2.6.3) and will be summarised by dose level group and overall using descriptive statistics ( $T_{ra}$ ) and  $T_{ra}$ 



The maximum level of sensory block ( $SB_{max}$ ) will be listed (Listing 16.2.6.3) and will be summarised by dose level group and overall using tables of frequency (Table 14.2.1.3, Table 14.2.1.4).

Due to the small sample size, collected data will be compared using nonparametric tests.  $T_{ea}$ ,  $T_{sb}$ ,  $T_{mb}$ ,  $T_{rs}$ ,  $T_{S1}$ ,  $T_{rmb}$ ,  $T_{ua}$ ,  $SB_{max}$ ,  $T_{SBmax}$ ,  $T_{rd}$ ,  $T_{hd}$ ,  $T_{uv}$ ,  $T_{ra}$  and  $T_{pa}$  will be analysed using the Kruskal-Wallis test. Pairwise comparisons between dose level groups will be performed using the Wilcoxon rank-sum test (Table 14.2.2.1, Table 14.2.2.2, Table 14.2.2.3, Table 14.2.2.4). Comparisons will be performed according to the following hierarchical order:

- 1. Overall comparison
- 2. D1 (30 mg) vs. D3 (50 mg) comparison
- 3. D2 (40 mg) vs. D3 (50 mg) comparison
- 4. D1 (30 mg) vs. D2 (40 mg) comparison

Due to the hierarchical testing procedure, no formal adjustment of the alpha level is necessary (7). However, if a null hypothesis of a comparison cannot be rejected, all the null hypotheses of the subsequent comparisons cannot be rejected.

# 12.5.4 Effectiveness of anaesthesia and quality of spinal block

The date and time of assessment and the evaluations of effectiveness of anaesthesia and quality of spinal block will be listed (Listing 16.2.6.4) and will be summarised by dose level group and overall using tables of frequencies (Table 14.2.1.5, Table 14.2.1.6, Table 14.2.1.7, Table 14.2.1.8).

# 12.6 Analysis of pharmacokinetic parameters

The date and time of blood samples collection, the plasma concentrations of chloroprocaine and CABA, the date and time of urine sample collection and the urinary excretion of CABA will be listed (Listing 16.2.5.3, Listing 16.2.5.4).

A descriptive PK will be presented. The results will be displayed and summarised in tables (Table 14.2.3.1, Table 14.2.3.2) and figures (Figure 16.2.5.j, Figure 14.2.3.1, Figure 14.2.3.2). Individual and mean curves (+SD at sampling times), indicating inter-subject variability, will be plotted. Data below the lower quantification limit (BLQL) will be considered as 0 in the calculations and presented as BLQL in listings and tables. As a consequence of BLQL (i.e. 0) values, calculated geometric means (if requested) could be null. For this reason, in the presence of any null value, the geometric mean will be reported as not calculated (NC). PK analysis will be performed using SAS® version 9.3 (TS1M1) (4) and the figures will be generated using Phoenix WinNonlin® version 6.3 (5).

Urinary excretion of CABA will be calculated as the amount of metabolite excreted as a percentage of the administered dose (molar ratio).



#### 12.7 Safety and tolerability evaluation

Continuous variables will be summarised by dose level group using classic descriptive statistics (i.e. mean, SD, CV%, min, median and max) and categorical variables will be summarised by dose level group using tables of frequencies.

#### 12.7.1 Adverse events

A summary of AE definition, classification and management is reported in the section 11 of the study protocol (1).

Adverse events (AEs) will be coded by System Organ Class (SOC) and Preferred Term (PT), using the Medical Dictionary for Regulatory Activities (MedDRA) version 18.1.

AEs will be classified as pre-treatment AEs (PTAEs) and TEAEs according to the period of their occurrence, as follows:

- PTAEs: all AEs occurring before the IMP spinal injection and not worsening after the IMP spinal injection
- TEAEs: all AEs occurring or worsening after the IMP spinal injection

Individual TEAEs and PTAEs will be listed in two different subject data listings (Listing 16.2.7.1, Listing 16.2.7.2).

No summary table will be provided for PTAEs.

TEAEs will be summarised by dose level group and overall using frequency tables. The number and proportion of subjects with any TEAE, the number of TEAEs, the number and proportion of subjects with any TEAE by severity, the number of TEAEs by severity, the number and proportion of subjects with any TEAE related to the IMP, the number of TEAEs related to the IMP will be presented (Table 14.3.1.1, Table 14.3.1.2, Table 14.3.1.3, Table 14.3.1.4).

Should any serious TEAE occur, serious TEAEs will be summarised using frequency tables. The number and proportion of subjects with any serious TEAE, the number of serious TEAEs, the number and proportion of subjects with any serious TEAE related to the IMP and the number of serious TEAEs related to the IMP would be presented (Table 14.3.1.5, Table 14.3.1.6).

Additionally, all TEAEs leading to death, serious TEAEs and TEAEs leading to discontinuation will be listed separately, if applicable (Table 14.3.2.1).

#### 12.7.2 Vital signs

For screening, baseline and discharge (i.e. final/early termination visit) assessments of haemodynamic variables and for any other assessment judged clinical significant, the date and time of vital signs assessment and the values of Systolic Blood Pressure, Diastolic Blood Pressure, Heart Rate and Oxygen Saturation will be listed (Listing 16.2.9.1).



Screening, baseline and discharge (i.e. final/early termination visit) values of Systolic Blood Pressure, Diastolic Blood Pressure, Heart Rate and Oxygen Saturation will be summarised by dose level group and overall using descriptive statistics (Table 14.3.5.1).

#### 12.7.3 ECG

For any ECG assessment judged clinical significant, the date and time of ECG recording, overall investigator's interpretation (as normal, abnormal not clinically significant [NCS] or abnormal clinically significant [CS]) and the values Heart Rate, PR Interval, QRS Duration and QT Interval parameters will be listed (Listing 16.2.9.2).

#### 12.7.4 Pain assessment at the site of injection and at the site of surgery

Pain assessment at the site of injection and at the site of surgery immediately after regression of spinal block, at discharge (final visit/ETV), 24 h (day 2) and 6±1 days (day 7±1) after spinal injection will be listed (Listing 16.2.9.3) and will be summarised by dose level group and overall using frequency tables (Table 14.3.5.2).

# 12.7.5 Incidence of TNS at 24 h (day 2) and 6 days $\pm 1$ (day 7 $\pm 1$ ) after spinal injection $(T_{sp})$

The incidence of TNS at 24 h (day 2) and  $6\pm1$  days (day  $7\pm1$ ) after spinal injection ( $T_{sp}$ ) will be listed (Listing 16.2.9.4) and will be summarised by dose level group and overall using tables of frequency (Table 14.3.5.3).

# 12.7.6 Modified Aldrete's scoring scale

The assessments of the modified Aldrete's scoring scale will be listed (Listing 16.2.9.5).

# 12.7.7 Spinal injection

The date/time of spinal injection, the anatomical location of spinal injection, the identifier of the kit used and whether or not the planned volume was administered as per protocol will be listed (Listing 16.2.5.1).

# 12.7.8 Sedation and premedication

The administration of i.v. midazolam, the date and time of injection and the injected dose (if applicable), the administration of Ringer's solution, the date and time of infusion start and end and the infused volume (if applicable) will be listed (Listing 16.2.5.2).



#### 13 REFERENCES

- 1. Study Protocol CRO-14-122 / CHL.1/02-2014. Spinal anaesthesia with Chloroprocaine HCl 1% for elective lower limb procedures of short duration: a prospective, randomised, observer-blind study in adult patients. Final version 2.0, 28JAN2015
- 2. Study Protocol CRO-14-122 / CHL.1/02-2014. Spinal anaesthesia with Chloroprocaine HCl 1% for elective lower limb procedures of short duration: a prospective, randomised, observer-blind study in adult patients. Amendment Nr. 3, Final version 1.0, 03NOV2015
- 3. U.S. Department of Health and Human Services and U.S. Department of Agriculture, Nutrition and your health: Dietary Guidelines for Americans, 2010
- 4. SAS/STAT® 9.3 User's Guide
- 5. WinNonlin® Getting Started Guide, Pharsight Corporation
- 6. Casati A, Danelli G, Berti M, Fioro A, Fanelli A, Benassi C, Petronella G, Fanelli G. Intrathecal 2-chloroprocaine for lower limb outpatient surgery: a prospective, randomized, double-blind, clinical evaluation. Anesth Analg. 2006 Jul;103(1):234-8, table of contents
- 7. EMA CPMP/EWP/908/99 guideline "Points to consider on multiplicity issues in clinical trials", 19 September 2002




Statistical analysis plan CRO-14-122 Sponsor code CHL.1/02-2014 Chloroprocaine 1% - Spinal block Final version 1.0, 02FEB2016

# 14 APPENDICES

Appendix 1. Section 14 - Tables and Figures Shells

Appendix 2. Section 16.2 - Individual Subject Data Listings and Figures Shells



#### Section 14 - Tables and Figures Shells

- Table 14.1.1.1 Subjects' disposition (Enrolled set)
- Table 14.1.1.2 Analysis sets (Enrolled set)
- Table 14.1.1.3 Demography (Enrolled set, Safety set, Full analysis set and Per protocol set)
- Table 14.1.1.4 Inclusion/Exclusion criteria not met (Enrolled set)
- Table 14.1.1.5 Protocol deviations (Enrolled set, Full analysis set and Per protocol set)
- Table 14.1.1.6 Medical and surgical history (Safety set)
- Table 14.1.1.7 Prior and concomitant medications (Safety set)
- Table 14.2.1.1 Time to events (Per protocol set)
- Table 14.2.1.2 Time to events (Full analysis set)
- Table 14.2.1.3 Maximum level of sensory block (Per protocol set)
- Table 14.2.1.4 Maximum level of sensory block (Full analysis set)
- Table 14.2.1.5 Effectiveness of anaesthesia (Per protocol set)
- Table 14.2.1.6 Effectiveness of anaesthesia (Full analysis set)
- Table 14.2.1.7 Quality of spinal block (Per protocol set)
- Table 14.2.1.8 Quality of spinal block (Full analysis set)
- Table 14.2.2.1 Comparison of time to events (Per protocol set)
- Table 14.2.2.2 Comparison of time to events (Full analysis set)
- Table 14.2.2.3 Comparison of maximum level of sensory block (Per protocol set)
- Table 14.2.2.4 Comparison of maximum level of sensory block (Full analysis set)
- Table 14.2.3.1 Plasma concentrations (PK set 1)
- Table 14.2.3.2 Urinary concentration and excretion (PK set 2)
- Table 14.3.1.1 Global incidence of treatment emergent adverse events (Safety set)
- Table 14.3.1.2 Subjects with treatment emergent adverse events by system organ class and preferred term (Safety set)
- Table 14.3.1.3 Subjects with treatment emergent adverse events by system organ class, preferred term and severity (Safety set)
- Table 14.3.1.4 Subjects with treatment emergent adverse events related to the IMP by system organ class and preferred term (Safety set)
- Table 14.3.1.5 Subjects with serious treatment emergent adverse events by system organ class and preferred term (Safety set)
- Table 14.3.1.6 Subjects with serious treatment emergent adverse events related to the IMP by system organ class and preferred term (Safety set)
- Table 14.3.2.1 Treatment emergent adverse events leading to death, serious or leading to discontinuation (Safety set)
- Table 14.3.5.1 Vital signs (Safety set)
- Table 14.3.5.2 Pain assessment at the site of injection and at the site of surgery (Safety set)

CROSS Metrics S.A.


Statistical analysis plan CRO-14-122 Sponsor code CHL.1/02-2014 Chloroprocaine 1% - Spinal block Final version 1.0, 02FEB2016

# CROSS ALLIANCE Contract Research Organisation for Scientific Services

# Section 14 - Tables and Figures Shells

Table 14.3.5.3 - Transient neurological symptoms (Safety set)

Figure 14.2.3.1 - Mean plasma concentration curves of Chloroprocaine (PK set 1)

Figure 14.2.3.2 - Mean plasma concentration curves of CABA (PK set 1)

CROSS Metrics S.A.



#### Table 14.1.1.1 - Subjects' disposition (Enrolled set)

# Chloroprocaine 1% 40 mg 50 mg Overall

**Enrolled Set** 

| | 30 mg<br>N=XX<br>n (%) | 40 mg<br>N=XX<br>n (%) | 50 mg<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
|---|---|---|---|---|
| Randomised | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Discontinued before treatment | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Treated | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Completed | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Discontinued | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Reason A<br>Reason B | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) |
| | ••• | ••• | ••• | ••• |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the enrolled set

Source: Listing 16.2.4.1 - Subjects' disposition

Program: Tables\c122-ds-tbl.sas



#### **Table 14.1.1.2 - Analysis sets (Enrolled set)**

# Enrolled Set Chloroprocaine 1%

| | Chloroprocaine 1% | | | |
|---|---|---|---|---|
| | 30 mg<br>N=XX<br>n (%) | 40 mg<br>N=XX<br>n (%) | 50 mg<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
| Safety Set | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Full Analysis Set | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Per Protocol Set | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| PK Set 1 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| PK Set 2 | nn(xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the enrolled set

Source: Listing 16.2.4.2 - Analysis sets

Program: Tables\c122-ds-tbl.sas


Table 14.1.1.3 - Demography (Enrolled set, Safety set, Full analysis set and Per protocol set)

## Enrolled Set

| | | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|---|
| | | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Sex | Female | n (%) | nn (xx.x) | nn(xx.x) | nn (xx.x) | nn(xx.x) |
| | Male | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn(xx.x) |
| Race | American Indian or Alaska Native | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Asian | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Native Hawaiian or Other Pacific Islander | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Black or African American | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | White | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Other | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Age (years) | | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XX | XX | XX | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the enrolled set

Source: Listing 16.2.4.3 - Demography Program: Tables\c122-dm-tbl.sas



Table 14.1.1.3 - Demography (Enrolled set, Safety set, Full analysis set and Per protocol set)

## Enrolled Set

| | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|
| | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Height (cm) | N | nn | nn | nn | nn |
| | Mean | xxx.x | XXX.X | XXX.X | XXX.X |
| | SD | XX.X | XX.X | XX.X | xx.x |
| | CV% | XX.X | XX.X | XX.X | XX.X |
| | Min | XXX | XXX | XXX | XXX |
| | Median | XXX.X | XXX.X | xxx.x | XXX.X |
| | Max | xxx | XXX | XXX | xxx |
| Weight (kg) | N | nn | nn | nn | nn |
| | Mean | xx.xx | XX.XX | xx.xx | XX.XX |
| | SD | xx.xx | XX.XX | xx.xx | XX.XX |
| | CV% | xx.xx | xx.xx | xx.xx | xx.xx |
| | Min | XX.X | XX.X | XX.X | XX.X |
| | Median | xx.xx | xx.xx | xx.xx | XX.XX |
| | Max | XX.X | XX.X | XX.X | XX.X |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the enrolled set

Source: Listing 16.2.4.3 - Demography Program: Tables\c122-dm-tbl.sas



Table 14.1.1.3 - Demography (Enrolled set, Safety set, Full analysis set and Per protocol set)

## Enrolled Set

| | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|
| | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Body Mass Index (kg/m²) | N | nn | nn | nn | nn |
| | Mean | xx.xx | XX.XX | xx.xx | XX.XX |
| | SD | xx.xx | XX.XX | xx.xx | xx.xx |
| | CV% | XX.XX | XX.XX | XX.XX | XX.XX |
| | Min | XX.X | XX.X | XX.X | XX.X |
| | Median | xx.xx | XX.XX | XX.XX | xx.xx |
| | Max | XX.X | XX.X | XX.X | XX.X |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the enrolled set

Source: Listing 16.2.4.3 - Demography Program: Tables\c122-dm-tbl.sas



Table 14.1.1.3 - Demography (Enrolled set, Safety set, Full analysis set and Per protocol set)

Safety Set

| | | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|---|
| | | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| S | Famala | ·· (0/) | ( | () | () | |
| Sex | Female | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Male | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Race | American Indian or Alaska Native | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Asian | n (%) | nn (xx.x) | nn(xx.x) | nn(xx.x) | nn (xx.x) |
| | Native Hawaiian or Other Pacific Islander | n (%) | nn (xx.x) | nn(xx.x) | nn(xx.x) | nn (xx.x) |
| | Black or African American | n (%) | nn (xx.x) | nn (xx.x) | nn(xx.x) | nn (xx.x) |
| | White | n (%) | nn (xx.x) | nn(xx.x) | nn(xx.x) | nn (xx.x) |
| | Other | n (%) | nn (xx.x) | nn (xx.x) | nn(xx.x) | nn (xx.x) |
| Age (years) | | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | xx.x |
| | | SD | XX.X | XX.X | XX.X | xx.x |
| | | CV% | XX.X | XX.X | XX.X | xx.x |
| | | Min | XX | xx | xx | XX |
| | | Median | xx.x | XX.X | XX.X | xx.x |
| | | Max | XX | XX | XX | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the safety set

Source: Listing 16.2.4.3 - Demography Program: Tables\c122-dm-tbl.sas



Table 14.1.1.3 - Demography (Enrolled set, Safety set, Full analysis set and Per protocol set)

Safety Set

| | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|
| | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Height (cm) | N | nn | nn | nn | nn |
| | Mean | XXX.X | XXX.X | XXX.X | xxx.x |
| | SD | XX.X | XX.X | XX.X | XX.X |
| | CV% | xx.x | XX.X | XX.X | xx.x |
| | Min | XXX | XXX | XXX | xxx |
| | Median | XXX.X | xxx.x | XXX.X | xxx.x |
| | Max | xxx | XXX | XXX | xxx |
| Weight (kg) | N | nn | nn | nn | nn |
| | Mean | XX.XX | xx.xx | xx.xx | xx.xx |
| | SD | XX.XX | XX.XX | xx.xx | xx.xx |
| | CV% | XX.XX | xx.xx | xx.xx | xx.xx |
| | Min | xx.x | xx.x | XX.X | xx.x |
| | Median | xx.xx | XX.XX | xx.xx | xx.xx |
| | Max | XX.X | XX.X | XX.X | XX.X |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the safety set

Source: Listing 16.2.4.3 - Demography Program: Tables\c122-dm-tbl.sas



Table 14.1.1.3 - Demography (Enrolled set, Safety set, Full analysis set and Per protocol set)

## Safety Set

| | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|
| | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Body Mass Index (kg/m²) | N | nn | nn | nn | nn |
| | Mean | xx.xx | XX.XX | xx.xx | XX.XX |
| | SD | xx.xx | XX.XX | xx.xx | xx.xx |
| | CV% | xx.xx | XX.XX | xx.xx | XX.XX |
| | Min | XX.X | XX.X | XX.X | XX.X |
| | Median | xx.xx | XX.XX | xx.xx | XX.XX |
| | Max | XX.X | XX.X | XX.X | XX.X |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the safety set

Source: Listing 16.2.4.3 - Demography Program: Tables\c122-dm-tbl.sas



Table 14.1.1.3 - Demography (Enrolled set, Safety set, Full analysis set and Per protocol set)

#### Full Analysis Set Chloroprocaine 1%

| | | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|---|
| | | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Sex | Female | m (0/) | nn (222 22) | an (*** **) | an () | nn (vvv v) |
| Sex | | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Male | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Race | American Indian or Alaska Native | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Asian | n (%) | nn (xx.x) | nn (xx.x) | nn(xx.x) | nn(xx.x) |
| | Native Hawaiian or Other Pacific Islander | n (%) | nn (xx.x) | nn (xx.x) | nn(xx.x) | nn (xx.x) |
| | Black or African American | n (%) | nn (xx.x) | nn (xx.x) | nn(xx.x) | nn (xx.x) |
| | White | n (%) | nn (xx.x) | nn (xx.x) | nn(xx.x) | nn (xx.x) |
| | Other | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Age (years) | | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | XX.X |
| | | Min | XX | xx | xx | XX |
| | | Median | XX.X | XX.X | XX.X | XX.X |
| | | Max | XX | XX | XX | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the full analysis set

Source: Listing 16.2.4.3 - Demography Program: Tables\c122-dm-tbl.sas



Table 14.1.1.3 - Demography (Enrolled set, Safety set, Full analysis set and Per protocol set)

## Full Analysis Set

| | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|
| | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Height (cm) | N | nn | nn | nn | nn |
| | Mean | XXX.X | XXX.X | XXX.X | XXX.X |
| | SD | XX.X | XX.X | XX.X | XX.X |
| | CV% | XX.X | xx.x | XX.X | xx.x |
| | Min | XXX | xxx | XXX | xxx |
| | Median | XXX.X | xxx.x | xxx.x | xxx.x |
| | Max | XXX | XXX | xxx | xxx |
| Weight (kg) | N | nn | nn | nn | nn |
| | Mean | XX.XX | XX.XX | XX.XX | xx.xx |
| | SD | xx.xx | xx.xx | xx.xx | xx.xx |
| | CV% | xx.xx | xx.xx | xx.xx | xx.xx |
| | Min | xx.x | XX.X | xx.x | xx.x |
| | Median | XX.XX | XX.XX | XX.XX | xx.xx |
| | Max | XX.X | xx.x | XX.X | xx.x |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the full analysis set

Source: Listing 16.2.4.3 - Demography Program: Tables\c122-dm-tbl.sas



Table 14.1.1.3 - Demography (Enrolled set, Safety set, Full analysis set and Per protocol set)

# Full Analysis Set

| | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|
| | Statistics | 30 mg | 40 mg | 50 mg | Overall |
| | | N=XX | N=XX | N=XX | N=XX |
| Body Mass Index (kg/m²) | N | nn | nn | nn | nn |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | xx.xx | XX.XX | xx.xx | XX.XX |
| | CV% | XX.XX | XX.XX | XX.XX | xx.xx |
| | Min | XX.X | XX.X | XX.X | XX.X |
| | Median | xx.xx | XX.XX | xx.xx | xx.xx |
| | Max | xx.x | xx.x | XX.X | XX.X |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the full analysis set

Source: Listing 16.2.4.3 - Demography Program: Tables\c122-dm-tbl.sas



Table 14.1.1.3 - Demography (Enrolled set, Safety set, Full analysis set and Per protocol set)

#### Per Protocol Set Chloroprocaine 1%

| | | | | Chloropr | ocaine 1% | |
|---|---|---|---|---|---|---|
| | | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| G. | Percel | (0/) | | ( | ( | |
| Sex | Female | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Male | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Race | American Indian or Alaska Native | n (%) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Asian | n (%) | nn (xx.x) | nn(xx.x) | nn(xx.x) | nn(xx.x) |
| | Native Hawaiian or Other Pacific Islander | n (%) | nn (xx.x) | nn(xx.x) | nn(xx.x) | nn(xx.x) |
| | Black or African American | n (%) | nn (xx.x) | nn(xx.x) | nn(xx.x) | nn(xx.x) |
| | White | n (%) | nn (xx.x) | nn(xx.x) | nn(xx.x) | nn(xx.x) |
| | Other | n (%) | nn(xx.x) | nn(xx.x) | nn (xx.x) | nn (xx.x) |
| Age (years) | | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | xx.x |
| | | Min | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | xx.x |
| | | Max | XX | XX | XX | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Source: Listing 16.2.4.3 - Demography Program: Tables\c122-dm-tbl.sas



Table 14.1.1.3 - Demography (Enrolled set, Safety set, Full analysis set and Per protocol set)

## Per Protocol Set

| | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|
| | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Height (cm) | N | nn | nn | nn | nn |
| | Mean | xxx.x | XXX.X | XXX.X | XXX.X |
| | SD | XX.X | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X | XX.X |
| | Min | XXX | XXX | XXX | XXX |
| | Median | XXX.X | XXX.X | XXX.X | XXX.X |
| | Max | xxx | xxx | xxx | xxx |
| Waight (Isa) | N | nn | 22 | nn | nn |
| Weight (kg) | | nn | nn | nn | nn |
| | Mean | XX.XX | XX.XX | XX.XX | XX.XX |
| | SD | XX.XX | XX.XX | XX.XX | XX.XX |
| | CV% | XX.XX | xx.xx | XX.XX | XX.XX |
| | Min | XX.X | XX.X | XX.X | XX.X |
| | Median | xx.xx | xx.xx | xx.xx | XX.XX |
| | Max | xx.x | XX.X | XX.X | xx.x |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Source: Listing 16.2.4.3 - Demography Program: Tables\c122-dm-tbl.sas

XX.X



Statistical analysis plan CRO-14-122 Sponsor code CHL.1/02-2014 Chloroprocaine 1% - Spinal block Final version 1.0, 02FEB2016

Table 14.1.1.3 - Demography (Enrolled set, Safety set, Full analysis set and Per protocol set)

#### **Per Protocol Set** Chloroprocaine 1% 30 mg 40 mg 50 mg **Statistics Overall** N=XXN=XX N=XXN=XXBody Mass Index (kg/m<sup>2</sup>) N nn nn nn nn Mean XX.XX XX.XX XX.XXXX.XX SD XX.XX XX.XX XX.XX XX.XX CV% XX.XX XX.XX XX.XX XX.XX Min XX.X XX.X XX.X XX.X Median XX.XX XX.XX XX.XX XX.XX

XX.X

XX.X

XX.X

Max

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Source: Listing 16.2.4.3 - Demography Program: Tables\c122-dm-tbl.sas



#### **Table 14.1.1.4 - Inclusion/Exclusion criteria not met (Enrolled set)**

## Chloroprocaine 1% 40 mg 50 mg Overall N=XXN=XXN=XX

**Enrolled Set** 

| | n (%) | n (%) | n (%) | n (%) |
|---|---|---|---|---|
| Number of subjects who did not meet any inclusion/exclusion criterion | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criterion 1 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Inclusion criterion 2 | nn(xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criterion 1 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Exclusion criterion 2 | nn(xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | | | ••• |

30 mg

N=XX

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the enrolled set

Source: Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

Program: Tables\c122-ie-tbl.sas



Table 14.1.1.5 - Protocol deviations (Enrolled set, Full analysis set and Per protocol set)

#### **Enrolled Set** Chloroprocaine 1% 30 mg 40 mg 50 mg Overall N=XXN=XXN=XXN=XXn (%) n (%) n (%) n (%) Number of subjects with any protocol deviation nn (xx.x) nn (xx.x) nn (xx.x) nn (xx.x) Major nn (xx.x) nn (xx.x) nn (xx.x) nn (xx.x) Deviation Coded Term A nn(xx.x)nn(xx.x)nn(xx.x)nn (xx.x) Deviation Coded Term B nn (xx.x) nn(xx.x)nn(xx.x)nn (xx.x) ••• ••• Minor nn (xx.x) nn (xx.x) nn (xx.x) nn (xx.x) Deviation Coded Term C nn (xx.x) nn (xx.x) nn(xx.x)nn(xx.x)Deviation Coded Term D nn(xx.x)nn(xx.x)nn(xx.x)nn (xx.x)

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the enrolled set

Source: Listing 16.2.2.1 - Protocol deviations

 $Program: Tables \verb|\c122-dv-tbl.sas|$ 



Table 14.1.1.5 - Protocol deviations (Enrolled set, Full analysis set and Per protocol set)

#### Full Analysis Set Chloroprocaine 1%

| | Chloroprocaine 1% | | | |
|---|---|---|---|---|
| | 30 mg<br>N=XX<br>n (%) | 40 mg<br>N=XX<br>n (%) | 50 mg<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
| Number of subjects with any protocol deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Major | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation Coded Term A Deviation Coded Term B | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) |
| Minor | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation Coded Term C | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation Coded Term D | nn(xx.x) | nn (xx.x) | nn(xx.x) | nn (xx.x) |
| | | | ••• | ••• |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the full analysis set

Source: Listing 16.2.2.1 - Protocol deviations

Program: Tables\c122-dv-tbl.sas



Table 14.1.1.5 - Protocol deviations (Enrolled set, Full analysis set and Per protocol set)

# Per Protocol Set Chloroprocaine 1%

| | Chloroprocaine 1% | | | |
|---|---|---|---|---|
| | 30 mg<br>N=XX<br>n (%) | 40 mg<br>N=XX<br>n (%) | 50 mg<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
| Number of subjects with any protocol deviation | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Minor | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| Deviation Coded Term C Deviation Coded Term D | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) |
| | ••• | ••• | ••• | ••• |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Source: Listing 16.2.2.1 - Protocol deviations

Program: Tables\c122-dv-tbl.sas



#### Table 14.1.1.6 - Medical and surgical history (Safety set)

## Safety Set Chloroprocaine 1%

| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | 30 mg | 40 mg | 40 mg | Overall |
|---|---|---|---|---|
| | N=XX | N=XX | N=XX | N=XX |
| | n (%) [n MH/SH] | n (%) [n MH/SH] | n (%) [n MH/SH] | n (%) [n MH/SH] |
| Number of subjects with any disease or surgery | nn (xx.x) [nn] | nn (xx.x) [nn] | nn (xx.x) [nn] | nn (xx.x) [nn] |
| System Organ Class A | nn(xx.x)[nn] | nn (xx.x) [nn] | nn (xx.x) [nn] | nn(xx.x)[nn] |
| Preferred Term A | nn (xx.x) [nn] | nn (xx.x) [nn] | nn (xx.x) [nn] | nn (xx.x) [nn] |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the safety set

Note 1: MedDRA version 18.1

Source: Listing 16.2.10.1 - Medical and surgical history

Program: Tables\c122-mh-tbl.sas



#### Table 14.1.1.7 - Prior and concomitant medications (Safety set)

#### Safety Set Chloroprocaine 1%

| | Chioroprocaine 1% | | | |
|---|---|---|---|---|
| Prior or Concomitant ATC level 4 <sup>1</sup> Standardised name <sup>1</sup> | 30 mg<br>N=XX<br>n (%) [n CM] | 40 mg<br>N=XX<br>n (%) [n CM] | 50 mg<br>N=XX<br>n (%) [n CM] | Overall<br>N=XX<br>n (%) [n CM] |
| Number of patients with any prior or concomitant medication | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] | nn (xx.x) [nn] |
| Prior | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] |
| ATC level 4 Term A | nn(xx.x)[nn] | nn (xx.x) [nn] | nn(xx.x)[nn] | nn(xx.x)[nn] |
| Standardised name A Standardised name B | nn (xx.x) [nn]<br>nn (xx.x) [nn]<br> | nn (xx.x) [nn]<br>nn (xx.x) [nn]<br> | nn (xx.x) [nn]<br>nn (xx.x) [nn]<br> | nn (xx.x) [nn]<br>nn (xx.x) [nn]<br> |
| Concomitant | nn(xx.x)[nn] | nn (xx.x) [nn] | nn (xx.x) [nn] | nn(xx.x)[nn] |
| ATC level 4 Term A | nn(xx.x)[nn] | nn (xx.x) [nn] | nn(xx.x)[nn] | nn(xx.x)[nn] |
| Standardised name A Standardised name B | nn (xx.x) [nn]<br>nn (xx.x) [nn]<br> | nn (xx.x) [nn]<br>nn (xx.x) [nn]<br> | nn (xx.x) [nn]<br>nn (xx.x) [nn]<br> | nn (xx.x) [nn]<br>nn (xx.x) [nn]<br> |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the safety set

Note 1: WHODDE September 1, 2015

Source: Listing 16.2.10.3 - Prior and concomitant medications

Program: Tables\c122-cm-tbl.sas



#### **Table 14.2.1.1 - Time to events (Per protocol set)**

## Per Protocol Set Chloroprocaine 1%

| | Chloroprocaine 1% | | | |
|---|---|---|---|---|
| Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| N | nn | nn | nn | nn |
| Mean | XX.X | XX.X | XX.X | xx.x |
| SD | XX.X | XX.X | XX.X | xx.x |
| CV% | XX.X | xx.x | XX.X | xx.x |
| Min | XX | xx | XX | XX |
| Median | XX.X | xx.x | XX.X | xx.x |
| Max | XX | xx | xx | XX |
| N | nn | nn | nn | nn |
| Mean | XX.X | xx.x | XX.X | xx.x |
| SD | XX.X | xx.x | XX.X | xx.x |
| CV% | xx.x | xx.x | XX.X | XX.X |
| Min | XX | xx | XX | xx |
| Median | XX.X | xx.x | xx.x | xx.x |
| Max | XX | xx | XX | xx |
| | N Mean SD CV% Min Median Max N Mean SD CV% Min Mean Man SD CV% Min Median | N nn Mean xx.x SD xx.x CV% xx.x Min xx Median xx.x N nn Mean xx.x SD xx.x CV% xx.x Min xx Median xx.x Median xx.x | Statistics 30 mg N=XX 40 mg N=XX N nn nn Mean xx.x xx.x SD xx.x xx.x CV% xx.x xx.x Min xx xx.x Median xx.x xx.x N nn nn Mean xx.x xx.x SD xx.x xx.x CV% xx.x xx.x Min xx xx Median xx.x xx.x | Statistics 30 mg N=XX 40 mg N=XX 50 mg N=XX N nn nn nn Mean xx.x xx.x xx.x SD xx.x xx.x xx.x CV% xx.x xx.x xx.x Min xx xx.x xx.x Median xx.x xx.x xx.x N nn nn nn Mean xx.x xx.x xx.x SD xx.x xx.x xx.x CV% xx.x xx.x xx.x Min xx xx xx Median xx.x xx.x xx.x |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



#### **Table 14.2.1.1 - Time to events (Per protocol set)**

#### Per Protocol Set Chloroprocaine 1%

| | | Chioroprocaine 1% | | | |
|---|---|---|---|---|---|
| Time to | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Onset of Motor Block (min) | N | nn | nn | nn | nn |
| Onset of Motor Block (mm) | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X | XX.X |
| | CV% | XX.X | xx.x | XX.X | XX.X |
| | Min | XX | xx | xx | XX |
| | Median | XX.X | xx.x | XX.X | xx.x |
| | Max | XX | XX | XX | XX |
| D 1: 0 0 ( ; ) | N | | | | |
| Readiness for Surgery (min) | N | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | xx | XX |
| | Median | XX.X | xx.x | xx.x | xx.x |
| | Max | XX | xx | XX | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



**Table 14.2.1.1 - Time to events (Per protocol set)** 

#### Per Protocol Set Chloroprocaine 1%

| | Chioroprocaine 1% | | | | |
|---|---|---|---|---|---|
| Time to | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Regression of Sensory Block (h) | N | nn | nn | nn | nn |
| regression of sensory block (ii) | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X | XX.X |
| | CV% | XX.X | xx.x | XX.X | xx.x |
| | Min | XX | XX | xx | XX |
| | Median | xx.x | xx.x | xx.x | xx.x |
| | Max | XX | XX | XX | XX |
| Regression of Motor Block h) | N | nn | nn | nn | nn |
| Regression of Wotor Block II) | Mean | nn<br>xx.x | nn<br>xx.x | nn<br>xx.x | nn |
| | SD | XX.X | XX.X | XX.X | XX.X<br>XX.X |
| | CV% | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX |
| | Median | XX.X | XX.X | xx.x | xx.x |
| | Max | XX | xx | XX | xx |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



**Table 14.2.1.1 - Time to events (Per protocol set)** 

#### Per Protocol Set Chloroprocaine 1%

| | Chloroprocaine 1% | | | |
|---|---|---|---|---|
| Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| N | nn | nn | nn | nn |
| Mean | XX.X | xx.x | XX.X | xx.x |
| SD | XX.X | xx.x | XX.X | xx.x |
| CV% | XX.X | xx.x | XX.X | xx.x |
| Min | XX | xx | XX | xx |
| Median | XX.X | xx.x | XX.X | xx.x |
| Max | XX | xx | xx | xx |
| N | nn | nn | nn | nn |
| Mean | XX.X | xx.x | XX.X | xx.x |
| SD | XX.X | xx.x | XX.X | xx.x |
| CV% | xx.x | xx.x | XX.X | XX.X |
| Min | XX | xx | XX | XX |
| Median | XX.X | xx.x | XX.X | xx.x |
| Max | XX | xx | XX | XX |
| | N Mean SD CV% Min Median Max N Mean SD CV% Min Mean SD CV% Min Median | N=XX N nn Mean xx.x SD xx.x CV% xx.x Min xx Median xx.x N nn Mean xx.x SD xx.x CV% xx.x Min xx Median xx.x Median xx.x | Statistics 30 mg N=XX 40 mg N=XX N nn nn Mean xx.x xx.x SD xx.x xx.x CV% xx.x xx.x Min xx xx.x Median xx.x xx.x N nn nn Mean xx.x xx.x SD xx.x xx.x CV% xx.x xx.x Min xx xx Median xx.x xx.x | Statistics 30 mg N=XX 40 mg N=XX 50 mg N=XX N nn nn nn Mean xx.x xx.x xx.x SD xx.x xx.x xx.x CV% xx.x xx.x xx.x Min xx xx.x xx.x Median xx.x xx xx N nn nn nn Mean xx.x xx.x xx.x SD xx.x xx.x xx.x CV% xx.x xx.x xx.x Min xx xx xx Median xx.x xx.x xx.x |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



**Table 14.2.1.1 - Time to events (Per protocol set)** 

#### Per Protocol Set Chloroprocaine 1%

| | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|
| Time to | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Regression of Two Dermatomers (h) | N | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | xx.x | XX.X |
| | SD | XX.X | XX.X | xx.x | XX.X |
| | CV% | XX.X | XX.X | XX.X | xx.x |
| | Min | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | xx.x |
| | Max | XX | XX | XX | XX |
| Eligibility for Home Discharge (h) | N | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | xx.x | XX.X |
| | SD | XX.X | XX.X | XX.X | xx.x |
| | CV% | XX.X | XX.X | xx.x | xx.x |
| | Min | XX | xx | xx | XX |
| | Median | XX.X | XX.X | xx.x | XX.X |
| | Max | XX | xx | xx | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



#### **Table 14.2.1.1 - Time to events (Per protocol set)**

#### Per Protocol Set Chloroprocaine 1%

| | Chioroprocaine 1% | | | | |
|---|---|---|---|---|---|
| Time to | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| First Spontaneous Urine Voiding (h) | N | nn | nn | nn | nn |
| That openaneous erme volume (ii) | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X | XX.X |
| | CV% | XX.X | xx.x | xx.x | xx.x |
| | Min | XX | xx | XX | xx |
| | Median | XX.X | xx.x | xx.x | xx.x |
| | Max | XX | XX | xx | XX |
| Rescue Anaesthesia/Analgesia (h) | N | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Max | XX | XX | xx | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



#### **Table 14.2.1.1 - Time to events (Per protocol set)**

#### Per Protocol Set Chloroprocaine 1%

| | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|
| Time to | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| First Post-Operative Analgesia (h) | N | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | xx.x |
| | SD | XX.X | XX.X | XX.X | XX.X |
| | CV% | XX.X | XX.X | XX.X | xx.x |
| | Min | XX | xx | XX | XX |
| | Median | XX.X | xx.x | XX.X | xx.x |
| | Max | XX | XX | XX | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



## Table 14.2.1.2 - Time to events (Full analysis set)

#### Full Analysis Set Chloroprocaine 1%

| | | | Chloroprocaine 1% | | |
|---|---|---|---|---|---|
| Time to | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Regression of Spinal Block (h) | N | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | xx.x | XX.X |
| | SD | XX.X | XX.X | xx.x | XX.X |
| | CV% | XX.X | xx.x | xx.x | xx.x |
| | Min | XX | XX | XX | XX |
| | Median | XX.X | xx.x | xx.x | xx.x |
| | Max | XX | xx | xx | XX |
| Onset of Sensory Block (min) | N | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | xx.x | XX.X |
| | SD | XX.X | XX.X | xx.x | XX.X |
| | CV% | XX.X | xx.x | xx.x | xx.x |
| | Min | XX | XX | XX | XX |
| | Median | XX.X | xx.x | xx.x | XX.X |
| | Max | XX | xx | xx | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



## Table 14.2.1.2 - Time to events (Full analysis set)

#### Full Analysis Set Chloroprocaine 1%

| | | | Chloroprocaine 1% | | |
|---|---|---|---|---|---|
| Time to | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Onset of Motor Block (min) | N | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | xx.x | XX.X |
| | SD | XX.X | XX.X | xx.x | XX.X |
| | CV% | XX.X | XX.X | xx.x | XX.X |
| | Min | XX | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | XX.X |
| | Max | XX | XX | XX | XX |
| Readiness for Surgery (min) | N | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | xx.x | XX.X |
| | SD | XX.X | XX.X | xx.x | XX.X |
| | CV% | XX.X | XX.X | xx.x | xx.x |
| | Min | XX | XX | xx | XX |
| | Median | XX.X | xx.x | xx.x | XX.X |
| | Max | XX | xx | xx | xx |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



## Table 14.2.1.2 - Time to events (Full analysis set)

#### Full Analysis Set Chloroprocaine 1%

| | | | Chloroprocaine 1% | | |
|---|---|---|---|---|---|
| Time to | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Regression of Sensory Block (h) | N | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | xx.x |
| | SD | XX.X | XX.X | XX.X | xx.x |
| | CV% | XX.X | XX.X | XX.X | xx.x |
| | Min | XX | XX | xx | XX |
| | Median | XX.X | XX.X | XX.X | xx.x |
| | Max | XX | xx | xx | xx |
| Regression of Motor Block h) | N | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | xx.x |
| | SD | XX.X | XX.X | XX.X | xx.x |
| | CV% | XX.X | XX.X | xx.x | xx.x |
| | Min | XX | xx | xx | XX |
| | Median | XX.X | XX.X | xx.x | xx.x |
| | Max | XX | xx | xx | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



Table 14.2.1.2 - Time to events (Full analysis set)

#### Full Analysis Set Chloroprocaine 1%

| | Chloroprocaine 1% | | | |
|---|---|---|---|---|
| Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| N | nn | nn | nn | nn |
| Mean | XX.X | xx.x | XX.X | xx.x |
| SD | XX.X | xx.x | XX.X | xx.x |
| CV% | XX.X | xx.x | XX.X | xx.x |
| Min | XX | xx | XX | xx |
| Median | XX.X | xx.x | XX.X | xx.x |
| Max | XX | xx | xx | xx |
| N | nn | nn | nn | nn |
| Mean | XX.X | xx.x | XX.X | xx.x |
| SD | XX.X | xx.x | XX.X | xx.x |
| CV% | xx.x | xx.x | XX.X | XX.X |
| Min | XX | xx | XX | XX |
| Median | XX.X | xx.x | XX.X | xx.x |
| Max | XX | xx | xx | xx |
| | N Mean SD CV% Min Median Max N Mean SD CV% Min Mean SD CV% Min Median | N=XX N nn Mean xx.x SD xx.x CV% xx.x Min xx Median xx.x N nn Mean xx.x SD xx.x CV% xx.x Min xx Median xx.x Median xx.x | Statistics 30 mg N=XX 40 mg N=XX N nn nn Mean xx.x xx.x SD xx.x xx.x CV% xx.x xx.x Min xx xx.x Median xx.x xx.x N nn nn Mean xx.x xx.x SD xx.x xx.x CV% xx.x xx.x Min xx xx Median xx.x xx.x | Statistics 30 mg N=XX 40 mg N=XX 50 mg N=XX N nn nn nn Mean xx.x xx.x xx.x SD xx.x xx.x xx.x CV% xx.x xx.x xx.x Min xx xx.x xx.x Median xx.x xx xx N nn nn nn Mean xx.x xx.x xx.x SD xx.x xx.x xx.x CV% xx.x xx.x xx.x Min xx xx xx Median xx.x xx.x xx.x |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



#### Table 14.2.1.2 - Time to events (Full analysis set)

#### Full Analysis Set Chloroprocaine 1%

| Chioroprocaine 1% | | | | |
|---|---|---|---|---|
| Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| N | nn | nn | nn | nn |
| Mean | xx.x | XX.X | XX.X | XX.X |
| SD | XX.X | xx.x | XX.X | XX.X |
| CV% | XX.X | XX.X | XX.X | XX.X |
| Min | XX | XX | xx | XX |
| Median | XX.X | XX.X | xx.x | XX.X |
| Max | XX | XX | xx | xx |
| N | nn | nn | nn | nn |
| Mean | XX.X | XX.X | XX.X | XX.X |
| SD | XX.X | XX.X | XX.X | XX.X |
| CV% | XX.X | XX.X | xx.x | XX.X |
| Min | XX | XX | XX | XX |
| Median | XX.X | XX.X | XX.X | XX.X |
| Max | XX | XX | XX | xx |
| | N Mean SD CV% Min Median Max N Mean SD CV% Min Mean Man Man Modian | N=XX N nn Mean xx.x SD xx.x CV% xx.x Min xx Median xx.x N nn Mean xx.x SD xx.x CV% xx.x Min xx Median xx.x Median xx.x | Statistics 30 mg N=XX 40 mg N=XX N nn nn Mean xx.x xx.x SD xx.x xx.x CV% xx.x xx.x Min xx xx.x Median xx.x xx.x N nn nn Mean xx.x xx.x SD xx.x xx.x CV% xx.x xx.x Min xx xx Median xx.x xx.x | Statistics 30 mg N=XX 40 mg N=XX 50 mg N=XX N nn nn nn Mean xx.x xx.x xx.x SD xx.x xx.x xx.x CV% xx.x xx.x xx.x Min xx.x xx.x xx.x Median xx.x xx.x xx.x N nn nn nn Mean xx.x xx.x xx.x SD xx.x xx.x xx.x CV% xx.x xx.x xx.x Min xx xx xx Median xx.x xx.x xx.x |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



## Table 14.2.1.2 - Time to events (Full analysis set)

#### Full Analysis Set Chloroprocaine 1%

| | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|
| Time to | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| First Spontaneous Urine Voiding (h) | N | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | xx.x |
| | SD | XX.X | XX.X | XX.X | xx.x |
| | CV% | XX.X | XX.X | XX.X | XX.X |
| | Min | XX | xx | XX | XX |
| | Median | XX.X | XX.X | XX.X | xx.x |
| | Max | XX | xx | xx | XX |
| Rescue Anaesthesia/Analgesia (h) | N | nn | nn | nn | nn |
| | Mean | XX.X | XX.X | XX.X | xx.x |
| | SD | XX.X | XX.X | XX.X | xx.x |
| | CV% | XX.X | xx.x | xx.x | xx.x |
| | Min | XX | xx | xx | XX |
| | Median | XX.X | XX.X | xx.x | xx.x |
| | Max | XX | xx | xx | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



#### Table 14.2.1.2 - Time to events (Full analysis set)

#### Full Analysis Set Chloroprocaine 1%

| | | | Chioroprocaine 1% | | |
|---|---|---|---|---|---|
| Time to | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| First Post-Operative Analgesia (h) | N | nn | nn | nn | nn |
| | Mean | XX.X | xx.x | xx.x | xx.x |
| | SD | XX.X | xx.x | xx.x | xx.x |
| | CV% | XX.X | xx.x | XX.X | xx.x |
| | Min | XX | xx | XX | XX |
| | Median | XX.X | xx.x | XX.X | xx.x |
| | Max | XX | XX | XX | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



Table 14.2.1.3 - Maximum level of sensory block (Per protocol set)

#### **Per Protocol Set** Chloroprocaine 1% 40 mg Metameric 30 mg 50 mg **Overall** N=XXN=XXN=XXN=XXLevel n (%) n (%) n (%) n (%) Maximum Level of Sensory Block T1 nn (xx.x) nn (xx.x) nn (xx.x) nn (xx.x) T2 nn (xx.x) nn(xx.x)nn(xx.x)nn (xx.x) T3 nn (xx.x) nn (xx.x) nn (xx.x) nn (xx.x) T4 nn (xx.x) nn (xx.x) nn (xx.x) nn (xx.x) ...

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



#### Table 14.2.1.4 - Maximum level of sensory block (Full analysis set)

#### Full Analysis Set Chloroprocaine 1%

| | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|
| | Metameric<br>Level | 30 mg<br>N=XX<br>n (%) | 40 mg<br>N=XX<br>n (%) | 50 mg<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
| Maximum Level of Sensory Block | T1 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | T2 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Т3 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | T4 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | | ••• | ••• | ••• |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the full analysis set

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-01-tbl.sas



#### Table 14.2.1.5 - Effectiveness of anaesthesia (Per protocol set)

# Per Protocol Set Chloroprocaine 1% 40 mg 50 mg Overall N=XX N=XX N=XX n (%) n (%) n (%)

| | | 30 mg<br>N=XX<br>n (%) | 40 mg<br>N=XX<br>n (%) | 50 mg<br>N=XX<br>n (%) | N=XX<br>n (%) |
|---|---|---|---|---|---|
| Achievement of an Effective Anaesthesia | Y | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | N | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

20 ----

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Source: Listing 16.2.6.4 - Effectiveness of anaesthesia and quality of spinal block

Program: Tables\c122-qs-01-tbl.sas



#### Table 14.2.1.6 - Effectiveness of anaesthesia (Full analysis set)

## Full Analysis Set

| | | | Chloroprocaine 1% | | |
|---|---|---|---|---|---|
| | | 30 mg<br>N=XX<br>n (%) | 40 mg<br>N=XX<br>n (%) | 50 mg<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
| Achievement of an Effective Anaesthesia | Y | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | N | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the full analysis set

Source: Listing 16.2.6.4 - Effectiveness of anaesthesia and quality of spinal block

Program: Tables\c122-qs-01-tbl.sas


#### Table 14.2.1.7 - Quality of spinal block (Per protocol set)

# Per Protocol Set Chloroprocaine 1% 40 mg 50 mg Overall N=XX N=XX N=XX n (%) n (%) n (%)

| | | N=XX<br>n (%) | N=XX<br>n (%) | N=XX<br>n (%) | N=XX<br>n (%) |
|---|---|---|---|---|---|
| Quality of Spinal Block | Adequate Spinal Block | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Inadequate Spinal Block | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Failed Spinal Block | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

20 ----

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Source: Listing 16.2.6.4 - Effectiveness of anaesthesia and quality of spinal block

Program: Tables\c122-qs-01-tbl.sas



#### Table 14.2.1.8 - Quality of spinal block (Full analysis set)

# Full Analysis Set

| | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|
| | | 30 mg<br>N=XX<br>n (%) | 40 mg<br>N=XX<br>n (%) | 50 mg<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
| Quality of Spinal Block | Adequate Spinal Block | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Inadequate Spinal Block | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | Failed Spinal Block | nn (xx.x) | nn (xx.x) | nn(xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the full analysis set

Source: Listing 16.2.6.4 - Effectiveness of anaesthesia and quality of spinal block

Program: Tables\c122-qs-01-tbl.sas



**Table 14.2.2.1 - Comparison of time to events (Per protocol set)** 

| | | | Per Protocol Set | |
|---|---|---|---|---|
| Time to | Comparison | Test | Statistic | p-value <sup>1</sup> |
| Regression of Spinal Block (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| Onset of Sensory Block (min) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxxx |
| , | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX,X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| Onset of Motor Block (min) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxx |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | xxxx.x | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| Readiness for Surgery (min) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxx |
| Readilless for Surgery (IIIII) | | Wilcoxon Rank-Sum | | |
| | Chloroprocaine 1% 30 mg vs. 50 mg | | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |

Note: Subjects are analysed according to the dose level of the product they actually received

Note 1: p-values of Wilcoxon Rank-Sum test were calculated using t approximation

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-02-tbl.sas



**Table 14.2.2.1 - Comparison of time to events (Per protocol set)** 

| | | | Per Protocol Set | |
|---|---|---|---|---|
| Time to | Comparison | Test | Statistic | p-value <sup>1</sup> |
| Regression of Sensory Block (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| Regression of Motor Block h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxxx |
| , | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| Unassisted Ambulation (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| Maximum Level of Sensory Block (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | VVVV V | V VVVV |
| Maximum Level of Sensory Block (II) | | | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| <u></u> | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |

Note: Subjects are analysed according to the dose level of the product they actually received

Note 1: p-values of Wilcoxon Rank-Sum test were calculated using t approximation

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-02-tbl.sas



**Table 14.2.2.1 - Comparison of time to events (Per protocol set)** 

| | | | Per Protocol Set | |
|---|---|---|---|---|
| Time to | Comparison | Test | Statistic | p-value <sup>1</sup> |
| Regression of Two Dermatomers (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| Eligibility for Home Discharge (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxxx |
| <b>3</b> • <b>3</b> • | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| First Spontaneous Urine Voiding (h | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxx |
| 3( | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxx |
| Rescue Anaesthesia/Analgesia (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxx |
| Rescue I maesunesia I margesia (II) | Chloroprocaine 1% 30 mg vs. 50 mg Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | | |
| | | | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |

Note: Subjects are analysed according to the dose level of the product they actually received

Note 1: p-values of Wilcoxon Rank-Sum test were calculated using t approximation

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-02-tbl.sas



#### Table 14.2.2.1 - Comparison of time to events (Per protocol set)

| | | | Per Protocol Set | |
|---|---|---|---|---|
| Time to | Comparison | Test | Statistic | p-value <sup>1</sup> |
| First Post-Operative Analgesia (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |

Note: Subjects are analysed according to the dose level of the product they actually received

Note 1: p-values of Wilcoxon Rank-Sum test were calculated using t approximation

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-02-tbl.sas



Table 14.2.2.2 - Comparison of time to events (Full analysis set)

| | | Full Analysis Set | | |
|---|---|---|---|---|
| Time to | Comparison | Test | Statistic | p-value <sup>1</sup> |
| Regression of Spinal Block (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| Onset of Sensory Block (min) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| Onset of Motor Block (min) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| Readiness for Surgery (min) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |

Note: Subjects are analysed according to the dose level of the product they actually received

Note 1: p-values of Wilcoxon Rank-Sum test were calculated using t approximation

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-02-tbl.sas



Table 14.2.2.2 - Comparison of time to events (Full analysis set)

| | | | Full Analysis Set | |
|---|---|---|---|---|
| Time to | Comparison | Test | Statistic | p-value <sup>1</sup> |
| D : (C D) 1 (1) | CI 10/20 40 50 | 77 1 1 777 11 | | |
| Regression of Sensory Block (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| Regression of Motor Block h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | X.XXXX |
| Unassisted Ambulation (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | X.XXXX |
| Maximum Level of Sensory Block (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |

Note: Subjects are analysed according to the dose level of the product they actually received

Note 1: p-values of Wilcoxon Rank-Sum test were calculated using t approximation

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-02-tbl.sas



Table 14.2.2.2 - Comparison of time to events (Full analysis set)

| | | Full Analysis Set | | |
|---|---|---|---|---|
| Time to | Comparison | Test | Statistic | p-value <sup>1</sup> |
| Regression of Two Dermatomers (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| Eligibility for Home Discharge (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| First Spontaneous Urine Voiding (h | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| Rescue Anaesthesia/Analgesia (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | xxxx.x | x.xxxx |

Note: Subjects are analysed according to the dose level of the product they actually received

Note 1: p-values of Wilcoxon Rank-Sum test were calculated using t approximation

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-02-tbl.sas



#### Table 14.2.2.2 - Comparison of time to events (Full analysis set)

#### **Full Analysis Set**

| Time to | Comparison | Test | Statistic | p-value <sup>1</sup> |
|---|---|---|---|---|
| First Part Organization Application (b) | Chlanaura sina 10/20 mana 40 mana 50 ma | Variabel Wellia | | |
| First Post-Operative Analgesia (h) | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |

Note: Subjects are analysed according to the dose level of the product they actually received

Note 1: p-values of Wilcoxon Rank-Sum test were calculated using t approximation

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-02-tbl.sas



#### Table 14.2.2.3 - Comparison of maximum level of sensory block (Per protocol set)

| | Per Protocol Set | | | |
|---|---|---|---|---|
| | Comparison | Test | Statistic | p-value <sup>1</sup> |
| Maximum Level of Sensory Block | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | xxxx.x | x.xxxx |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | XXXX.X | x.xxxx |

Note: Subjects are analysed according to the dose level of the product they actually received

Note 1: p-values of Wilcoxon Rank-Sum test were calculated using t approximation

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-02-tbl.sas



#### Table 14.2.2.4 - Comparison of maximum level of sensory block (Full analysis set)

| | | | Full Analysis Set | |
|---|---|---|---|---|
| | Comparison | Test | Statistic | p-value <sup>1</sup> |
| Maximum Level of Sensory Block | Chloroprocaine 1% 30 mg vs. 40 mg vs. 50 mg | Kruskal-Wallis | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 40 mg vs. 50 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |
| | Chloroprocaine 1% 30 mg vs. 40 mg | Wilcoxon Rank-Sum | XXXX.X | X.XXXX |

Note: Subjects are analysed according to the dose level of the product they actually received

Note 1: p-values of Wilcoxon Rank-Sum test were calculated using t approximation

Source: Listing 16.2.6.3 - Time to events and maximum level of sensory block

Program: Tables\c122-qs-02-tbl.sas



#### Table 14.2.3.1 - Plasma concentrations (PK set 1)

PK Set 1

| | | Chloroprocaine 1% | | | | |
|---|---|---|---|---|---|---|
| | Time Point | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Chloroprocaine Plasma Concentration (ng/mL) | Pre-dose (0) | N | nn | nn | nn | nn |
| | | Geo.Mean | xx.x | XX.X | XX.X | XX.X |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | xx.x | XX.X | XX.X | XX.X |
| | | Min | XX | XX | XX | XX |
| | | Median | xx.x | XX.X | XX.X | XX.X |
| | | Max | XX | XX | XX | XX |
| Chloroprocaine Plasma Concentration (ng/mL) | 5 min after spinal injection | N | nn | nn | nn | nn |
| | | Geo.Mean | XX.X | XX.X | XX.X | XX.X |
| | | Mean | xx.x | XX.X | XX.X | XX.X |
| | | SD | xx.x | XX.X | XX.X | XX.X |
| | | CV% | xx.x | XX.X | XX.X | xx.x |
| | | Min | XX | XX | XX | XX |
| | | Median | xx.x | XX.X | XX.X | XX.X |
| | | Max | XX | XX | XX | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.5.3 - PK blood samples collection and plasma concentrations

Program: Tables\c122-pc-tbl.sas



#### Table 14.2.3.1 - Plasma concentrations (PK set 1)

PK Set 1

| | | Chloroprocaine 1% | | | | |
|---|---|---|---|---|---|---|
| | Time Point | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Chloroprocaine Plasma Concentration (ng/mL) | 10 min after spinal injection | N | nn | nn | nn | nn |
| | | Geo.Mean | XX.X | XX.X | XX.X | XX.X |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | xx.x |
| | | CV% | XX.X | xx.x | XX.X | xx.x |
| | | Min | XX | XX | xx | XX |
| | | Median | XX.X | XX.X | XX.X | xx.x |
| | | Max | XX | XX | XX | XX |
| Chloroprocaine Plasma Concentration (ng/mL) | 30 min after spinal injection | N | nn | nn | nn | nn |
| | | Geo.Mean | xx.x | XX.X | XX.X | xx.x |
| | | Mean | XX.X | xx.x | xx.x | xx.x |
| | | SD | xx.x | XX.X | XX.X | XX.X |
| | | CV% | xx.x | XX.X | XX.X | XX.X |
| | | Min | xx | XX | XX | XX |
| | | Median | xx.x | xx.x | xx.x | xx.x |
| | | Max | XX | XX | XX | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.5.3 - PK blood samples collection and plasma concentrations

Program: Tables\c122-pc-tbl.sas



#### Table 14.2.3.1 - Plasma concentrations (PK set 1)

PK Set 1

| | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|
| Time Point | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| 60 min after spinal injection | | nn | nn | nn | nn |
| | Geo.Mean | XX.X | XX.X | XX.X | XX.X |
| | Mean | XX.X | XX.X | XX.X | XX.X |
| | SD | XX.X | XX.X | XX.X | xx.x |
| | CV% | xx.x | xx.x | xx.x | xx.x |
| | Min | xx | XX | XX | XX |
| | Median | XX.X | XX.X | XX.X | xx.x |
| | Max | XX | XX | XX | XX |
| Pre-dose (0) | N | nn | nn | nn | nn |
| | Geo.Mean | XX.X | XX.X | XX.X | xx.x |
| | Mean | XX.X | xx.x | xx.x | XX.X |
| | SD | XX.X | xx.x | xx.x | XX.X |
| | CV% | XX.X | xx.x | xx.x | xx.x |
| | Min | xx | XX | XX | XX |
| | Median | XX.X | xx.x | xx.x | xx.x |
| | Max | xx | XX | XX | XX |
| | 60 min after spinal injection | 60 min after spinal injection N Geo.Mean Mean SD CV% Min Median Max Pre-dose (0) N Geo.Mean Mean SD CV% Min Mean SD CV% Min Mean Mean Mean Mean Mean Mean Mean Mea | N=XX | Time Point Statistics 30 mg N=XX 40 mg N=XX 60 min after spinal injection N nn nn Geo.Mean xx.x xx.x Mean xx.x xx.x SD xx.x xx.x Min xx xx Median xx.x xx.x Pre-dose (0) N nn nn Geo.Mean xx.x xx.x Mean xx.x xx.x SD xx.x xx.x CV% xx.x xx.x Min xx xx Median xx.x xx.x | Time Point Statistics 30 mg N=XX 40 mg N=XX 50 mg N=XX 60 min after spinal injection N nn nn nn Geo.Mean xx.x xx.x xx.x xx.x Mean xx.x xx.x xx.x xx.x CV% xx.x xx.x xx.x xx.x Min xx xx xx.x xx.x Pre-dose (0) N nn nn nn Pre-dose (0) N nn nn nn Geo.Mean xx.x xx.x xx.x Mean xx.x xx.x xx.x SD xx.x xx.x xx.x CV% xx.x xx.x xx.x CV% xx.x xx.x xx.x Min xx xx.x xx.x Median xx.x xx.x xx.x |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.5.3 - PK blood samples collection and plasma concentrations

Program: Tables\c122-pc-tbl.sas



#### Table 14.2.3.1 - Plasma concentrations (PK set 1)

PK Set 1

| | | Chloroprocaine 1% | | | | |
|---|---|---|---|---|---|---|
| | Time Point | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| CABA Plasma Concentration (ng/mL) | 5 min after spinal injection | N | nn | nn | nn | nn |
| | | Geo.Mean | XX.X | XX.X | XX.X | XX.X |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | xx.x | XX.X | xx.x |
| | | Min | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | xx.x |
| | | Max | XX | XX | XX | XX |
| CABA Plasma Concentration (ng/mL) | 10 min after spinal injection | N | nn | nn | nn | nn |
| | | Geo.Mean | XX.X | XX.X | XX.X | XX.X |
| | | Mean | xx.x | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | xx.x |
| | | Min | xx | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | xx.x |
| | | Max | XX | XX | XX | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.5.3 - PK blood samples collection and plasma concentrations

Program: Tables\c122-pc-tbl.sas



#### Table 14.2.3.1 - Plasma concentrations (PK set 1)

PK Set 1

| | | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|---|
| | Time Point | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| CABA Plasma Concentration (ng/mL) | 30 min after spinal injection | N | nn | nn | nn | nn |
| | | Geo.Mean | XX.X | XX.X | XX.X | XX.X |
| | | Mean | XX.X | XX.X | xx.x | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | xx.x |
| | | Min | xx | xx | XX | XX |
| | | Median | XX.X | XX.X | XX.X | xx.x |
| | | Max | XX | XX | XX | XX |
| CABA Plasma Concentration (ng/mL) | 60 min after spinal injection | N | nn | nn | nn | nn |
| | | Geo.Mean | XX.X | XX.X | XX.X | xx.x |
| | | Mean | XX.X | XX.X | XX.X | xx.x |
| | | SD | XX.X | XX.X | XX.X | xx.x |
| | | CV% | XX.X | XX.X | XX.X | xx.x |
| | | Min | xx | xx | xx | XX |
| | | Median | XX.X | XX.X | XX.X | xx.x |
| | | Max | XX | XX | XX | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.5.3 - PK blood samples collection and plasma concentrations

Program: Tables\c122-pc-tbl.sas



#### Table 14.2.3.2 - Urinary concentration and excretion (PK set 2)

PK Set 2

| | | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|---|
| | Time Point | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| CABA Urinary Concentration (ng/mL) | First Spontaneous Urine Voiding | N | nn | nn | nn | nn |
| | | Geo.Mean | XX.X | XX.X | XX.X | XX.X |
| | | Mean | XX.X | XX.X | xx.x | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | xx.x | XX.X | XX.X | XX.X |
| | | Min | XX | XX | XX | XX |
| | | Median | xx.x | XX.X | XX.X | XX.X |
| | | Max | XX | XX | xx | XX |
| CABA Urinary Excretion (%) | First Spontaneous Urine Voiding | N | nn | nn | nn | nn |
| | | Geo.Mean | xx.x | XX.X | XX.X | XX.X |
| | | Mean | xx.x | XX.X | XX.X | XX.X |
| | | SD | xx.x | XX.X | xx.x | XX.X |
| | | CV% | xx.x | XX.X | xx.x | XX.X |
| | | Min | xx | xx | xx | xx |
| | | Median | xx.x | XX.X | xx.x | XX.X |
| | | Max | XX | XX | XX | xx |

Note: Subjects are summarised according to the dose level of the product they actually received Source: Listing 16.2.5.4 - PK urine sample collection, urinary concentration and urinary excretion

Program: Tables\c122-pc-tbl.sas



Table 14.3.1.1 - Global incidence of treatment emergent adverse events (Safety set)

#### Safety Set Chloroprocaine 1%

| | | Chioropr | ocame 170 | |
|---|---|---|---|---|
| | 30 mg<br>N=XX<br>n (%) [n AE] | 40 mg<br>N=XX<br>n (%) [n AE] | 50 mg<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| Treatment Emergent Adverse Events | nn (xx.x) [nn] | nn (xx.x) [nn] | nn (xx.x) [nn] | nn (xx.x) [nn] |
| Related | nn(xx.x)[nn] | nn (xx.x) [nn] | nn(xx.x)[nn] | nn (xx.x) [nn] |
| Not related | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] |
| Mild | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] |
| Moderate | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] |
| Severe | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] |
| Leading to discontinuation | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] |
| Serious Treatment Emergent Adverse Events | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] | nn (xx.x) [nn] |
| Related | nn(xx.x)[nn] | nn (xx.x) [nn] | nn (xx.x) [nn] | nn (xx.x) [nn] |
| Not related | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] |
| Leading to discontinuation | nn(xx.x)[nn] | nn (xx.x) [nn] | nn (xx.x) [nn] | nn (xx.x) [nn] |
| Life-threatening | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] |
| Leading to death | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] | nn (xx.x) [nn] |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the safety set

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\c122-ae-01-tbl.sas



#### Table 14.3.1.2 - Subjects with treatment emergent adverse events by system organ class and preferred term (Safety set)

### Safety Set Chloroprocaine 1%

| | Chioroprocame 1/0 | | | |
|---|---|---|---|---|
| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | 30 mg<br>N=XX<br>n (%) [n AE] | 40 mg<br>N=XX<br>n (%) [n AE] | 50 mg<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| Treatment Emergent Adverse Events | $\operatorname{nn}(xx.x)[\operatorname{nn}]$ | nn (xx.x) [nn] | nn (xx.x) [nn] | nn (xx.x) [nn] |
| Injury, poisoning and procedural complications | nn(xx.x)[nn] | nn(xx.x)[nn] | nn (xx.x) [nn] | nn (xx.x) [nn] |
| Procedural pain Injection site pain | nn (xx.x) [nn]<br>nn (xx.x) [nn] | nn (xx.x) [nn]<br>nn (xx.x) [nn] | nn (xx.x) [nn]<br>nn (xx.x) [nn] | nn (xx.x) [nn]<br>nn (xx.x) [nn] |
| | | ••• | | |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the safety set

Note 1: MedDRA version 18.1

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\c122-ae-02-tbl.sas



Table 14.3.1.3 - Subjects with treatment emergent adverse events by system organ class, preferred term and severity (Safety set)

#### Safety Set Chloroprocaine 1%

| | | | | | | Cinoropi | ocume 1 /0 | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 30 mg<br>N=XX | | | 40 mg<br>N=XX | | | 50 mg<br>N=XX | | | Overall<br>N=XX | |
| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | Mild | Moderate | Severe | Mild | Moderate | Severe | Mild | Moderate | Severe | Mild | Moderate | Severe |
| | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) | n (%) |
| | [n AE] | [n AE] | [n AE] | [n AE] | [n AE] | [n AE] | [n AE] | [n AE] | [n AE] | [n AE] | [n AE] | [n AE] |
| Treatment Emergent Adverse Events | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] |
| Injury, poisoning and procedural complications | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] |
| Procedural pain | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] |
| Injection site pain | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] | [nn] |
| | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• | ••• |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the safety set

Note 1: MedDRA version 18.1

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\c122-ae-02-tbl.sas



Table 14.3.1.4 - Subjects with treatment emergent adverse events related to the IMP by system organ class and preferred term (Safety set)

Safety Set Chloroprocaine 1%

| | Chioroprocame 1 76 | | | |
|---|---|---|---|---|
| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | 30 mg<br>N=XX<br>n (%) [n AE] | 40 mg<br>N=XX<br>n (%) [n AE] | 50 mg<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| Treatment Emergent Adverse Events related to study IMP | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] | nn (xx.x) [nn] |
| Injury, poisoning and procedural complications | nn(xx.x)[nn] | nn(xx.x)[nn] | nn (xx.x) [nn] | nn(xx.x)[nn] |
| Procedural pain Injection site pain | nn (xx.x) [nn]<br>nn (xx.x) [nn] | nn (xx.x) [nn]<br>nn (xx.x) [nn] | nn (xx.x) [nn]<br>nn (xx.x) [nn] | nn (xx.x) [nn]<br>nn (xx.x) [nn] |
| <del></del> | | | | |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the safety set

Note 1: MedDRA version 18.1

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\c122-ae-02-tbl.sas



Table 14.3.1.5 - Subjects with serious treatment emergent adverse events by system organ class and preferred term (Safety set)

Safety Set Chloroprocaine 1%

| Chloroprocaine 1% | | | |
|---|---|---|---|
| 30 mg<br>N=XX<br>n (%) [n AE] | 40 mg<br>N=XX<br>n (%) [n AE] | 50 mg<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] | nn (xx.x) [nn] |
| nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] | nn(xx.x)[nn] |
| nn (xx.x) [nn]<br>nn (xx.x) [nn]<br> | nn (xx.x) [nn]<br>nn (xx.x) [nn]<br> | nn (xx.x) [nn]<br>nn (xx.x) [nn]<br> | nn (xx.x) [nn]<br>nn (xx.x) [nn]<br> |
| | N=XX<br>n (%) [n AE]<br>nn (xx.x) [nn]<br>nn (xx.x) [nn]<br>nn (xx.x) [nn]<br>nn (xx.x) [nn] | 30 mg | N=XX<br>n (%) [n AE] N=XX<br>n (%) [n AE] N=XX<br>n (%) [n AE] nn (xx.x) [nn] nn (xx.x) [nn] nn (xx.x) [nn] nn (xx.x) [nn] nn (xx.x) [nn] nn (xx.x) [nn] nn (xx.x) [nn] nn (xx.x) [nn] nn (xx.x) [nn] nn (xx.x) [nn] nn (xx.x) [nn] nn (xx.x) [nn] |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the safety set

Note 1: MedDRA version 18.1

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\c122-ae-02-tbl.sas



Table 14.3.1.6 - Subjects with serious treatment emergent adverse events related to the IMP by system organ class and preferred term (Safety set)

#### Safety Set Chloroprocaine 1%

| | Chioroprocame 178 | | | |
|---|---|---|---|---|
| System Organ Class <sup>1</sup> Preferred Term <sup>1</sup> | 30 mg<br>N=XX<br>n (%) [n AE] | 40 mg<br>N=XX<br>n (%) [n AE] | 50 mg<br>N=XX<br>n (%) [n AE] | Overall<br>N=XX<br>n (%) [n AE] |
| Serious Treatment Emergent Adverse Events related to study IMP | nn (xx.x) [nn] | nn (xx.x) [nn] | nn (xx.x) [nn] | nn (xx.x) [nn] |
| Injury, poisoning and procedural complications | nn(xx.x)[nn] | nn (xx.x) [nn] | nn (xx.x) [nn] | nn(xx.x)[nn] |
| Procedural pain Injection site pain | nn (xx.x) [nn]<br>nn (xx.x) [nn] | nn (xx.x) [nn]<br>nn (xx.x) [nn] | nn (xx.x) [nn]<br>nn (xx.x) [nn] | nn (xx.x) [nn]<br>nn (xx.x) [nn] |
| | | ••• | ••• | ••• |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the safety set

Note 1: MedDRA version 18.1

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

 $Program: Tables \verb|\c122-ae-02-tbl.sas|$ 



#### Table 14.3.2.1 - Treatment emergent adverse events leading to death, serious or leading to discontinuation (Safety set)

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | AE<br>Nr<br>/<br>FU<br>Nr | Verbatim /<br>Preferred Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> | Start or Follow-up Date/time / Start or Follow-up Day / End Date/time / End Day / Duration | IMP injection Date/time / Day / Time from IMP injection | Seriousness /<br>Severity /<br>Related to IMP /<br>Other relationship | Outcome / Action taken with IMP / Other action taken | Therapy required / Leading to discontinuation / Comments |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | 1 | Headache /<br>Headache /<br>Nervous system disorders | ddMMMyyyy hh:mm / Day j / Ongoing / / | ddMMMyyyy hh:mm /<br>Day j /<br>xx h xx min | Y /<br>Moderate /<br>Not related /<br>Weather condition | Recovering/resolving / Not applicable / | Y /<br>N /<br> |
| Skkk/ppp | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: MedDRA version 18.1

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\c122-ae-03-tbl.sas



#### Table 14.3.2.1 - Treatment emergent adverse events leading to death, serious or leading to discontinuation (Safety set)

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | AE<br>Nr<br>/<br>FU<br>Nr | Verbatim /<br>Preferred Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> | Start or Follow-up Date/time / Start or Follow-up Day / End Date/time / End Day / Duration | IMP injection Date/time / Day / Time from IMP injection | Seriousness /<br>Severity /<br>Related to IMP /<br>Other relationship | Outcome / Action taken with IMP / Other action taken | Therapy required / Leading to discontinuation / Comments |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | 1 | Headache /<br>Headache /<br>Nervous system disorders | ddMMMyyyy hh:mm / Day j / Ongoing / / | ddMMMyyyy hh:mm /<br>Day j /<br>xx h xx min | Y /<br>Moderate /<br>Not related /<br>Weather condition | Recovering/resolving / Not applicable / | Y /<br>N /<br> |
| Skkk/ppp | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: MedDRA version 18.1

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\c122-ae-03-tbl.sas



#### Table 14.3.2.1 - Treatment emergent adverse events leading to death, serious or leading to discontinuation (Safety set)

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | AE<br>Nr<br>/<br>FU<br>Nr | Verbatim /<br>Preferred Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> | Start or Follow-up Date/time / Start or Follow-up Day / End Date/time / End Day / Duration | IMP injection Date/time / Day / Time from IMP injection | Seriousness /<br>Severity /<br>Related to IMP /<br>Other relationship | Outcome / Action taken with IMP / Other action taken | Therapy required / Leading to discontinuation / Comments |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | 1 | Headache /<br>Headache /<br>Nervous system disorders | ddMMMyyyy hh:mm / Day j / Ongoing / / | ddMMMyyyy hh:mm /<br>Day j /<br>xx h xx min | Y /<br>Moderate /<br>Not related /<br>Weather condition | Recovering/resolving / Not applicable / | Y /<br>N /<br> |
| Skkk/ppp | ••• | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: MedDRA version 18.1

Source: Listing 16.2.7.1 - Treatment-emergent adverse events

Program: Tables\c122-ae-03-tbl.sas



#### Table 14.2.3.1 - Vital signs (Safety set)

## Safety Set

| | | | ocaine 1% | | | |
|---|---|---|---|---|---|---|
| Parameter | Time Point | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Systolic Blood Pressure (mmHg) | Screening | N | nn | nn | nn | nn |
| | | Mean | XXX.X | XXX.X | XXX.X | xxx.x |
| | | SD | XXX.X | XXX.X | XXX.X | xxx.x |
| | | CV% | XXX.X | XXX.X | XXX.X | xxx.x |
| | | Min | XXX | XXX | XXX | xxx |
| | | Median | XXX.X | XXX.X | XXX.X | xxx.x |
| | | Max | XXX | XXX | XXX | XXX |
| Systolic Blood Pressure (mmHg) | Baseline | N | nn | nn | nn | nn |
| | | Mean | XXX.X | XXX.X | XXX.X | xxx.x |
| | | SD | XXX.X | XXX.X | XXX.X | xxx.x |
| | | CV% | XXX.X | XXX.X | XXX.X | xxx.x |
| | | Min | XXX | XXX | XXX | xxx |
| | | Median | XXX.X | XXX.X | XXX.X | xxx.x |
| | | Max | XXX | XXX | XXX | xxx |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.9.1 - Vital signs Program: Tables\c122-vs-tbl.sas



#### Table 14.2.3.1 - Vital signs (Safety set)

# Safety Set

| | | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|---|
| Parameter | Time Point | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Systolic Blood Pressure (mmHg) | Discharge | N | nn | nn | nn | nn |
| | | Mean | XXX.X | XXX.X | XXX.X | xxx.x |
| | | SD | XXX.X | XXX.X | XXX.X | xxx.x |
| | | CV% | XXX.X | XXX.X | XXX.X | xxx.x |
| | | Min | XXX | XXX | XXX | xxx |
| | | Median | XXX.X | XXX.X | XXX.X | xxx.x |
| | | Max | xxx | XXX | XXX | XXX |
| Diastolic Blood Pressure (mmHg) | Screening | N | nn | nn | nn | nn |
| | | Mean | XXX.X | XXX.X | XXX.X | xxx.x |
| | | SD | XXX.X | XXX.X | XXX.X | xxx.x |
| | | CV% | XXX.X | XXX.X | XXX.X | xxx.x |
| | | Min | XXX | XXX | XXX | xxx |
| | | Median | XXX.X | XXX.X | XXX.X | xxx.x |
| | | Max | XXX | XXX | XXX | xxx |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.9.1 - Vital signs Program: Tables\c122-vs-tbl.sas



#### Table 14.2.3.1 - Vital signs (Safety set)

# Safety Set

| | | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|---|
| Parameter | Time Point | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Diastolic Blood Pressure (mmHg) | Baseline | N | nn | nn | nn | nn |
| | | Mean | XXX.X | XXX.X | XXX.X | xxx.x |
| | | SD | XXX.X | XXX.X | XXX.X | xxx.x |
| | | CV% | XXX.X | XXX.X | XXX.X | xxx.x |
| | | Min | XXX | XXX | XXX | xxx |
| | | Median | XXX.X | XXX.X | XXX.X | xxx.x |
| | | Max | xxx | XXX | XXX | XXX |
| Diastolic Blood Pressure (mmHg) | Discharge | N | nn | nn | nn | nn |
| | | Mean | XXX.X | XXX.X | XXX.X | xxx.x |
| | | SD | XXX.X | XXX.X | XXX.X | XXX.X |
| | | CV% | XXX.X | XXX.X | XXX.X | XXX.X |
| | | Min | XXX | XXX | XXX | xxx |
| | | Median | XXX.X | XXX.X | XXX.X | xxx.x |
| | | Max | XXX | XXX | XXX | xxx |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.9.1 - Vital signs Program: Tables\c122-vs-tbl.sas



#### Table 14.2.3.1 - Vital signs (Safety set)

# Safety Set Chloroproceine 1%

| | | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|---|
| Parameter | Time Point | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Heart Rate (beats/min) | Screening | N | nn | nn | nn | nn |
| | | Mean | XX.X | xx.x | XX.X | xx.x |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | xx.x |
| | | Min | XX | XX | XX | xx |
| | | Median | XX.X | XX.X | XX.X | xx.x |
| | | Max | XX | XX | XX | XX |
| Heart Rate (beats/min) | Baseline | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | xx.x |
| | | SD | XX.X | XX.X | XX.X | xx.x |
| | | CV% | XX.X | XX.X | XX.X | xx.x |
| | | Min | XX | XX | XX | XX |
| | | Median | XX.X | XX.X | XX.X | xx.x |
| | | Max | XX | XX | XX | XX |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.9.1 - Vital signs Program: Tables\c122-vs-tbl.sas



#### Table 14.2.3.1 - Vital signs (Safety set)

## Safety Set

| | | | Chloroprocaine 1% | | | |
|---|---|---|---|---|---|---|
| Parameter | Time Point | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Heart Rate (beats/min) | Discharge | N | nn | nn | nn | nn |
| | | Mean | XX.X | XX.X | XX.X | XX.X |
| | | SD | XX.X | XX.X | XX.X | XX.X |
| | | CV% | XX.X | XX.X | XX.X | xx.x |
| | | Min | XX | XX | XX | xx |
| | | Median | XX.X | XX.X | XX.X | xx.x |
| | | Max | XX | XX | XX | XX |
| Oxygen Saturation (%) | Screening | N | nn | nn | nn | nn |
| | | Mean | XX.XX | XX.XX | XX.XX | xx.xx |
| | | SD | XX.XX | XX.XX | XX.XX | xx.xx |
| | | CV% | XX.XX | XX.XX | XX.XX | xx.xx |
| | | Max | XX.X | XX.X | XX.X | xx.x |
| | | Median | XX.XX | XX.XX | XX.XX | xx.xx |
| | | Max | XX.X | XX.X | XX.X | xx.x |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.9.1 - Vital signs Program: Tables\c122-vs-tbl.sas



#### Table 14.2.3.1 - Vital signs (Safety set)

# Safety Set

| | | Chloroprocaine 1% | | | | |
|---|---|---|---|---|---|---|
| Parameter | Time Point | Statistics | 30 mg<br>N=XX | 40 mg<br>N=XX | 50 mg<br>N=XX | Overall<br>N=XX |
| Oxygen Saturation (%) | Baseline | N | nn | nn | nn | nn |
| | | Mean | XX.XX | xx.xx | XX.XX | XX.XX |
| | | SD | XX.XX | XX.XX | XX.XX | xx.xx |
| | | CV% | XX.XX | XX.XX | XX.XX | xx.xx |
| | | Max | XX.X | XX.X | XX.X | XX.X |
| | | Median | XX.XX | XX.XX | XX.XX | xx.xx |
| | | Max | XX.X | XX.X | XX.X | XX.X |
| Oxygen Saturation (%) | Discharge | N | nn | nn | nn | nn |
| | | Mean | XX.XX | XX.XX | XX.XX | xx.xx |
| | | SD | XX.XX | XX.XX | XX.XX | xx.xx |
| | | CV% | XX.XX | XX.XX | XX.XX | xx.xx |
| | | Max | XX.X | XX.X | XX.X | XX.X |
| | | Median | XX.XX | XX.XX | xx.xx | xx.xx |
| | | Max | XX.X | XX.X | XX.X | xx.x |

Note: Subjects are summarised according to the dose level of the product they actually received

Source: Listing 16.2.9.1 - Vital signs Program: Tables\c122-vs-tbl.sas



Table 14.3.5.2 - Pain assessment at the site of injection and at the site of surgery (Safety set)

| | | Safety Set Chloroprocaine 1% | | | | |
|---|---|---|---|---|---|---|
| Parameter | Time Point | Pain<br>Assessment <sup>1</sup> | 30 mg<br>N=XX<br>n (%) | 40 mg<br>N=XX<br>n (%) | 50 mg<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
| Pain at the Injection Site | Immediately after regression of spinal block | 0 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 1 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 2 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 3 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 4 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 5 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 6 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 7 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 8 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 9 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 10 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Note 1: Pain was assessed according to a numerical rating scale ranging from 0 (no pain) to 10 (worst imaginable pain)

Source: Listing 16.2.9.3 - Pain assessment at the site of injection and at the site of surgery

Program: Tables\c122-qs-03-tbl.sas



Table 14.3.5.2 - Pain assessment at the site of injection and at the site of surgery (Safety set)

| | | | | Safet | - | |
|---|---|---|---|---|---|---|
| | | | | Chloropro | | |
| Parameter | Time Point | Pain | 30 mg | 40 mg | 50 mg | Overall |
| | | Assessment 1 | N=XX | N=XX | N=XX | N=XX |
| | | | n (%) | n (%) | n (%) | n (%) |
| Pain at the Injection Site | Discharge | 0 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 1 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 2 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 3 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 4 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 5 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 6 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 7 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 8 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 9 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 10 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Note 1: Pain was assessed according to a numerical rating scale ranging from 0 (no pain) to 10 (worst imaginable pain)

Source: Listing 16.2.9.3 - Pain assessment at the site of injection and at the site of surgery

Program: Tables\c122-qs-03-tbl.sas



Table 14.3.5.2 - Pain assessment at the site of injection and at the site of surgery (Safety set)

| | | | | Safet | • | |
|---|---|---|---|---|---|---|
| | | | | Chloropro | | |
| Parameter | Time Point | Pain | 30 mg | 40 mg | 50 mg | Overall |
| | | Assessment 1 | N=XX | N=XX | N=XX | N=XX |
| | | | n (%) | n (%) | n (%) | n (%) |
| Pain at the Injection Site | Day 2 | 0 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 1 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 2 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 3 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 4 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 5 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 6 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 7 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 8 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 9 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 10 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Note 1: Pain was assessed according to a numerical rating scale ranging from 0 (no pain) to 10 (worst imaginable pain)

Source: Listing 16.2.9.3 - Pain assessment at the site of injection and at the site of surgery

Program: Tables\c122-qs-03-tbl.sas


Table 14.3.5.2 - Pain assessment at the site of injection and at the site of surgery (Safety set)

| | | | | Safet <sub>y</sub><br>Chloropro | • | |
|---|---|---|---|---|---|---|
| Parameter | Time Point | Pain<br>Assessment <sup>1</sup> | 30 mg<br>N=XX<br>n (%) | 40 mg<br>N=XX<br>n (%) | 50 mg<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
| Pain at the Injection Site | Day 7±1 | 0 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 1 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 2 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 3 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 4 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 5 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 6 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 7 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 8 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 9 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 10 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Note 1: Pain was assessed according to a numerical rating scale ranging from 0 (no pain) to 10 (worst imaginable pain)

Source: Listing 16.2.9.3 - Pain assessment at the site of injection and at the site of surgery

Program: Tables\c122-qs-03-tbl.sas



Table 14.3.5.2 - Pain assessment at the site of injection and at the site of surgery (Safety set)

| | | | | Safet<br>Chloropro | • | |
|---|---|---|---|---|---|---|
| Parameter | Time Point | Pain<br>Assessment <sup>1</sup> | 30 mg<br>N=XX<br>n (%) | 40 mg<br>N=XX<br>n (%) | 50 mg<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
| Pain at the Surgery Site | Immediately after regression of spinal block | 0 | nn (vv. v.) | nn (vv v) | nn (vv v) | nn (vv v) |
| rain at the Surgery Site | miniediately after regression of spinar block | 1 | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) | nn (xx.x)<br>nn (xx.x) |
| | | 2 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 3 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 4 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 5 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 6 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 7 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 8 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn(xx.x) |
| | | 9 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 10 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn(xx.x) |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Note 1: Pain was assessed according to a numerical rating scale ranging from 0 (no pain) to 10 (worst imaginable pain)

Source: Listing 16.2.9.3 - Pain assessment at the site of injection and at the site of surgery

Program: Tables\c122-qs-03-tbl.sas



Table 14.3.5.2 - Pain assessment at the site of injection and at the site of surgery (Safety set)

| | | | | Safet <sub>y</sub><br>Chloropro | • | |
|---|---|---|---|---|---|---|
| Parameter | Time Point | Pain<br>Assessment <sup>1</sup> | 30 mg<br>N=XX<br>n (%) | 40 mg<br>N=XX<br>n (%) | 50 mg<br>N=XX<br>n (%) | Overall<br>N=XX<br>n (%) |
| Pain at the Surgery Site | Discharge | 0 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn(xx.x) |
| | | 1 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 2 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 3 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 4 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 5 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 6 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 7 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 8 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 9 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 10 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Note 1: Pain was assessed according to a numerical rating scale ranging from 0 (no pain) to 10 (worst imaginable pain)

Source: Listing 16.2.9.3 - Pain assessment at the site of injection and at the site of surgery

Program: Tables\c122-qs-03-tbl.sas



Table 14.3.5.2 - Pain assessment at the site of injection and at the site of surgery (Safety set)

| | | | | Safet | - | |
|---|---|---|---|---|---|---|
| | | | | Chloropro | caine 1% | |
| Parameter | Time Point | Pain | 30 mg | 40 mg | 50 mg | Overall |
| | | Assessment 1 | N=XX | N=XX | N=XX | N=XX |
| | | | n (%) | n (%) | n (%) | n (%) |
| Pain at the Surgery Site | Day 2 | 0 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 1 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 2 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 3 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 4 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 5 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 6 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 7 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 8 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 9 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 10 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Note 1: Pain was assessed according to a numerical rating scale ranging from 0 (no pain) to 10 (worst imaginable pain)

Source: Listing 16.2.9.3 - Pain assessment at the site of injection and at the site of surgery

Program: Tables\c122-qs-03-tbl.sas



Table 14.3.5.2 - Pain assessment at the site of injection and at the site of surgery (Safety set)

| | | | | Safet | y Set | |
|---|---|---|---|---|---|---|
| | | | | Chloropro | | |
| Parameter | Time Point | Pain | 30 mg | 40 mg | 50 mg | Overall |
| | | Assessment 1 | N=XX | N=XX | N=XX | N=XX |
| | | | n (%) | n (%) | n (%) | n (%) |
| Pain at the Surgery Site | Day 7±1 | 0 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 1 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 2 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 3 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 4 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 5 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 6 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 7 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 8 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 9 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |
| | | 10 | nn (xx.x) | nn (xx.x) | nn (xx.x) | nn (xx.x) |

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Note 1: Pain was assessed according to a numerical rating scale ranging from 0 (no pain) to 10 (worst imaginable pain)

Source: Listing 16.2.9.3 - Pain assessment at the site of injection and at the site of surgery

Program: Tables\c122-qs-03-tbl.sas



#### Table 14.3.5.3 - Transient neurological symptoms (Safety set)

#### Safety Set Chloroprocaine 1% 40 mg **Time Point** Assessment 30 mg 50 mg **Overall** N=XXN=XX N=XXN=XXn (%) n (%) n (%) n (%) Transient Neurological Symptoms Day 2 Y nn (xx.x) nn (xx.x) nn(xx.x)nn (xx.x) N nn (xx.x) nn (xx.x) nn(xx.x)nn (xx.x) Transient Neurological Symptoms Day 7±1 Y nn(xx.x)nn(xx.x)nn (xx.x) nn (xx.x) N nn (xx.x) nn (xx.x) nn (xx.x) nn (xx.x)

Note: Subjects are summarised according to the dose level of the product they actually received

The denominator for calculating the proportions is the number of subjects in each dose level and overall in the per protocol set

Source: Listing 16.2.9.4 - Transient neurological symptoms

Program: Tables\c122-qs-03-tbl.sas


Statistical analysis plan CRO-14-122 Sponsor code CHL.1/02-2014 Chloroprocaine 1% - Spinal block Final version 1.0, 02FEB2016



Figure 14.2.3.1 - Mean plasma concentration curves of Chloroprocaine (PK set 1)

Mean plasma concentration curves of Chloroprocaine (linear scale and logarithmic/linear scale)


Statistical analysis plan CRO-14-122 Sponsor code CHL.1/02-2014 Chloroprocaine 1% - Spinal block Final version 1.0, 02FEB2016



Figure 14.2.3.2 - Mean plasma concentration curves of CABA (PK set 1)

Mean plasma concentration curves of CABA (linear scale and logarithmic/linear scale)




Statistical analysis plan CRO-14-122 Sponsor code CHL.1/02-2014 Chloroprocaine 1% - Spinal block Final version 1.0, 02FEB2016

#### Section 16.2 - Individual Subject Data Listings and Figures Shells

| Listing 16.2.1.1 - Discontinued subjects |
|---|
| Listing 16.2.2.1 - Protocol deviations |
| Listing 16.2.3.1 - Subjects excluded from the efficacy, PK or safety analysis |
| Listing 16.2.4.1 - Subjects' disposition |
| Listing 16.2.4.2 - Analysis sets |
| Listing 16.2.4.3 - Demography |
| Listing 16.2.4.4 - Inclusion/Exclusion criteria not met |
| Listing 16.2.5.1 - IMP spinal injection |
| Listing 16.2.5.2 - Sedation and premedication |
| Listing 16.2.5.3 - PK blood samples collection and plasma concentrations |
| Listing 16.2.5.4 - PK urine sample collection, urinary concentration and urinary excretion |
| Listing 16.2.6.1 - Surgical procedure |

Listing 16.2.6.2 - Sensory and motor block assessment

Listing 16.2.6.3 - Time to events and maximum level of sensory block

Listing 16.2.6.4 - Effectiveness of anaesthesia and quality of spinal block

Listing 16.2.7.1 - Treatment-emergent adverse events

Listing 16.2.7.2 - Pre-treatment adverse events

Listing 16.2.9.1 - Vital signs

Listing 16.2.9.2 - ECG

Listing 16.2.9.3 - Pain assessment at the site of injection and at the site of surgery

Listing 16.2.9.4 - Transient neurological symptoms

Listing 16.2.9.5 - Modified Aldrete's scoring scale

Listing 16.2.10.1 - Medical and surgical history

Listing 16.2.10.2 - Physical examination

Listing 16.2.10.3 - Prior and concomitant medications

Listing 16.2.10.4 - Subjects study visits

Listing 16.2.10.5 - Pregnancy test

Figure 16.2.5.j - Subject [Sxxx]/[nnn] - Individual plasma concentration curves of Chloroprocaine and CABA



**Listing 16.2.1.1 - Discontinued Subjects** 

| Subject<br>ID | IMP administered | Sex | Age<br>(years) | Last<br>visit | Time elapsed<br>from IMP<br>spinal injection<br>(days) | Date of premature discontinuation | Primary reason for subject premature discontinuation |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | Chloroprocaine 1% - 30 mg | M | XX | Visit A | X | ddMMMyyyy | Reason A |
| Sjjj/nnn | Chloroprocaine 1% - 40 mg | F | XX | Visit B | X | ddMMMyyyy | Reason B |
| Sjjj/nnn | Chloroprocaine 1% - 50 mg | F | XX | Visit C | X | ddMMMyyyy | Reason C |
| Sjjj/nnn | Not Treated | F | XX | Visit C | X | ddMMMyyyy | Reason D |
| Sjjj/nnn | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ds-lst.sas



# **Listing 16.2.2.1 - Protocol deviations**

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | <b>Deviation</b><br><b>Number</b> | Deviation<br>Category | Deviation<br>Coded<br>Term | Deviation Description |
|---|---|---|---|---|
| Sjjj/nnn | 1 | Major | Coded Term A | Description A |
| Sjjj/nnn | 2 | Minor | Coded Term B | Description B |
| Sxxx/ppp | 1 | Major | Coded Term A | Description A |
| Sxxx/ppp | 2 | Minor | Coded Term B | Description B |
| Sxxx/ppp | | | | |

Note: Only subjects with protocol deviations are listed. Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-dv-lst.sas



# **Listing 16.2.2.1 - Protocol deviations**

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Deviation<br>Number | Deviation<br>Category | Deviation<br>Coded<br>Term | Deviation Description |
|---|---|---|---|---|
| Sjjj/nnn | 1 | Major | Coded Term A | Description A |
| Sjjj/nnn | 2 | Minor | Coded Term B | Description B |
| Sxxx/ppp | 1 | Major | Coded Term A | Description A |
| Sxxx/ppp | 2 | Minor | Coded Term B | Description B |
| Sxxx/ppp | | | | |

Note: Only subjects with protocol deviations are listed. Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-dv-lst.sas



# **Listing 16.2.2.1 - Protocol deviations**

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Deviation<br>Number | Deviation<br>Category | Deviation<br>Coded<br>Term | Deviation Description |
|---|---|---|---|---|
| Sjjj/nnn | 1 | Major | Coded Term A | Description A |
| Sjjj/nnn | 2 | Minor | Coded Term B | Description B |
| Sxxx/ppp | 1 | Major | Coded Term A | Description A |
| Sxxx/ppp | 2 | Minor | Coded Term B | Description B |
| Sxxx/ppp | | | | |

Note: Only subjects with protocol deviations are listed. Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-dv-lst.sas



# **Listing 16.2.2.1 - Protocol deviations**

**Investigational Medicinal Product: Not Assigned** 

| Subject<br>ID | Deviation<br>Number | <b>Deviation Category</b> | Deviation<br>Coded<br>Term | Deviation Description |
|---|---|---|---|---|
| Sjjj/nnn | 1 | Major | Coded Term A | Description A |
| Sjjj/nnn | 2 | Minor | Coded Term B | Description B |
| Sxxx/ppp | 1 | Major | Coded Term A | Description A |
| Sxxx/ppp | 2 | Minor | Coded Term B | Description B |
| Sxxx/ppp | | | | |

Note: Only subjects with protocol deviations are listed. Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-dv-lst.sas



# **Listing 16.2.2.1 - Protocol deviations**

**Investigational Medicinal Product: Not Treated** 

| Subject<br>ID | Deviation<br>Number | <b>Deviation Category</b> | Deviation<br>Coded<br>Term | Deviation Description |
|---|---|---|---|---|
| Sjjj/nnn | 1 | Major | Coded Term A | Description A |
| Sjjj/nnn | 2 | Minor | Coded Term B | Description B |
| Sxxx/ppp | 1 | Major | Coded Term A | Description A |
| Sxxx/ppp | 2 | Minor | Coded Term B | Description B |
| Sxxx/ppp | | | | |

Note: Only subjects with protocol deviations are listed. Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-dv-lst.sas



Listing 16.2.3.1 - Subjects excluded from the efficacy and/or PK and/or safety analysis

| Subject<br>ID | Investigational<br>Medicinal<br>Product | Sex | Age<br>(years) | Enrolled<br>Set | Randomised | Safety<br>Set | Full<br>Analysis<br>Set | Per<br>Protocol<br>Set | PK<br>Set 1 | PK<br>Set 2 | Reason for the exclusion |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Sjjj | Not Assigned | M | XX | N | N | N | N | N | N | N | Reason D |
| Sjjj/nnn | Chloroprocaine 1% - 30 mg | M | XX | Y | Y | Y | Y | N | Y | N | Reason A |
| Sjjj/nnn | Chloroprocaine 1% - 40 mg | M | XX | Y | Y | Y | Y | Y | N | Y | Reason B |
| Sjjj/nnn | Chloroprocaine 1% - 50 mg | M | XX | Y | Y | N | N | N | N | Y | Reason C |
| Sjjj/nnn | Not Treated | F | XX | Y | Y | N | N | N | N | N | Reason E |
| Sjjj/nnn | | | | | • | | • | | | •• | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ds-lst.sas



#### Listing 16.2.4.1 - Subjects' disposition

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Date of<br>Informed<br>Consent | Date of<br>Screening | Date of<br>Randomisation | Date of<br>Spinal<br>Injection | Completed or Discontinued | Date of Study<br>Completion or<br>Discontinuation | Date of<br>End of<br>Partecipation | Comments<br>Reason for discontinuation |
|---|---|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Discontinued | ddMMMyyyy | ddMMMyyyy | Reason A |
| Sjjj/nnn | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Completed | ddMMMyyyy | ddMMMyyyy | |
| Sjjj/nnn | | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ds-lst.sas



#### Listing 16.2.4.1 - Subjects' disposition

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Date of<br>Informed<br>Consent | Date of<br>Screening | Date of<br>Randomisation | Date of<br>Spinal<br>Injection | Completed or<br>Discontinued | Date of Study<br>Completion or<br>Discontinuation | Date of<br>End of<br>Partecipation | Comments<br>Reason for discontinuation |
|---|---|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Discontinued | ddMMMyyyy | ddMMMyyyy | Reason B |
| Sjjj/nnn | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Completed | ddMMMyyyy | ddMMMyyyy | |
| Sjjj/nnn | | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ds-lst.sas



#### Listing 16.2.4.1 - Subjects' disposition

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Date of<br>Informed<br>Consent | Date of<br>Screening | Date of<br>Randomisation | Date of<br>Spinal<br>Injection | Completed or<br>Discontinued | Date of Study<br>Completion or<br>Discontinuation | Date of<br>End of<br>Partecipation | Comments<br>Reason for discontinuation |
|---|---|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Discontinued | ddMMMyyyy | ddMMMyyyy | Reason C |
| Sjjj/nnn | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | Completed | ddMMMyyyy | ddMMMyyyy | |
| Sjjj/nnn | | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ds-lst.sas



# Listing 16.2.4.1 - Subjects' disposition

**Investigational Medicinal Product: Not Assigned** 

| Subject<br>ID | Date of<br>Informed<br>Consent | Date of<br>Screening | Date of<br>Randomisation | Date of<br>Spinal<br>Injection | Completed or Discontinued | Date of Study<br>Completion or<br>Discontinuation | Date of<br>End of<br>Partecipation | Comments<br>Reason for discontinuation |
|---|---|---|---|---|---|---|---|---|
| Sjjj | ddMMMyyyy | ddMMMyyyy | | | | | | Reason D |
| Sjjj | | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ds-lst.sas



# Listing 16.2.4.1 - Subjects' disposition

**Investigational Medicinal Product: Not Treated** 

| Subject<br>ID | Date of<br>Informed<br>Consent | Date of<br>Screening | Date of Randomisation | Date of<br>Spinal<br>Injection | Completed or Discontinued | Date of Study<br>Completion or<br>Discontinuation | Date of<br>End of<br>Partecipation | Comments<br>Reason for discontinuation |
|---|---|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy | ddMMMyyyy | ddMMMyyyy | | Discontinued | ddMMMyyyy | ddMMMyyyy | Reason E |
| Sjjj/nnn | | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ds-lst.sas



#### Listing 16.2.4.2 - Analysis sets

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Enrolled<br>Set | Randomised | Safety<br>Set | Full<br>Analysis<br>Set | Per<br>Protocol<br>Set | PK<br>Set 1 | PK<br>Set 2 | Reason for the exclusion |
|---|---|---|---|---|---|---|---|---|
| Sjjj/nnn | Y | Y | Y | Y | N | Y | N | Reason A |
| Sjjj/nnn | | • | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ds-lst.sas



#### Listing 16.2.4.2 - Analysis sets

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Enrolled<br>Set | Randomised | Safety<br>Set | Full<br>Analysis<br>Set | Per<br>Protocol<br>Set | PK<br>Set 1 | PK<br>Set 2 | Reason for the exclusion |
|---|---|---|---|---|---|---|---|---|
| Sjjj/nnn | Y | Y | Y | Y | Y | N | Y | Reason B |
| Sjjj/nnn | | | | | • | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ds-lst.sas



#### Listing 16.2.4.2 - Analysis sets

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Enrolled<br>Set | Randomised | Safety<br>Set | Full<br>Analysis<br>Set | Per<br>Protocol<br>Set | PK<br>Set 1 | PK<br>Set 2 | Reason for the exclusion |
|---|---|---|---|---|---|---|---|---|
| Sjjj/nnn | Y | Y | N | N | N | N | Y | Reason C |
| Sjjj/nnn | | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ds-lst.sas



#### Listing 16.2.4.2 - Analysis sets

**Investigational Medicinal Product: Not Assigned** 

| Subject<br>ID | Enrolled<br>Set | Randomised | Safety<br>Set | Full<br>Analysis<br>Set | Per<br>Protocol<br>Set | PK<br>Set 1 | PK<br>Set 2 | Reason for the exclusion |
|---|---|---|---|---|---|---|---|---|
| Sjjj | N | N | N | N | N | N | N | Reason D |
| Sjjj | •• | • | •• | • | • | •• | •• | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ds-lst.sas



#### Listing 16.2.4.2 - Analysis sets

**Investigational Medicinal Product: Not Treated** 

| Subject<br>ID | Enrolled<br>Set | Randomised | Safety<br>Set | Full<br>Analysis<br>Set | Per<br>Protocol<br>Set | PK<br>Set 1 | PK<br>Set 2 | Reason for the exclusion |
|---|---|---|---|---|---|---|---|---|
| Sjjj/nnn | Y | Y | N | N | N | N | N | Reason E |
| Sjjj/nnn | | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ds-lst.sas



# Listing 16.2.4.3 - Demography

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Sex | Race | Age<br>(years) | Height<br>(cm) | Weight (kg) | Body Mass Index<br>(kg/m²) |
|---|---|---|---|---|---|---|
| Sjjj/nnn | M | Race A | XX | XXX | XX.X | XX.X |
| Sxxx/ppp | F | Race B | XX | XXX | XX.X | xx.x |
| Szzz/ttt | | | | | | ••• |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-dm-lst.sas



# **Listing 16.2.4.3 - Demography**

# Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Sex | Race | Age<br>(years) | Height<br>(cm) | Weight (kg) | Body Mass Index (kg/m²) |
|---|---|---|---|---|---|---|
| Sjjj/nnn | M | Race A | XX | XXX | XX.X | XX.X |
| Sxxx/ppp | F | Race B | XX | XXX | XX.X | XX.X |
| Szzz/ttt | | ••• | | ••• | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-dm-lst.sas



# Listing 16.2.4.3 - Demography

#### Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Sex | Race | Age<br>(years) | Height<br>(cm) | Weight<br>(kg) | Body Mass Index<br>(kg/m²) |
|---|---|---|---|---|---|---|
| Sjjj/nnn | M | Race A | XX | XXX | XX.X | XX.X |
| Sxxx/ppp | F | Race B | XX | XXX | XX.X | XX.X |
| Szzz/ttt | | | | ••• | | ••• |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-dm-lst.sas



# Listing 16.2.4.3 - Demography

**Investigational Medicinal Product: Not Assigned** 

| Subject<br>ID | Sex | Race | Age<br>(years) | Height (cm) | Weight (kg) | Body Mass Index<br>(kg/m²) |
|---|---|---|---|---|---|---|
| Sjjj | M | Race A | XX | XXX | XX.X | XX.X |
| Sxxx | F | Race B | XX | xxx | XX.X | xx.x |
| Szzz | | | | | ••• | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-dm-lst.sas



# **Listing 16.2.4.3 - Demography**

# **Investigational Medicinal Product: Not Treated**

| Subject<br>ID | Sex | Race | Age<br>(years) | Height<br>(cm) | Weight (kg) | Body Mass Index<br>(kg/m²) |
|---|---|---|---|---|---|---|
| Sjjj/nnn | M | Race A | XX | XXX | XX.X | XX.X |
| Sxxx/ppp | F | Race B | XX | XXX | XX.X | XX.X |
| Szzz/ttt | | ••• | | ••• | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-dm-lst.sas



# Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Patient<br>ID | Time point | Assessment<br>Date | Inclusion/<br>Exclusion | Criterion<br>Number | Criterion |
|---|---|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy | Exclusion | 1 | Physical findings: clinically significant abnormal physical findings |
| ••• | ••• | | ••• | | <b></b> |

Note: Subjects are listed according to the dose level of the product they were assigned to

Program: Listings\c122-ie-lst.sas



# Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Patient<br>ID | Time point | Assessment<br>Date | Inclusion/<br>Exclusion | Criterion<br>Number | Criterion |
|---|---|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy | Exclusion | 1 | Physical findings: clinically significant abnormal physical findings |

Note: Subjects are listed according to the dose level of the product they were assigned to

Program: Listings\c122-ie-lst.sas



# Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Patient<br>ID | Time point | Assessment<br>Date | Inclusion/<br>Exclusion | Criterion<br>Number | Criterion |
|---|---|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy | Exclusion | 1 | Physical findings: clinically significant abnormal physical findings |
| ••• | ••• | ••• | ••• | | <b></b> |

Note: Subjects are listed according to the dose level of the product they were assigned to

Program: Listings\c122-ie-lst.sas



# Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

**Investigational Medicinal Product: Not Assigned** 

| Patient<br>ID | Time point | Assessment<br>Date | Inclusion/<br>Exclusion | Criterion<br>Number | Criterion |
|---|---|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy | Exclusion | 1 | Physical findings: clinically significant abnormal physical findings |

Note: Subjects are listed according to the dose level of the product they were assigned to

Program: Listings\c122-ie-lst.sas



# Listing 16.2.4.4 - Inclusion/Exclusion criteria not met

**Investigational Medicinal Product: Not Treated** 

| Patient<br>ID | Time point | Assessment<br>Date | Inclusion/<br>Exclusion | Criterion<br>Number | Criterion |
|---|---|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy | Exclusion | 1 | Physical findings: clinically significant abnormal physical findings |
| ••• | ••• | | | | |

Note: Subjects are listed according to the dose level of the product they were assigned to

Program: Listings\c122-ie-lst.sas


# Listing 16.2.5.1 - IMP spinal injection

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Anatomical location of the spinal injection | Kit<br>Identifier | Injection<br>Date/time | Was the planned volume administered as per protocol? | Comments |
|---|---|---|---|---|---|
| Sjjj/nnn | L3/L4 | Knnn | ddMMMyyyy hh:mm | Y | |
| Skkk/ttt | L4/L5 | Kttt | ddMMMyyyy hh:mm | Y | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ex-lst.sas



# Listing 16.2.5.1 - IMP spinal injection

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Anatomical location of the spinal injection | Kit<br>Identifier | Injection<br>Date/time | Was the planned volume administered as per protocol? | Comments |
|---|---|---|---|---|---|
| Sjjj/nnn | L3/L4 | Knnn | ddMMMyyyy hh:mm | Y | |
| Skkk/ttt | L4/L5 | Kttt | ddMMMyyyy hh:mm | Y | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ex-lst.sas



# Listing 16.2.5.1 - IMP spinal injection

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Anatomical location of the spinal injection | Kit<br>Identifier | Injection<br>Date/time | Was the planned volume administered as per protocol? | Comments |
|---|---|---|---|---|---|
| Sjjj/nnn | L3/L4 | Knnn | ddMMMyyyy hh:mm | Y | |
| Skkk/ttt | L4/L5 | Kttt | ddMMMyyyy hh:mm | Y | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ex-lst.sas



# Listing 16.2.5.1 - IMP spinal injection

**Investigational Medicinal Product: Not Treated** 

| Subject<br>ID | Anatomical location of the spinal injection | Kit<br>Identifier | Injection<br>Date/time | Was the planned volume administered as per protocol? | Comments |
|---|---|---|---|---|---|
| Sjjj/nnn | L3/L4 | Knnn | | N | |
| Skkk/ttt | L4/L5 | Kttt | | N | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ex-lst.sas



# Listing 16.2.5.2 - Sedation and premedication

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Sedation with i.v. Midazolam? | Injection<br>Date/time | Injected<br>Dose | Premedication with Ringer's solution? | Infusion start<br>Date/time | Infusion start<br>End/time | Infused<br>Volume |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | Y | ddMMMyyyy hh:mm | 2 mg | Y | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | 500 mL |
| Sjjj/nnn | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-cm-lst.sas



## Listing 16.2.5.2 - Sedation and premedication

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Sedation with i.v. Midazolam? | Injection<br>Date/time | Injected<br>Dose | Premedication with Ringer's solution? | Infusion start<br>Date/time | Infusion start<br>End/time | Infused<br>Volume |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | Y | ddMMMyyyy hh:mm | 2 mg | Y | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | 500 mL |
| Sjjj/nnn | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-cm-lst.sas



## Listing 16.2.5.2 - Sedation and premedication

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Sedation with i.v. Midazolam? | Injection<br>Date/time | Injected<br>Dose | Premedication with Ringer's solution? | Infusion start<br>Date/time | Infusion start<br>End/time | Infused<br>Volume |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | Y | ddMMMyyyy hh:mm | 2 mg | Y | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | 500 mL |
| Sjjj/nnn | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-cm-lst.sas



# Listing 16.2.5.2 - Sedation and premedication

**Investigational Medicinal Product: Not Treated** 

| Subject<br>ID | Sedation with i.v. Midazolam? | Injection<br>Date/time | Injected<br>Dose | Premedication with Ringer's solution? | Infusion start<br>Date/time | Infusion start<br>End/time | Infused<br>Volume |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | Y | ddMMMyyyy hh:mm | 2 mg | Y | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | 500 mL |
| Sjjj/nnn | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-cm-lst.sas



# Listing 16.2.5.3 - PK blood samples collection and plasma concentrations

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | IMP Injection<br>Date/time | Sample<br>Number | Time Point | Collection<br>Date/time | Time from<br>IMP<br>Injection | Chloroprocaine<br>Plasma<br>Concentration<br>(ng/mL) | CABA Plasma Concentration (ng/mL) |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | 1 | Pre-dose (0) - Within 60 min before IMP administration | ddMMMyyyy hh:mm | -xx min | XX.XX | XX.XX |
| Sjjj/nnn | ddMMMyyyy hh:mm | 2 | 5 min after spinal injection | ddMMMyyyy hh:mm | xx min | XX.XX | XX.XX |
| Sjjj/nnn | ddMMMyyyy hh:mm | 3 | 10 min after spinal injection | ddMMMyyyy hh:mm | xx min | XX.XX | XX.XX |
| Sjjj/nnn | ddMMMyyyy hh:mm | 4 | 30 min after spinal injection $\pm 1$ min | ddMMMyyyy hh:mm | xx min | XX.XX | XX.XX |
| Sjjj/nnn | ddMMMyyyy hh:mm | 5 | 60 min after spinal injection $\pm$ 3 min | ddMMMyyyy hh:mm | xx min | XX.XX | XX.XX |
| Skkk/ttt | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-pc-lst.sas



# Listing 16.2.5.3 - PK blood samples collection and plasma concentrations

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | IMP Injection<br>Date/time | Sample<br>Number | Time Point | Collection<br>Date/time | Time from<br>IMP<br>Injection | Chloroprocaine<br>Plasma<br>Concentration<br>(ng/mL) | CABA Plasma Concentration (ng/mL) |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | 1 | Pre-dose (0) - Within 60 min before IMP administration | ddMMMyyyy hh:mm | -xx min | XX.XX | XX.XX |
| Sjjj/nnn | ddMMMyyyy hh:mm | 2 | 5 min after spinal injection | ddMMMyyyy hh:mm | xx min | XX.XX | XX.XX |
| Sjjj/nnn | ddMMMyyyy hh:mm | 3 | 10 min after spinal injection | ddMMMyyyy hh:mm | xx min | XX.XX | XX.XX |
| Sjjj/nnn | ddMMMyyyy hh:mm | 4 | 30 min after spinal injection $\pm 1$ min | ddMMMyyyy hh:mm | xx min | XX.XX | XX.XX |
| Sjjj/nnn | ddMMMyyyy hh:mm | 5 | 60 min after spinal injection $\pm$ 3 min | ddMMMyyyy hh:mm | xx min | XX.XX | XX.XX |
| Skkk/ttt | ••• | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-pc-lst.sas



# Listing 16.2.5.3 - PK blood samples collection and plasma concentrations

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | IMP Injection<br>Date/time | Sample<br>Number | Time Point | Collection<br>Date/time | Time from<br>IMP<br>Injection | Chloroprocaine<br>Plasma<br>Concentration<br>(ng/mL) | CABA Plasma Concentration (ng/mL) |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | 1 | Pre-dose (0) - Within 60 min before IMP administration | ddMMMyyyy hh:mm | -xx min | XX.XX | XX.XX |
| Sjjj/nnn | ddMMMyyyy hh:mm | 2 | 5 min after spinal injection | ddMMMyyyy hh:mm | xx min | XX.XX | XX.XX |
| Sjjj/nnn | ddMMMyyyy hh:mm | 3 | 10 min after spinal injection | ddMMMyyyy hh:mm | xx min | XX.XX | xx.xx |
| Sjjj/nnn | ddMMMyyyy hh:mm | 4 | 30 min after spinal injection $\pm 1$ min | ddMMMyyyy hh:mm | xx min | XX.XX | XX.XX |
| Sjjj/nnn | ddMMMyyyy hh:mm | 5 | 60 min after spinal injection $\pm$ 3 min | ddMMMyyyy hh:mm | xx min | XX.XX | XX.XX |
| Skkk/ttt | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-pc-lst.sas



# Listing 16.2.5.4 - PK urine sample collection, urinary concentration and urinary excretion

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | IMP Injection<br>Date/time | Time Point | Collection<br>Date/time | Time from<br>IMP Injection | Urine<br>Volume<br>(mL) | CABA<br>Urinary<br>Concentration<br>(ng/mL) | CABA Urinary Excretion (%) |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | First Spontaneous Urine Voiding | ddMMMyyyy hh:mm | zz h xx min | XXX | XX.XX | XXX.XX |
| Skkk/ttt | ••• | <b></b> | | | ••• | | ••• |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-pc-lst.sas



# Listing 16.2.5.4 - PK urine sample collection, urinary concentration and urinary excretion

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | IMP Injection<br>Date/time | Time Point | Collection<br>Date/time | Time from<br>IMP Injection | Urine<br>Volume<br>(mL) | CABA<br>Urinary<br>Concentration<br>(ng/mL) | CABA<br>Urinary<br>Excretion<br>(%) |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | First Spontaneous Urine Voiding | ddMMMyyyy hh:mm | zz h xx min | XXX | XX.XX | XXX.XX |
| Skkk/ttt | ••• | <b></b> | ••• | ••• | ••• | ••• | ••• |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-pc-lst.sas



# Listing 16.2.5.4 - PK urine sample collection, urinary concentration and urinary excretion

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | IMP Injection<br>Date/time | Time Point | Collection<br>Date/time | Time from IMP Injection | Urine<br>Volume<br>(mL) | CABA<br>Urinary<br>Concentration<br>(ng/mL) | CABA<br>Urinary<br>Excretion<br>(%) |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | First Spontaneous Urine Voiding | ddMMMyyyy hh:mm | zz h xx min | XXX | XX.XX | XXX.XX |
| Skkk/ttt | | | | | ••• | ••• | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-pc-lst.sas



# **Listing 16.2.6.1 - Surgical procedure**

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Type of Lower Limb Surgery / Preferred Term <sup>1</sup> / System Organ Class <sup>1</sup> | Required<br>Metameric<br>Level<br>of<br>Sensory<br>Block | Surgery<br>Executed? | Surgery start Date/time / Surgery end Date/time / Duration | Rescue<br>Anaesthesia<br>or<br>Analgesia? | Rescue<br>Anaesthesia<br>or Analgesia<br>Date/time | General<br>Anaesthesia<br>Required? | General<br>Anaesthesia<br>Date/time |
|---|---|---|---|---|---|---|---|---|
| Sjjj/nnn | Arthroscopic meniscectomy (right knee) / Meniscus removal / Surgical and medical procedures | T12 | Y | ddMMMyyyy hh:mm<br>ddMMMyyyy hh:mm<br>xx min | Y | ddMMMyyyy hh:mm | Y | ddMMMyyyy hh:mm |
| Skkk/ttt | | | | ••• | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-ce-lst.sas



# Listing 16.2.6.2 - Sensory and motor block assessment

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Spinal Injection,<br>Readiness for Surgery<br>or Regression of<br>Two Dermatomers<br>Date/time | Time Point | Assessment<br>Date/time | Elapsed<br>Time | Metameric<br>Level of<br>Sensory<br>Block | Bromage<br>Score |
|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | 2 min after spinal injection | ddMMMyyyy hh:mm | zz h xx min | L4 | 0 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 4 min after spinal injection | ddMMMyyyy hh:mm | zz h xx min | L1 | 1 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 6 min after spinal injection | ddMMMyyyy hh:mm | zz h xx min | T12 | 2 |
| Sjjj/nnn | ddMMMyyyy hh:mm | | ddMMMyyyy hh:mm | zz h xx min | ••• | ••• |
| Sjjj/nnn | ddMMMyyyy hh:mm | 5 min after readiness for surgery $\pm 1$ min | ddMMMyyyy hh:mm | zz h xx min | T11 | 2 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 10 min after readiness for surgery $\pm$ 1 min | ddMMMyyyy hh:mm | zz h xx min | T10 | 3 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 15 min after readiness for surgery $\pm$ 1 min | ddMMMyyyy hh:mm | zz h xx min | Т8 | 3 |
| Sjjj/nnn | ddMMMyyyy hh:mm | | ddMMMyyyy hh:mm | zz h xx min | | |
| Sjjj/nnn | ddMMMyyyy hh:mm | 30 min after regression of two dermatomers $\pm$ 5 min | ddMMMyyyy hh:mm | zz h xx min | T12 | 3 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 1 hour after regression of two dermatomers $\pm$ 5 min | ddMMMyyyy hh:mm | zz h xx min | L1 | 2 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 1 hour and 30 min after regression of two dermatomers $\pm$ 5 min | ddMMMyyyy hh:mm | zz h xx min | L3 | 1 |
| Sjjj/nnn | ddMMMyyyy hh:mm | | ddMMMyyyy hh:mm | zz h xx min | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



Listing 16.2.6.2 - Sensory and motor block assessment

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Spinal Injection,<br>Readiness for Surgery<br>or Regression of<br>Two Dermatomers<br>Date/time | Time Point | Assessment<br>Date/time | Elapsed<br>Time | Metameric<br>Level of<br>Sensory<br>Block | Bromage<br>Score |
|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | 2 min after spinal injection | ddMMMyyyy hh:mm | zz h xx min | L4 | 0 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 4 min after spinal injection | ddMMMyyyy hh:mm | zz h xx min | L1 | 1 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 6 min after spinal injection | ddMMMyyyy hh:mm | zz h xx min | T12 | 2 |
| Sjjj/nnn | ddMMMyyyy hh:mm | | ddMMMyyyy hh:mm | zz h xx min | ••• | ••• |
| Sjjj/nnn | ddMMMyyyy hh:mm | 5 min after readiness for surgery $\pm 1$ min | ddMMMyyyy hh:mm | zz h xx min | T11 | 2 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 10 min after readiness for surgery $\pm$ 1 min | ddMMMyyyy hh:mm | zz h xx min | T10 | 3 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 15 min after readiness for surgery $\pm$ 1 min | ddMMMyyyy hh:mm | zz h xx min | T8 | 3 |
| Sjjj/nnn | ddMMMyyyy hh:mm | <b></b> | ddMMMyyyy hh:mm | zz h xx min | | |
| Sjjj/nnn | ddMMMyyyy hh:mm | 30 min after regression of two dermatomers $\pm$ 5 min | ddMMMyyyy hh:mm | zz h xx min | T12 | 3 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 1 hour after regression of two dermatomers $\pm$ 5 min | ddMMMyyyy hh:mm | zz h xx min | L1 | 2 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 1 hour and 30 min after regression of two dermatomers $\pm$ 5 min | ddMMMyyyy hh:mm | zz h xx min | L3 | 1 |
| Sjjj/nnn | ddMMMyyyy hh:mm | | ddMMMyyyy hh:mm | zz h xx min | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



# Listing 16.2.6.2 - Sensory and motor block assessment

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Spinal Injection,<br>Readiness for Surgery<br>or Regression of<br>Two Dermatomers<br>Date/time | Time Point | Assessment<br>Date/time | Elapsed<br>Time | Metameric<br>Level of<br>Sensory<br>Block | Bromage<br>Score |
|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | 2 min after spinal injection | ddMMMyyyy hh:mm | zz h xx min | L4 | 0 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 4 min after spinal injection | ddMMMyyyy hh:mm | zz h xx min | L1 | 1 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 6 min after spinal injection | ddMMMyyyy hh:mm | zz h xx min | T12 | 2 |
| Sjjj/nnn | ddMMMyyyy hh:mm | | ddMMMyyyy hh:mm | zz h xx min | ••• | ••• |
| Sjjj/nnn | ddMMMyyyy hh:mm | 5 min after readiness for surgery $\pm 1$ min | ddMMMyyyy hh:mm | zz h xx min | T11 | 2 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 10 min after readiness for surgery $\pm$ 1 min | ddMMMyyyy hh:mm | zz h xx min | T10 | 3 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 15 min after readiness for surgery $\pm$ 1 min | ddMMMyyyy hh:mm | zz h xx min | T8 | 3 |
| Sjjj/nnn | ddMMMyyyy hh:mm | <b></b> | ddMMMyyyy hh:mm | zz h xx min | | |
| Sjjj/nnn | ddMMMyyyy hh:mm | 30 min after regression of two dermatomers $\pm$ 5 min | ddMMMyyyy hh:mm | zz h xx min | T12 | 3 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 1 hour after regression of two dermatomers $\pm$ 5 min | ddMMMyyyy hh:mm | zz h xx min | L1 | 2 |
| Sjjj/nnn | ddMMMyyyy hh:mm | 1 hour and 30 min after regression of two dermatomers $\pm$ 5 min | ddMMMyyyy hh:mm | zz h xx min | L3 | 1 |
| Sjjj/nnn | ddMMMyyyy hh:mm | | ddMMMyyyy hh:mm | zz h xx min | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



# Listing 16.2.6.3 - Time to events and maximum level of sensory block

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Spinal Injection Date/time | Spinal Injection Event Date/time | | Time<br>to Event | Metameric<br>Level |
|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | Regression of Spinal Block | Date/time<br>ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Onset of Sensory Block | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Onset of Motor Block | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Readiness for Surgery | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Regression of Sensory Block | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Regression of Motor Block | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Unassisted Ambulation | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Maximum Level of Sensory Block | ddMMMyyyy hh:mm | yy h xx min | T8 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Regression of Two Dermatomers | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Eligibility for Home Discharge | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | First Spontaneous Urine Voiding | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Rescue Anaesthesia/Analgesia | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | First Post-Operative Analgesia | ddMMMyyyy hh:mm | yy h xx min | |
| Skkk/ttt | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



# Listing 16.2.6.3 - Time to events and maximum level of sensory block

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Spinal Injection Date/time | Spinal Injection Event Date/time | | Time<br>to Event | Metameric<br>Level |
|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | Regression of Spinal Block | Date/time<br>ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Onset of Sensory Block | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Onset of Motor Block | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Readiness for Surgery | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Regression of Sensory Block | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Regression of Motor Block | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Unassisted Ambulation | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Maximum Level of Sensory Block | ddMMMyyyy hh:mm | yy h xx min | T8 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Regression of Two Dermatomers | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Eligibility for Home Discharge | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | First Spontaneous Urine Voiding | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Rescue Anaesthesia/Analgesia | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | First Post-Operative Analgesia | ddMMMyyyy hh:mm | yy h xx min | |
| Skkk/ttt | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



# Listing 16.2.6.3 - Time to events and maximum level of sensory block

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Spinal Injection Date/time | Spinal Injection Event Date/time | | Time<br>to Event | Metameric<br>Level |
|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | Regression of Spinal Block | Date/time<br>ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Onset of Sensory Block | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Onset of Motor Block | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Readiness for Surgery | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Regression of Sensory Block | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Regression of Motor Block | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Unassisted Ambulation | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Maximum Level of Sensory Block | ddMMMyyyy hh:mm | yy h xx min | T8 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Regression of Two Dermatomers | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Eligibility for Home Discharge | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | First Spontaneous Urine Voiding | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | Rescue Anaesthesia/Analgesia | ddMMMyyyy hh:mm | yy h xx min | |
| Sjjj/nnn | ddMMMyyyy hh:mm | First Post-Operative Analgesia | ddMMMyyyy hh:mm | yy h xx min | |
| Skkk/ttt | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



## Listing 16.2.6.4 - Effectiveness of anaesthesia and quality of spinal block

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Spinal Injection<br>Date/time | Assessment Date/time | Elapsed<br>Time | Parameter | Assessment |
|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Achievement of an Effective Anaesthesia | Y |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Quality of Spinal Block | Adequate Spinal Block |
| Skkk/ttt | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Achievement of an Effective Anaesthesia | N |
| Skkk/ttt | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Quality of Spinal Block | Inadequate Spinal Block |
| Snnn/xxx | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



## Listing 16.2.6.4 - Effectiveness of anaesthesia and quality of spinal block

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Spinal Injection<br>Date/time | Assessment Date/time | Elapsed<br>Time | Parameter | Assessment |
|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Achievement of an Effective Anaesthesia | Y |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Quality of Spinal Block | Adequate Spinal Block |
| Skkk/ttt | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Achievement of an Effective Anaesthesia | N |
| Skkk/ttt | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Quality of Spinal Block | Inadequate Spinal Block |
| Snnn/xxx | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



## Listing 16.2.6.4 - Effectiveness of anaesthesia and quality of spinal block

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Spinal Injection<br>Date/time | Assessment Date/time | Elapsed<br>Time | Parameter | Assessment |
|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Achievement of an Effective Anaesthesia | Y |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Quality of Spinal Block | Adequate Spinal Block |
| Skkk/ttt | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Achievement of an Effective Anaesthesia | N |
| Skkk/ttt | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Quality of Spinal Block | Inadequate Spinal Block |
| Snnn/xxx | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



## Listing 16.2.7.1 - Treatment-emergent adverse events

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | AE<br>Nr<br>/<br>FU<br>Nr | Verbatim /<br>Preferred Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> | Start or Follow-up Date/time / Start or Follow-up Day / End Date/time / End Day / Duration | IMP injection Date/time / Day / Time from IMP injection | Seriousness /<br>Severity /<br>Related to IMP /<br>Other relationship | Outcome /<br>Action taken with IMP /<br>Other action taken | Therapy required / Leading to discontinuation / Comments |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | 1 | Headache /<br>Headache /<br>Nervous system disorders | ddMMMyyyy hh:mm / Day j / Ongoing / / | ddMMMyyyy hh:mm /<br>Day j /<br>xx h xx min | N /<br>Moderate /<br>Not related /<br>Weather condition | Recovering/resolving / Not applicable / | Y /<br>N /<br> |
| Sjjj/nnn | 1/1 | Headache /<br>Headache /<br>Nervous system disorders | ddMMMyyyy hh:mm /<br>Day k /<br>ddMMMyyyy hh:mm /<br>Day k /<br>x h | ddMMMyyyy hh:mm /<br>Day j /<br>xx h xx min | N /<br>Mild /<br>Not related /<br>Weather condition | Recovered/resolved / Not applicable / | Y /<br>N /<br> |
| Skkk/ppp | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: MedDRA version 18.1 Program: Listings\c122-ae-lst.sas



## Listing 16.2.7.1 - Treatment-emergent adverse events

## Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | AE<br>Nr<br>/<br>FU<br>Nr | Verbatim /<br>Preferred Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> | Start or Follow-up Date/time / Start or Follow-up Day / End Date/time / End Day / Duration | IMP injection Date/time / Day / Time from IMP injection | Seriousness /<br>Severity /<br>Related to IMP /<br>Other relationship | Outcome / Action taken with IMP / Other action taken | Therapy required / Leading to discontinuation / Comments |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | 1 | Headache /<br>Headache /<br>Nervous system disorders | ddMMMyyyy hh:mm / Day j / Ongoing / / | ddMMMyyyy hh:mm /<br>Day j /<br>xx h xx min | N /<br>Moderate /<br>Not related /<br>Weather condition | Recovering/resolving / Not applicable / | Y /<br>N /<br> |
| Sjjj/nnn | 1/1 | Headache /<br>Headache /<br>Nervous system disorders | ddMMMyyyy hh:mm /<br>Day k /<br>ddMMMyyyy hh:mm /<br>Day k /<br>x h | ddMMMyyyy hh:mm /<br>Day j /<br>xx h xx min | N /<br>Mild /<br>Not related /<br>Weather condition | Recovered/resolved / Not applicable / | Y /<br>N /<br> |
| Skkk/ppp | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: MedDRA version 18.1 Program: Listings\c122-ae-lst.sas



## Listing 16.2.7.1 - Treatment-emergent adverse events

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | AE<br>Nr<br>/<br>FU<br>Nr | Verbatim /<br>Preferred Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> | Start or Follow-up Date/time / Start or Follow-up Day / End Date/time / End Day / Duration | IMP injection Date/time / Day / Time from IMP injection | Seriousness /<br>Severity /<br>Related to IMP /<br>Other relationship | Outcome / Action taken with IMP / Other action taken | Therapy required / Leading to discontinuation / Comments |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | 1 | Headache /<br>Headache /<br>Nervous system disorders | ddMMMyyyy hh:mm /<br>Day j /<br>Ongoing /<br>/ | ddMMMyyyy hh:mm /<br>Day j /<br>xx h xx min | N /<br>Moderate /<br>Not related /<br>Weather condition | Recovering/resolving / Not applicable / | Y /<br>N /<br> |
| Sjjj/nnn | 1/1 | Headache /<br>Headache /<br>Nervous system disorders | ddMMMyyyy hh:mm /<br>Day k /<br>ddMMMyyyy hh:mm /<br>Day k /<br>x h | ddMMMyyyy hh:mm /<br>Day j /<br>xx h xx min | N /<br>Mild /<br>Not related /<br>Weather condition | Recovered/resolved / Not applicable / | Y /<br>N /<br> |
| Skkk/ppp | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: MedDRA version 18.1 Program: Listings\c122-ae-lst.sas



## **Listing 16.2.7.2 - Pre-treatment adverse events**

## Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | AE<br>Nr | Verbatim /<br>Preferred Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> | Start Date/time /<br>End Date/time /<br>Duration | Seriousness /<br>Severity /<br>Related to IMP /<br>Other relationship | Outcome /<br>Action taken with IMP /<br>Other Action Taken | Therapy<br>required /<br>Leading to<br>discontinuation /<br>Comments |
|---|---|---|---|---|---|---|
| Sjjj/nnn | 1 | Headache / | ddMMMyyyy hh:mm / | N / | Recovered/resolved / | Y / |
| - | | Headache / | Day k / | Mild / | Not applicable / | N / |
| | | Nervous system disorders | ddMMMyyyy hh:mm /<br>Day k /<br>x h | Not related /<br>Weather condition | ` <u></u> | <del></del> |
| Skkk/ppp | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: MedDRA version 18.1 Program: Listings\c122-ae-lst.sas



## **Listing 16.2.7.2 - Pre-treatment adverse events**

## Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | AE<br>Nr | Verbatim /<br>Preferred Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> | Start Date/time /<br>End Date/time /<br>Duration | Seriousness / Severity / Related to IMP / Other relationship | Outcome /<br>Action taken with IMP /<br>Other Action Taken | Therapy<br>required /<br>Leading to<br>discontinuation /<br>Comments |
|---|---|---|---|---|---|---|
| Sjjj/nnn | 1 | Headache / | ddMMMyyyy hh:mm/ | N / | Recovered/resolved / | Y / |
| | | Headache / | Day k / | Mild / | Not applicable / | N / |
| | | Nervous system disorders | ddMMMyyyy hh:mm /<br>Day k /<br>x h | Not related /<br>Weather condition | | |
| Skkk/ppp | | ••• | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: MedDRA version 18.1 Program: Listings\c122-ae-lst.sas



## **Listing 16.2.7.2 - Pre-treatment adverse events**

## Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | AE<br>Nr | Verbatim /<br>Preferred Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> | Start Date/time /<br>End Date/time /<br>Duration | Seriousness /<br>Severity /<br>Related to IMP /<br>Other relationship | Outcome /<br>Action taken with IMP /<br>Other Action Taken | Therapy<br>required /<br>Leading to<br>discontinuation /<br>Comments |
|---|---|---|---|---|---|---|
| Sjjj/nnn | 1 | Headache / | ddMMMyyyy hh:mm / | N / | Recovered/resolved / | Y / |
| - | | Headache / | Day k / | Mild / | Not applicable / | N / |
| | | Nervous system disorders | ddMMMyyyy hh:mm /<br>Day k /<br>x h | Not related /<br>Weather condition | ` <u></u> | <del></del> |
| Skkk/ppp | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: MedDRA version 18.1 Program: Listings\c122-ae-lst.sas



# Listing 16.2.7.2 - Pre-treatment adverse events

## **Investigational Medicinal Product: Not Assigned**

| Subject AE<br>ID Nr | Verbatim /<br>Preferred Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> | Start Date/time /<br>End Date/time /<br>Duration | Seriousness /<br>Severity /<br>Related to IMP /<br>Other relationship | Outcome /<br>Action taken with IMP /<br>Other Action Taken | Therapy<br>required /<br>Leading to<br>discontinuation /<br>Comments |
|---|---|---|---|---|---|
| Sjjj/nnn 1 | Headache / | ddMMMyyyy hh:mm / | N / | Recovered/resolved / | Y / |
| 355 | Headache / | Day k / | Mild / | Not applicable / | N / |
| | Nervous system disorders | ddMMMyyyy hh:mm /<br>Day k /<br>x h | Not related / Weather condition | <u></u> | |
| Skkk/ppp | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: MedDRA version 18.1 Program: Listings\c122-ae-lst.sas



# Listing 16.2.7.2 - Pre-treatment adverse events

## **Investigational Medicinal Product: Not Treated**

| Subject AE<br>ID Nr | _ | Start Date/time /<br>End Date/time /<br>Duration | Seriousness /<br>Severity /<br>Related to IMP /<br>Other relationship | Outcome /<br>Action taken with IMP /<br>Other Action Taken | Therapy<br>required /<br>Leading to<br>discontinuation /<br>Comments |
|---|---|---|---|---|---|
| Sjjj/nnn 1 | Headache / | ddMMMyyyy hh:mm / | N / | Recovered/resolved/ | Y / |
| | Headache / | Day k / | Mild / | Not applicable / | N / |
| | Nervous system disorders | ddMMMyyyy hh:mm /<br>Day k /<br>x h | Not related / Weather condition | <u></u> | |
| Skkk/ppp | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: MedDRA version 18.1 Program: Listings\c122-ae-lst.sas



## Listing 16.2.9.1 - Vital signs

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Time Point | Assessment<br>Date/time | Parameter | Value | Normal Range | Interpretation <sup>1</sup> |
|---|---|---|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure | xxx mmHg | 100-139 mmHg | X |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Diastolic Blood Pressure | xxx mmHg | 50-89 mmHg | X |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Oxygen Saturation | xxx.x % | >= 95 % | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Systolic Blood Pressure | xxx mmHg | 100-139 mmHg | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Diastolic Blood Pressure | xxx mmHg | 50-89 mmHg | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Oxygen Saturation | xxx.x % | >= 95 % | X |
| Sjjj/nnn | Discharge | ddMMMyyyy hh:mm | Systolic Blood Pressure | xxx mmHg | 100-139 mmHg | X |
| Sjjj/nnn | Discharge | ddMMMyyyy hh:mm | Diastolic Blood Pressure | xxx mmHg | 50-89 mmHg | X |
| Sjjj/nnn | Discharge | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Discharge | ddMMMyyyy hh:mm | Oxygen Saturation | XXX.X % | >= 95 % | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Systolic Blood Pressure | xxx mmHg | 100-139 mmHg | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Diastolic Blood Pressure | xxx mmHg | 50-89 mmHg | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Oxygen Saturation | xxx.x % | >= 95 % | X |
| Skkk/xxx | | | | | >= 95 % | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: N=Normal, NCS=Abnormal, Not Clinically Significant, CS=Abnormal, Clinically Significant

Program: Listings\c122-vs-lst.sas



## Listing 16.2.9.1 - Vital signs

## Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Time Point | Assessment<br>Date/time | Parameter | Value | Normal Range | Interpretation <sup>1</sup> |
|---|---|---|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure | xxx mmHg | 100-139 mmHg | X |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Diastolic Blood Pressure | xxx mmHg | 50-89 mmHg | X |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Oxygen Saturation | xxx.x % | >= 95 % | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Systolic Blood Pressure | xxx mmHg | 100-139 mmHg | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Diastolic Blood Pressure | xxx mmHg | 50-89 mmHg | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Oxygen Saturation | xxx.x % | >= 95 % | X |
| Sjjj/nnn | Discharge | ddMMMyyyy hh:mm | Systolic Blood Pressure | xxx mmHg | 100-139 mmHg | X |
| Sjjj/nnn | Discharge | ddMMMyyyy hh:mm | Diastolic Blood Pressure | xxx mmHg | 50-89 mmHg | X |
| Sjjj/nnn | Discharge | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Discharge | ddMMMyyyy hh:mm | Oxygen Saturation | XXX.X % | >= 95 % | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Systolic Blood Pressure | xxx mmHg | 100-139 mmHg | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Diastolic Blood Pressure | xxx mmHg | 50-89 mmHg | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Oxygen Saturation | xxx.x % | >= 95 % | X |
| Skkk/xxx | | | | | >= 95 % | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: N=Normal, NCS=Abnormal, Not Clinically Significant, CS=Abnormal, Clinically Significant

Program: Listings\c122-vs-lst.sas



Listing 16.2.9.1 - Vital signs

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Time Point | Assessment<br>Date/time | Parameter | Value | Normal Range | Interpretation <sup>1</sup> |
|---|---|---|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure | xxx mmHg | 100-139 mmHg | X |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Diastolic Blood Pressure | xxx mmHg | 50-89 mmHg | X |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Oxygen Saturation | xxx.x % | >= 95 % | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Systolic Blood Pressure | xxx mmHg | 100-139 mmHg | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Diastolic Blood Pressure | xxx mmHg | 50-89 mmHg | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Oxygen Saturation | xxx.x % | >= 95 % | X |
| Sjjj/nnn | Discharge | ddMMMyyyy hh:mm | Systolic Blood Pressure | xxx mmHg | 100-139 mmHg | X |
| Sjjj/nnn | Discharge | ddMMMyyyy hh:mm | Diastolic Blood Pressure | xxx mmHg | 50-89 mmHg | X |
| Sjjj/nnn | Discharge | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Discharge | ddMMMyyyy hh:mm | Oxygen Saturation | XXX.X % | >= 95 % | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Systolic Blood Pressure | xxx mmHg | 100-139 mmHg | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Diastolic Blood Pressure | xxx mmHg | 50-89 mmHg | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Oxygen Saturation | xxx.x % | >= 95 % | X |
| Skkk/xxx | | | | | >= 95 % | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: N=Normal, NCS=Abnormal, Not Clinically Significant, CS=Abnormal, Clinically Significant

Program: Listings\c122-vs-lst.sas



## Listing 16.2.9.1 - Vital signs

**Investigational Medicinal Product: Not Assigned** 

| Subject<br>ID | Time Point | Assessment Date/time | Parameter | Value | Normal Range | Interpretation <sup>1</sup> |
|---|---|---|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure | xxx mmHg | 100-139 mmHg | X |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Diastolic Blood Pressure | xxx mmHg | 50-89 mmHg | X |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Oxygen Saturation | xxx.x % | >= 95 % | X |
| Skkk/xxx | | | | | >= 95 % | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: N=Normal, NCS=Abnormal, Not Clinically Significant, CS=Abnormal, Clinically Significant

Program: Listings\c122-vs-lst.sas


#### Listing 16.2.9.1 - Vital signs

**Investigational Medicinal Product: Not Treated** 

| Subject<br>ID | Time Point | Assessment<br>Date/time | Parameter | Value | Normal Range | Interpretation <sup>1</sup> |
|---|---|---|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Systolic Blood Pressure | xxx mmHg | 100-139 mmHg | X |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Diastolic Blood Pressure | xxx mmHg | 50-89 mmHg | X |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Oxygen Saturation | xxx.x % | >= 95 % | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Systolic Blood Pressure | xxx mmHg | 100-139 mmHg | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Diastolic Blood Pressure | xxx mmHg | 50-89 mmHg | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Baseline | ddMMMyyyy hh:mm | Oxygen Saturation | xxx.x % | >= 95 % | X |
| Skkk/xxx | | | | | >= 95 % | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: N=Normal, NCS=Abnormal, Not Clinically Significant, CS=Abnormal, Clinically Significant

Program: Listings  $\c 122$ -vs-lst.sas



#### **Listing 16.2.9.2 - ECG**

# Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Time Point | Assessment Date/time | Parameter | Value | Normal Range | Interpretation <sup>1</sup> |
|---|---|---|---|---|---|---|
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Investigator's Interpretation | Abnormal, Not Clinically Significant | | |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Clinically Significant Abnormalities | XXXXX | | |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | PR Interval | xxx msec | 100-220 msec | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | QRS Duration | xxx msec | <= 120 msec | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | QT Interval | xxx msec | <= 500 msec | X |
| Skkk/xxx | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: N=Normal, NCS=Abnormal, Not Clinically Significant, CS=Abnormal, Clinically Significant

Program: Listings\c122-eg-lst.sas



#### **Listing 16.2.9.2 - ECG**

# Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Time Point | Assessment Date/time | Parameter | Value | Normal Range | Interpretation <sup>1</sup> |
|---|---|---|---|---|---|---|
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Investigator's Interpretation | Abnormal, Not Clinically Significant | | |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Clinically Significant Abnormalities | XXXXX | | |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | PR Interval | xxx msec | 100-220 msec | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | QRS Duration | xxx msec | <= 120 msec | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | QT Interval | xxx msec | <= 500 msec | X |
| Skkk/xxx | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: N=Normal, NCS=Abnormal, Not Clinically Significant, CS=Abnormal, Clinically Significant

Program: Listings\c122-eg-lst.sas



#### **Listing 16.2.9.2 - ECG**

# Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Time Point | Assessment Date/time | Parameter | Value | Normal Range | Interpretation <sup>1</sup> |
|---|---|---|---|---|---|---|
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Investigator's Interpretation | Abnormal, Not Clinically Significant | | |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Clinically Significant Abnormalities | XXXXX | | |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | PR Interval | xxx msec | 100-220 msec | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | QRS Duration | xxx msec | <= 120 msec | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | QT Interval | xxx msec | <= 500 msec | X |
| Skkk/xxx | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: N=Normal, NCS=Abnormal, Not Clinically Significant, CS=Abnormal, Clinically Significant

Program: Listings\c122-eg-lst.sas



#### **Listing 16.2.9.2 - ECG**

#### **Investigational Medicinal Product: Not Treated**

| Subject<br>ID | Time Point | Assessment<br>Date/time | Parameter | Value | Normal Range | Interpretation <sup>1</sup> |
|---|---|---|---|---|---|---|
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Investigator's Interpretation | Abnormal, Not Clinically Significant | | |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Clinically Significant Abnormalities | xxxxx | | |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | Heart Rate | xxx beats/min | 50-90 beats/min | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | PR Interval | xxx msec | 100-220 msec | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | QRS Duration | xxx msec | <= 120 msec | X |
| Sjjj/nnn | Unscheduled | ddMMMyyyy hh:mm | QT Interval | xxx msec | <= 500 msec | X |
| Skkk/xxx | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: N=Normal, NCS=Abnormal, Not Clinically Significant, CS=Abnormal, Clinically Significant

Program: Listings\c122-eg-lst.sas



#### Listing 16.2.9.3 - Pain assessment at the site of injection and at the site of surgery

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Spinal Injection<br>Date/time | Time Point | Assessment Date/time | Elapsed<br>Time | Parameter | Pain<br>Assessment <sup>1</sup> |
|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | Immediately after regression of spinal block | ddMMMyyyy hh:mm | yy h xx min | Pain at the Injection Site | 5 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Discharge | ddMMMyyyy hh:mm | yy h xx min | Pain at the Injection Site | 5 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Pain at the Injection Site | 5 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 7±1 | ddMMMyyyy hh:mm | yy days yy h xx min | Pain at the Injection Site | 5 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Immediately after regression of spinal block | ddMMMyyyy hh:mm | yy h xx min | Pain at the Surgery Site | 7 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Discharge | ddMMMyyyy hh:mm | yy h xx min | Pain at the Surgery Site | 7 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Pain at the Surgery Site | 7 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 7±1 | ddMMMyyyy hh:mm | yy days yy h xx min | Pain at the Surgery Site | 7 |
| Snnn/xxx | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: Pain was assessed according to a numerical rating scale ranging from 0 (no pain) to 10 (worst imaginable pain)

 $Program: Listings \verb|\c122-qs-lst.sas|$ 



#### Listing 16.2.9.3 - Pain assessment at the site of injection and at the site of surgery

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Spinal Injection<br>Date/time | Time Point | Assessment Date/time | Elapsed<br>Time | Parameter | Pain<br>Assessment <sup>1</sup> |
|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | Immediately after regression of spinal block | ddMMMyyyy hh:mm | yy h xx min | Pain at the Injection Site | 5 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Discharge | ddMMMyyyy hh:mm | yy h xx min | Pain at the Injection Site | 5 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Pain at the Injection Site | 5 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 7±1 | ddMMMyyyy hh:mm | yy days yy h xx min | Pain at the Injection Site | 5 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Immediately after regression of spinal block | ddMMMyyyy hh:mm | yy h xx min | Pain at the Surgery Site | 7 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Discharge | ddMMMyyyy hh:mm | yy h xx min | Pain at the Surgery Site | 7 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Pain at the Surgery Site | 7 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 7±1 | ddMMMyyyy hh:mm | yy days yy h xx min | Pain at the Surgery Site | 7 |
| Snnn/xxx | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: Pain was assessed according to a numerical rating scale ranging from 0 (no pain) to 10 (worst imaginable pain)

 $Program: Listings \verb|\c122-qs-lst.sas|$ 



#### Listing 16.2.9.3 - Pain assessment at the site of injection and at the site of surgery

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Spinal Injection<br>Date/time | Time Point | Assessment Date/time | Elapsed<br>Time | Parameter | Pain<br>Assessment <sup>1</sup> |
|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | Immediately after regression of spinal block | ddMMMyyyy hh:mm | yy h xx min | Pain at the Injection Site | 5 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Discharge | ddMMMyyyy hh:mm | yy h xx min | Pain at the Injection Site | 5 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Pain at the Injection Site | 5 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 7±1 | ddMMMyyyy hh:mm | yy days yy h xx min | Pain at the Injection Site | 5 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Immediately after regression of spinal block | ddMMMyyyy hh:mm | yy h xx min | Pain at the Surgery Site | 7 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Discharge | ddMMMyyyy hh:mm | yy h xx min | Pain at the Surgery Site | 7 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Pain at the Surgery Site | 7 |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 7±1 | ddMMMyyyy hh:mm | yy days yy h xx min | Pain at the Surgery Site | 7 |
| Snnn/xxx | | | | | | ••• |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: Pain was assessed according to a numerical rating scale ranging from 0 (no pain) to 10 (worst imaginable pain)

 $Program: Listings \verb|\c122-qs-lst.sas|$ 



**Listing 16.2.9.4 - Transient neurological symptoms** 

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Spinal Injection<br>Date/time | Time Point | Questionnaire<br>Date/time | Elapsed<br>Time | Parameter | Assessment |
|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Transient Neurological Symptoms | N |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Was the Patient Feeling Good? | N |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Reported Problems | Nausea/Vomiting |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Unusual Sensations? | Y |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Symptoms | Burning, Tingling |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Location of Symptoms | Thighs anterior, Lower limbs |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Laterality of Symptoms | Bilateral |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Previous Experience of Such Symptoms? | N |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 7±1 | ddMMMyyyy hh:mm | zz days yy h xx min | Transient Neurological Symptoms | N |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 7±1 | ddMMMyyyy hh:mm | zz days yy h xx min | Was the Patient Feeling Good? | Y |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 7±1 | ddMMMyyyy hh:mm | zz days yy h xx min | <b>Unusual Sensations?</b> | N |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



**Listing 16.2.9.4 - Transient neurological symptoms** 

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Spinal Injection<br>Date/time | Time Point | Questionnaire<br>Date/time | Elapsed<br>Time | Parameter | Assessment |
|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Transient Neurological Symptoms | N |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Was the Patient Feeling Good? | N |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Reported Problems | Nausea/Vomiting |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Unusual Sensations? | Y |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Symptoms | Burning, Tingling |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Location of Symptoms | Thighs anterior, Lower limbs |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Laterality of Symptoms | Bilateral |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Previous Experience of Such Symptoms? | N |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 7±1 | ddMMMyyyy hh:mm | zz days yy h xx min | Transient Neurological Symptoms | N |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 7±1 | ddMMMyyyy hh:mm | zz days yy h xx min | Was the Patient Feeling Good? | Y |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 7±1 | ddMMMyyyy hh:mm | zz days yy h xx min | <b>Unusual Sensations?</b> | N |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



**Listing 16.2.9.4 - Transient neurological symptoms** 

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Spinal Injection<br>Date/time | Time Point | Questionnaire<br>Date/time | Elapsed<br>Time | Parameter | Assessment |
|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Transient Neurological Symptoms | N |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Was the Patient Feeling Good? | N |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Reported Problems | Nausea/Vomiting |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Unusual Sensations? | Y |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Symptoms | Burning, Tingling |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Location of Symptoms | Thighs anterior, Lower limbs |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Laterality of Symptoms | Bilateral |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 2 | ddMMMyyyy hh:mm | yy h xx min | Previous Experience of Such Symptoms? | N |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 7±1 | ddMMMyyyy hh:mm | zz days yy h xx min | Transient Neurological Symptoms | N |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 7±1 | ddMMMyyyy hh:mm | zz days yy h xx min | Was the Patient Feeling Good? | Y |
| Sjjj/nnn | ddMMMyyyy hh:mm | Day 7±1 | ddMMMyyyy hh:mm | zz days yy h xx min | Unusual Sensations? | N |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



# **Listing 16.2.9.5 - Modified Aldrete's scoring scale**

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Spinal Injection<br>Date/time | Assessment<br>Date/time | Elapsed<br>Time | Parameter | Assessment |
|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Activity | 2 - Able to move 4 extremities voluntarily or on command |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Respiration | 2 - Able to breathe deeply and cough freely |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Circulation | 2 - Blood pressure $\pm$ 20% of pre-anaesthetic level |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Consciousness | 2 - Fully awake |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | O <sub>2</sub> saturation | 2 - Able to maintain $O_2$ saturation > 92% on room air |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Dressing | 2 - Dry and clean |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Pain | 2 - Pain free |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Ambulation | 2 - Able to stand up and walk straight |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Fasting-feeding | 2 - Able to drink fluids |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Urine output | 2 - Has voided |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Total Score | 20 |
| Snnn/xxx | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



# **Listing 16.2.9.5 - Modified Aldrete's scoring scale**

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Spinal Injection<br>Date/time | Assessment<br>Date/time | Elapsed<br>Time | Parameter | Assessment |
|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Activity | 2 - Able to move 4 extremities voluntarily or on command |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Respiration | 2 - Able to breathe deeply and cough freely |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Circulation | 2 - Blood pressure $\pm$ 20% of pre-anaesthetic level |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Consciousness | 2 - Fully awake |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | O <sub>2</sub> saturation | 2 - Able to maintain $O_2$ saturation > 92% on room air |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Dressing | 2 - Dry and clean |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Pain | 2 - Pain free |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Ambulation | 2 - Able to stand up and walk straight |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Fasting-feeding | 2 - Able to drink fluids |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Urine output | 2 - Has voided |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Total Score | 20 |
| Snnn/xxx | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



# **Listing 16.2.9.5 - Modified Aldrete's scoring scale**

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Spinal Injection<br>Date/time | Assessment<br>Date/time | Elapsed<br>Time | Parameter | Assessment |
|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Activity | 2 - Able to move 4 extremities voluntarily or on command |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Respiration | 2 - Able to breathe deeply and cough freely |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Circulation | 2 - Blood pressure $\pm$ 20% of pre-anaesthetic level |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Consciousness | 2 - Fully awake |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | O <sub>2</sub> saturation | 2 - Able to maintain $O_2$ saturation > 92% on room air |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Dressing | 2 - Dry and clean |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Pain | 2 - Pain free |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Ambulation | 2 - Able to stand up and walk straight |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Fasting-feeding | 2 - Able to drink fluids |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Urine output | 2 - Has voided |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Total Score | 20 |
| Snnn/xxx | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



# **Listing 16.2.9.5 - Modified Aldrete's scoring scale**

**Investigational Medicinal Product: Not Treated** 

| Subject<br>ID | Spinal Injection<br>Date/time | Assessment Date/time | Elapsed<br>Time | Parameter | Assessment |
|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Activity | 2 - Able to move 4 extremities voluntarily or on command |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Respiration | 2 - Able to breathe deeply and cough freely |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Circulation | 2 - Blood pressure $\pm$ 20% of pre-anaesthetic level |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Consciousness | 2 - Fully awake |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | O <sub>2</sub> saturation | 2 - Able to maintain $O_2$ saturation > 92% on room air |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Dressing | 2 - Dry and clean |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Pain | 2 - Pain free |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Ambulation | 2 - Able to stand up and walk straight |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Fasting-feeding | 2 - Able to drink fluids |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Urine output | 2 - Has voided |
| Sjjj/nnn | ddMMMyyyy hh:mm | ddMMMyyyy hh:mm | yy h xx min | Total Score | 20 |
| Snnn/xxx | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-qs-lst.sas



#### Listing 16.2.10.1 - Medical and surgical history

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Date of History<br>Collection | Verbatim /<br>Preferrec Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> | Date of<br>Diagnosis/<br>Surgery | Date of<br>Resolution<br>(Ongoing) |
|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy | Pollen allergy /<br>Seasonal allergy /<br>Immune system disorders | MMMyyyy | Ongoing |
| Sjjj/nnn | ddMMMyyyy | Appendectomy / Appendicectomy / Surgical and medical procedures | уууу | |
| Sjjj/nnn | ddMMMyyyy | Appendectomy / Appendicectomy / Surgical and medical procedures | уууу | |
| Skkk/xxx | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: N=Normal, NCS=Abnormal, Not Clinically Significant, CS=Abnormal, Clinically Significant

Program: Listings\c122-mh-lst.sas



#### Listing 16.2.10.1 - Medical and surgical history

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Date of History<br>Collection | Verbatim /<br>Preferrec Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> | Date of<br>Diagnosis/<br>Surgery | Date of<br>Resolution<br>(Ongoing) |
|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy | Pollen allergy /<br>Seasonal allergy /<br>Immune system disorders | MMMyyyy | Ongoing |
| Sjjj/nnn | ddMMMyyyy | Appendectomy / Appendicectomy / Surgical and medical procedures | уууу | |
| Sjjj/nnn | ddMMMyyyy | Appendectomy / Appendicectomy / Surgical and medical procedures | уууу | |
| Skkk/xxx | | <b></b> | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: N=Normal, NCS=Abnormal, Not Clinically Significant, CS=Abnormal, Clinically Significant

Program: Listings\c122-mh-lst.sas



#### Listing 16.2.10.1 - Medical and surgical history

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Date of History<br>Collection | Verbatim /<br>Preferrec Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> | Date of<br>Diagnosis/<br>Surgery | Date of<br>Resolution<br>(Ongoing) |
|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy | Pollen allergy /<br>Seasonal allergy /<br>Immune system disorders | MMMyyyy | Ongoing |
| Sjjj/nnn | ddMMMyyyy | Appendectomy / Appendicectomy / Surgical and medical procedures | уууу | |
| Sjjj/nnn | ddMMMyyyy | Appendectomy / Appendicectomy / Surgical and medical procedures | уууу | |
| Skkk/xxx | | <b></b> | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: N=Normal, NCS=Abnormal, Not Clinically Significant, CS=Abnormal, Clinically Significant

Program: Listings\c122-mh-lst.sas



#### Listing 16.2.10.1 - Medical and surgical history

**Investigational Medicinal Product: Not Assigned** 

| Subject<br>ID | Date of History<br>Collection | Verbatim /<br>Preferrec Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> | Date of<br>Diagnosis/<br>Surgery | Date of<br>Resolution<br>(Ongoing) |
|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy | Pollen allergy /<br>Seasonal allergy /<br>Immune system disorders | МММуууу | Ongoing |
| Sjjj/nnn | ddMMMyyyy | Appendectomy / Appendicectomy / Surgical and medical procedures | уууу | |
| Sjjj/nnn | ddMMMyyyy | Appendectomy / Appendicectomy / Surgical and medical procedures | уууу | |
| Skkk/xxx | | <b></b> | | ••• |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: N=Normal, NCS=Abnormal, Not Clinically Significant, CS=Abnormal, Clinically Significant

Program: Listings\c122-mh-lst.sas



#### Listing 16.2.10.1 - Medical and surgical history

**Investigational Medicinal Product: Not Treated** 

| Subject<br>ID | Date of History<br>Collection | Verbatim /<br>Preferrec Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> | Date of<br>Diagnosis/<br>Surgery | Date of<br>Resolution<br>(Ongoing) |
|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy | Pollen allergy /<br>Seasonal allergy /<br>Immune system disorders | MMMyyyy | Ongoing |
| Sjjj/nnn | ddMMMyyyy | Appendectomy / Appendicectomy / Surgical and medical procedures | уууу | |
| Sjjj/nnn | ddMMMyyyy | Appendectomy / Appendicectomy / Surgical and medical procedures | уууу | |
| Skkk/xxx | | <b></b> | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: N=Normal, NCS=Abnormal, Not Clinically Significant, CS=Abnormal, Clinically Significant

Program: Listings\c122-mh-lst.sas



# Listing 16.2.10.2 - Physical examination

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Time Point | Date of History<br>Collection | ASA<br>Physical<br>Status | Investigator's<br>Interpretation | Clinically Significant Findings /<br>Preferrec Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> |
|---|---|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy | III | Abnormal, Not Clinically Significant | |
| Skkk/ppp | Screening | ddMMMyyyy | II | Abnormal, Clinically Significant | Cardiac disorder /<br>Cardiac disorder /<br>Cardiac disorders |
| Snnn/xxx | Screening | ••• | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-pe-lst.sas



#### Listing 16.2.10.2 - Physical examination

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Time Point | Date of History<br>Collection | ASA<br>Physical<br>Status | Investigator's<br>Interpretation | Clinically Significant Findings /<br>Preferrec Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> |
|---|---|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy | III | Abnormal, Not Clinically Significant | |
| Skkk/ppp | Screening | ddMMMyyyy | II | Abnormal, Clinically Significant | Cardiac disorder /<br>Cardiac disorder /<br>Cardiac disorders |
| Snnn/xxx | Screening | ••• | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-pe-lst.sas



# Listing 16.2.10.2 - Physical examination

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Time Point | Date of History<br>Collection | ASA<br>Physical<br>Status | Investigator's<br>Interpretation | Clinically Significant Findings /<br>Preferrec Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> |
|---|---|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy | III | Abnormal, Not Clinically Significant | |
| Skkk/ppp | Screening | ddMMMyyyy | II | Abnormal, Clinically Significant | Cardiac disorder /<br>Cardiac disorder /<br>Cardiac disorders |
| Snnn/xxx | Screening | ••• | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-pe-lst.sas



# Listing 16.2.10.2 - Physical examination

**Investigational Medicinal Product: Not Assigned** 

| Subject<br>ID | Time Point | Date of History<br>Collection | ASA<br>Physical<br>Status | Investigator's<br>Interpretation | Clinically Significant Findings /<br>Preferrec Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> |
|---|---|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy | III | Abnormal, Not Clinically Significant | |
| Skkk/ppp | Screening | ddMMMyyyy | II | Abnormal, Clinically Significant | Cardiac disorder /<br>Cardiac disorder /<br>Cardiac disorders |
| Snnn/xxx | Screening | ••• | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-pe-lst.sas



# Listing 16.2.10.2 - Physical examination

**Investigational Medicinal Product: Not Treated** 

| Subject<br>ID | Time Point | Date of History<br>Collection | ASA<br>Physical<br>Status | Investigator's<br>Interpretation | Clinically Significant Findings /<br>Preferrec Term <sup>1</sup> /<br>System Organ Class <sup>1</sup> |
|---|---|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy | III | Abnormal, Not Clinically Significant | |
| Skkk/ppp | Screening | ddMMMyyyy | II | Abnormal, Clinically Significant | Cardiac disorder /<br>Cardiac disorder /<br>Cardiac disorders |
| Snnn/xxx | Screening | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-pe-lst.sas



# Listing 16.2.10.3 - Prior and concomitant medications

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | CM<br>Nr | Prior or<br>Concomitant | Verbatim /<br>Indication /<br>Related to<br>AE MH SH <sup>1</sup> | Standardised name <sup>2</sup> / Active ingredients <sup>2</sup> / ATC level 4 <sup>2</sup> | Dose | Start date/time /<br>End date/time<br>(Ongoing) | Frequency /<br>Dosage form /<br>Route |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | 1 | Concomitant | Paracetamol /<br>Analgesia /<br>AE Nr. 1 | Paracetamol / Paracetamol / Anilides | 500 mg | ddMMMyyyy<br>hh:mm /<br>ddMMMyyyy<br>hh:mm | Once /<br>Tablet /<br>Oral |
| Sjjj/nnn | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: AE=Adverve Event, MH=Medical History, SH=Surgical History

Note 2: WHODDE September 1, 2015 Program: Listings\k294-cm-lst.sas



# Listing 16.2.10.3 - Prior and concomitant medications

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | CM<br>Nr | Prior or<br>Concomitant | Verbatim /<br>Indication /<br>Related to<br>AE MH SH <sup>1</sup> | Standardised name <sup>2</sup> / Active ingredients <sup>2</sup> / ATC level 4 <sup>2</sup> | Dose | Start date/time /<br>End date/time<br>(Ongoing) | Frequency /<br>Dosage form /<br>Route |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | 1 | Concomitant | Paracetamol /<br>Analgesia /<br>AE Nr. 1 | Paracetamol / Paracetamol / Anilides | 500 mg | ddMMMyyyy<br>hh:mm /<br>ddMMMyyyy<br>hh:mm | Once /<br>Tablet /<br>Oral |
| Sjjj/nnn | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: AE=Adverve Event, MH=Medical History, SH=Surgical History

Note 2: WHODDE September 1, 2015 Program: Listings\k294-cm-lst.sas



# Listing 16.2.10.3 - Prior and concomitant medications

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | CM<br>Nr | Prior or<br>Concomitant | Verbatim /<br>Indication /<br>Related to<br>AE MH SH <sup>1</sup> | Standardised name <sup>2</sup> / Active ingredients <sup>2</sup> / ATC level 4 <sup>2</sup> | Dose | Start date/time /<br>End date/time<br>(Ongoing) | Frequency /<br>Dosage form /<br>Route |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | 1 | Concomitant | Paracetamol / Analgesia / AE Nr. 1 | Paracetamol / Paracetamol / Anilides | 500 mg | ddMMMyyyy<br>hh:mm/<br>ddMMMyyyy<br>hh:mm | Once /<br>Tablet /<br>Oral |
| Sjjj/nnn | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: AE=Adverve Event, MH=Medical History, SH=Surgical History

Note 2: WHODDE September 1, 2015 Program: Listings\k294-cm-lst.sas



# Listing 16.2.10.3 - Prior and concomitant medications

**Investigational Medicinal Product: Not Assigned** 

| Subject<br>ID | CM<br>Nr | Prior or<br>Concomitant | Verbatim /<br>Indication /<br>Related to<br>AE MH SH <sup>1</sup> | Standardised name <sup>2</sup> / Active ingredients <sup>2</sup> / ATC level 4 <sup>2</sup> | Dose | Start date/time /<br>End date/time<br>(Ongoing) | Frequency /<br>Dosage form /<br>Route |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | 1 | Concomitant | Ringer acetate / Fluid therapy / | Ringer acetate / Calcium chloride/Potassium chloride / Electrolyte solutions | 500 mL | ddMMMyyyy<br>hh:mm /<br>ddMMMyyyy<br>hh:mm | Continuous / Injection, solution / Intravenous |
| Sjjj/nnn | | •• | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: AE=Adverve Event, MH=Medical History, SH=Surgical History

Note 2: WHODDE September 1, 2015 Program: Listings\k294-cm-lst.sas



# Listing 16.2.10.3 - Prior and concomitant medications

**Investigational Medicinal Product: Not Treated** 

| Subject<br>ID | CM<br>Nr | Prior or<br>Concomitant | Verbatim /<br>Indication /<br>Related to<br>AE MH SH <sup>1</sup> | Standardised name <sup>2</sup> / Active ingredients <sup>2</sup> / ATC level 4 <sup>2</sup> | Dose | Start date/time /<br>End date/time<br>(Ongoing) | Frequency /<br>Dosage form /<br>Route |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | 1 | Concomitant | Ringer acetate /<br>Fluid therapy / | Ringer acetate / Calcium chloride/Potassium chloride / Electrolyte solutions | 500 mL | ddMMMyyyy<br>hh:mm /<br>ddMMMyyyy<br>hh:mm | Continuous / Injection, solution / Intravenous |
| Sjjj/nnn | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Note 1: AE=Adverve Event, MH=Medical History, SH=Surgical History

Note 2: WHODDE September 1, 2015 Program: Listings\k294-cm-lst.sas



# Listing 16.2.10.4 - Subjects study visits

Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Visit 1<br>Screening<br>Day -14/1<br>Date (Day) | Visit 2<br>Day 1<br>Date (Day) | Final<br>Visit<br>Date (Day) | Early<br>Termination<br>Visit<br>Date (Day) | Follow-up<br>Day 2<br>Date (Day) | Follow-up<br>Day 7±1<br>Date (Day) | Additional<br>Assessment<br>Date (Day) |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy (j) | ddMMMyyyy (j) | ddMMMyyyy (j) | ddMMMyyyy (j) | ddMMMyyyy (j) | ddMMMyyyy (j) | ddMMMyyyy (j) |
| Skkk/xxx | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-sv-lst.sas



# Listing 16.2.10.4 - Subjects study visits

Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Visit 1<br>Screening<br>Day -14/1<br>Date (Day) | Visit 2<br>Day 1<br>Date (Day) | Final<br>Visit<br>Date (Day) | Early<br>Termination<br>Visit<br>Date (Day) | Follow-up<br>Day 2<br>Date (Day) | Follow-up<br>Day 7±1<br>Date (Day) | Additional<br>Assessment<br>Date (Day) |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy (j) | ddMMMyyyy (j) | ddMMMyyyy (j) | ddMMMyyyy (j) | ddMMMyyyy (j) | ddMMMyyyy (j) | ddMMMyyyy (j) |
| Skkk/xxx | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-sv-lst.sas



# Listing 16.2.10.4 - Subjects study visits

Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Visit 1<br>Screening<br>Day -14/1<br>Date (Day) | Visit 2<br>Day 1<br>Date (Day) | Final<br>Visit<br>Date (Day) | Early<br>Termination<br>Visit<br>Date (Day) | Follow-up<br>Day 2<br>Date (Day) | Follow-up<br>Day 7±1<br>Date (Day) | Additional<br>Assessment<br>Date (Day) |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy (j) | ddMMMyyyy (j) | ddMMMyyyy (j) | ddMMMyyyy (j) | ddMMMyyyy (j) | ddMMMyyyy (j) | ddMMMyyyy (j) |
| Skkk/xxx | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-sv-lst.sas



# Listing 16.2.10.4 - Subjects study visits

**Investigational Medicinal Product: Not Assigned** 

| Subject<br>ID | Visit 1<br>Screening<br>Day -14/1<br>Date (Day) | Visit 2<br>Day 1<br>Date (Day) | Final<br>Visit<br>Date (Day) | Early<br>Termination<br>Visit<br>Date (Day) | Follow-up<br>Day 2<br>Date (Day) | Follow-up<br>Day 7±1<br>Date (Day) | Additional<br>Assessment<br>Date (Day) |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy (j) | | | | | | |
| Skkk/xxx | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-sv-lst.sas



# Listing 16.2.10.4 - Subjects study visits

# **Investigational Medicinal Product: Not Treated**

| Subject<br>ID | Visit 1<br>Screening<br>Day -14/1<br>Date (Day) | Visit 2<br>Day 1<br>Date (Day) | Final<br>Visit<br>Date (Day) | Early<br>Termination<br>Visit<br>Date (Day) | Follow-up<br>Day 2<br>Date (Day) | Follow-up<br>Day 7±1<br>Date (Day) | Additional<br>Assessment<br>Date (Day) |
|---|---|---|---|---|---|---|---|
| Sjjj/nnn | ddMMMyyyy (j) | ddMMMyyyy (j) | | | | | |
| Skkk/xxx | | | | | | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-sv-lst.sas



# Listing 16.2.10.5 - Pregnancy test

# Investigational Medicinal Product: Chloroprocaine 1% - 30 mg

| Subject<br>ID | Time Point | Urine Collection<br>Date/time | Pregnancy Test<br>Result |
|---|---|---|---|
| | - | | Result |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Negative |
| Skkk/ppp | Screening | ddMMMyyyy hh:mm | Negative |
| Snnn/xxx | Screening | <b></b> | <b></b> |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-xt-lst.sas



# Listing 16.2.10.5 - Pregnancy test

# Investigational Medicinal Product: Chloroprocaine 1% - 40 mg

| Subject<br>ID | Time Point | Urine Collection Date/time | Pregnancy Test<br>Result |
|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Negative |
| Skkk/ppp | Screening | ddMMMyyyy hh:mm | Negative |
| Snnn/xxx | Screening | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-xt-lst.sas



# Listing 16.2.10.5 - Pregnancy test

# Investigational Medicinal Product: Chloroprocaine 1% - 50 mg

| Subject<br>ID | Time Point | Urine Collection<br>Date/time | Pregnancy Test<br>Result |
|---|---|---|---|
| | - | | Result |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Negative |
| Skkk/ppp | Screening | ddMMMyyyy hh:mm | Negative |
| Snnn/xxx | Screening | <b></b> | <b></b> |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-xt-lst.sas



# Listing 16.2.10.5 - Pregnancy test

**Investigational Medicinal Product: Not Assigned** 

| Subject<br>ID | Time Point | Urine Collection<br>Date/time | Pregnancy Test<br>Result |
|---|---|---|---|
| | - | | Result |
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Negative |
| Skkk/ppp | Screening | ddMMMyyyy hh:mm | Negative |
| Snnn/xxx | Screening | <b></b> | <b></b> |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-xt-lst.sas



# Listing 16.2.10.5 - Pregnancy test

**Investigational Medicinal Product: Not Treated** 

| Subject<br>ID | Time Point | Urine Collection Date/time | Pregnancy Test<br>Result |
|---|---|---|---|
| Sjjj/nnn | Screening | ddMMMyyyy hh:mm | Negative |
| Skkk/ppp | Screening | ddMMMyyyy hh:mm | Negative |
| Snnn/xxx | Screening | | |

Note: Subjects are listed according to the dose level of the product they actually received

Program: Listings\c122-xt-lst.sas




Statistical analysis plan CRO-14-122 Sponsor code CHL.1/02-2014 Chloroprocaine 1% - Spinal block Final version 1.0, 02FEB2016

#### Figure 16.2.5.j - Subject [Sxxx]/[nnn] - Individual plasma concentration curves of Chloroprocaine and CABA

Individual plasma concentration curves of Chloroprocaine and CABA (linear scale and logarithmic/linear scale)